

## SAĞLIK BİLİMLERİ ÜNİVERSİTESİ HAMİDİYE SAĞLIK BİLİMLERİ ENSTİTÜSÜ

# FETAL GELİŞİMİN ÖĞRETİMİNDE SANAL GERÇEKLİK UYGULAMASININ GELİŞTİRİLMESİ VE KULLANILMASI

## REYHAN AYDIN DOĞAN

TEZ DANIŞMANI PROF. DR. SAADET YAZICI

EBELİK ANA BİLİM DALI EBELİK DOKTORA PROGRAMI

> DOKTORA TEZİ EYLÜL/2021

## **İTHAF**

"Bana her zaman destek olan eşime ve aileme ithaf ediyorum"

### **TEŞEKKÜR**

Tezin her aşamasına çok büyük emeği ile yanımda olduğunu hissettiren, desteği ile beni motive eden, değerli zamanını bana özveriyle ayıran ve öğrencisi olmaktan onur duyduğum tez danışmanım kıymetli hocam Prof. Dr. Saadet YAZICI'ya,

Doktora sürecimde beni destekleyen ve yolumu aydınlatan, sevgisi, sabrı ve güler yüzü ile bana rol model olan değerli hocalarım Prof. Dr. Neriman ZENGİN, Prof. Dr. Nurten KAYA, Doç. Dr. Handan ÖZCAN ve Dr. Öğr. Üyesi Asiye AYAR KOCATÜRK'e,

Doktora tez sürecimde bana yoldaşlık eden ve bu süreci birbirimizden güç alarak tamamladığımız sevgili dostum Öğr. Gör. Sebahat HÜSEYİNOĞLU'na,

Doktora eğitim hayatım boyunca gelişmeme katkıları olan Sağlık Bilimleri Üniversitesi, Ebelik Bölümü hocalarıma,

Doktora tez sürecimde varlığını her zaman yanımda hissettiğim değerli hocam Doç. Dr. Nazan KARAHAN'a,

Doktora sürecimde bana desteklerini esirgemeyen Karabük Üniversitesi Sağlık Bilimler Fakültesi Dekanı Prof. Dr. Mehmet ÖZDEMİR ve Ebelik Bölümü başkanı Doç. Dr. Raziye ÖZDEMİR'e,

Doktora tez sürecimde benim kahrımı çeken sevgili dostlarım, Dr. Öğr. Üyesi Neriman GÜDÜCÜ, Dr. Öğretim Üyesi Sevgi DİNÇ, Dr. Ebe Seda SERHATLIOĞLU, Öğr. Gör. Sibel KARAKOÇ ve Uzm. Ebe Esra YILMAZ'a,

Bu araştırmayı 2020/113 proje numarası ile destekleyen Sağlık Bilimleri Üniversitesi Bilimsel Bilimsel Araştırma Projeleri Birimine,

Hayatımın her döneminde beni destekleyen annem Zehra AYDIN, babam Ali AYDIN, kardeşim Huriye AYDIN ve eşim Mert DOĞAN'a,

En İçten Dileklerimle Teşekkür Ederim.

# İÇİNDEKİLER

| İTHAF | iii |
|------------------------------------------------------------|-----|
| TEŞEKKÜR | iv |
| İÇİNDEKİLER | v |
| TABLOLAR LİSTESİ | vii |
| ŞEKİLLER LİSTESİ | ix |
| SİMGELER VE KISALTMALAR | x |
| ÖZET | xi |
| ABSTRACT | xii |
| 1. GİRİŞ VE AMAÇ | 1 |
| 2. GENEL BİLGİLER | 3 |
| 2.1. ÜREME ORGANLARININ ANATOMİSİ | 3 |
| 2.1.1. Kadın Üreme Organlarının Anatomisi | 3 |
| 2.1.2. Erkek Üreme Organlarının Anatomisi | 7 |
| 2.2. EMBRİYONEL- FETAL GELİŞİM VE FİZYOLOJİSİ | 9 |
| 2.2.1. Preembriyonel Dönem (Fertilizasyon ve İmplantasyon) | 9 |
| 2.2.2. Embriyonel Dönem | 10 |
| 2.2.3. Fetal Dönem | 11 |
| 2.2.4. Embriyo ve Fetüs Dışı Oluşumlar | 12 |
| 2.3. SANAL GERÇEKLİK KAVRAMI VE UYGULAMALARI | 14 |
| 2.3.1. Sanal Gerçekliğin Eğitimde Kullanımı | 15 |
| 2.3.2. Sanal Gerçekliğin Ebelik Eğitiminde Kullanımı | 17 |
| 2.4. FETAL GELİŞİMİN ÖĞRETİMİNDE SANAL GERÇEKLİĞİN KULI | |
| 3. GEREÇ VE YÖNTEM | |
| 3.1. ARAŞTIRMANIN AMACI | |
| 3.2. ARAȘTIRMANI HİPOTEZLERİ | |
| 3.3. ARAŞTIRMANIN ŞEKLİ | |
| 3.4. ARAŞTIRMANIN DEĞİŞKENLERİ | |
| 3.5. ARAŞTIRMANIN YERİ VE ZAMANI | |
| 3.6. ARAŞTIRMANIN EVREN VE ÖRNEKLEMİ | |
| 3.6.1. Randomizasyon | |
| 3.7. VERİ TOPLAMA ARAÇLARI VE GEREÇLERİ | 25 |

| | 3.7.1. Veri Toplama Araçları | . 25 |
|---|---|---|
| | 3.8. ARAŞTIRMANIN AŞAMALARI | . 28 |
| | 3.8.1. Araştırmanın Hazırlık Aşaması | . 29 |
| | 3.8.2. Araştırmanın Uygulama Aşaması | . 32 |
| | 3.8.3. Araştırmanın İzlem Aşaması | . 35 |
| | 3.9. VERİLERİN ANALİZİ | . 36 |
| | 3.10. ARAŞTIRMANIN SINIRLILIKLAR VE TAMAMLANMA SÜRECİNDE<br>KARŞILAŞILAN DURUMLAR | . 37 |
| | 3.11. ARAŞTIRMA SÜRECİNDE ALINAN COVİD-19 TEDBİRLERİ | . 38 |
| | 3.12. ARAŞTIRMANIN YASAL VE ETİK BOYUTU | |
| 4. | BULGULAR | . 40 |
| | 4.1. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN SOSYO-<br>DEMOGRAFİK/TANIMLAYICI ÖZELLİKLERİNE İLİŞKİN BULGULAR | . 41 |
| | 4.2. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN ÖĞRETİM<br>MATERYALLERİNE (SG UYGULAMASI ve TEORİ EĞİTİMİ) İLİŞKİN BİLG<br>DÜZEYLERİNE AİT BULGULAR | i<br>. 45 |
| | 4.3. DENEY GRUBUNDAKİ ÖĞRENCİLERİN SANAL GERÇEKLİK<br>UYGULAMASINA AİT BİLİŞSEL YÜK VE BULUNUŞLUK HİSSİ<br>DÜZEYLERİNE AİT BULGULAR | . 55 |
| | 4.4. DENEY GRUBUNDAKİ ÖĞRENCİLERİN DENEYİMLEDİKLERİ SAN<br>GERÇEKLİK UYGULAMASINDAKİ KALİTATİF GERİ BİLDİRİMLERİ | |
| 5. | TARTIŞMA | . 61 |
| | 5.1. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN SOSYO-<br>DEMOGRAFİK ÖZELLİKLERİNİN KARŞILAŞTIRILMASI | . 61 |
| | 5.2. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN ÖĞRETİM MATERYALLERİNE (TEORİ EĞİTİMİ VE VR UYGULAMASI) İLİŞKİN BİLO DÜZEYLERİNE AİT BULGULARIN TARTIŞILMASI | Gİ<br>. 63 |
| | 5.3. DENEY GRUBUNDAKİ ÖĞRENCİLERİN SANAL GERÇEKLİK<br>UYGULAMASINA AİT BİLİŞSEL YÜK VE BULUNUŞLUK HİSSİ<br>DÜZEYLERİNE AİT BULGULARIN TARTIŞILMASI | . 70 |
| | 5.4. DENEY GRUBUNDAKİ ÖĞRENCİLERİN DENEYİMLEDİKLERİ SANAI<br>GERÇEKLİK UYGULAMASINDAKİ KALİTATİF GERİ BİLDİRİMLERİNE A<br>BULGULARIN TARTIŞILMASI | İΤ |
| | SONUÇLAR VE ÖNERİLER | |
| | 6.1. SONUÇLAR | |
| | 6.2. ÖNERİLER | |
| K | AYNAKLAR | . 78 |
| П | ZIED | 0.5 |

## TABLOLAR LİSTESİ

| <b>Tablo 3.1:</b> G-powers analizi sonuç protokolü |
|---|
| Tablo 3.2: Randomizasyon ile belirlene deney ve kontrol grupları 23 |
| Tablo 3.3: Örnekleme ait grupların atanması 23 |
| <b>Tablo 3.4:</b> Araştırmanın uygulama ve veri toplama aşamaları 28 |
| <b>Tablo 3.5:</b> Veri analiz parametre ve istatistik yöntemleri |
| Tablo 4.1: Deney ve kontrol grubunun sosyo-demografik ve tanımlayıcı özellikleri 41 |
| Tablo 4.2: Öğrencilerin bilgisayar oyunu oynama ve sanal gerçeklik uygulaması bilgileri 43 |
| <b>Tablo 4.3:</b> Deney ve kontrol grubunun bağımsız değişkenler ile binary lojistik regresyon analizi 44 |
| Tablo 4.4: Deney grubundaki öğrencilerin fetal gelişim ölçeğine verdikleri doğru ve yanlış cevaplar 46 |
| Tablo 4.5: Deney grubundaki öğrencilerin ön test ve son test sonrası doğru cevap veren kişi sayısı |
| Tablo 4.6: Deney grubundaki öğrencilerin ön test ve son test cevaplarının karşılaştırılması 48 |
| Tablo 4.7: Kontrol grubundaki öğrencilerin fetal gelişim ölçeğine verdikleri doğru ve yanlış cevaplar (n:42) |
| <b>Tablo 4.8:</b> Kontrol grubundaki öğrencilerin ön test ve son test sonrası doğru cevap veren kişi sayısı |
| Tablo 4.9: Kontrol grubundaki öğrencilerin ön test ve son test cevaplarının karşılaştırılması 52 |
| Tablo 4.10: Deney ve kontrol gruplarının ölçek toplam puanlarının ön test ve son testlerinin karşılaştırılması 53 |
| Tablo 4.11: Deney, kontrol ve tüm grupların ön test ve son test puanlarının karsılastırılması 53 |

| Tablo 4.12: Deney ve kontrol gruplarında yer alan öğrencilerin fetal gelişimi |
|---|
| değerlendirme son test toplam puanlarının kovaryans analizi sonuçları |
| <b>Tablo 4.13:</b> Deney grubundaki öğrencilerin bilişsel yük puanları 55 |
| Tablo 4.14: Sanal gerçeklik deneyimleyen öğrencilerin bulunuşluk hissi ölçek alt |
| boyutları puan ortalamaları |
| Tablo 4.15: Bilişsel yük ölçeği ile bulunuşluk hissi ölçeğinin alt boyutları arasındaki |
| ilişki |
| Tablo 4.16:Sanal gerçeklik ile ilgili bilgi durumunun bulunuşluk hissi ölçeğinin alt |
| boyutları ile binary lojistik regresyon analizi |
| Tablo 4.17: Sanal gerçeklik ile ilgili uygulamaya katılma durumunun bulunuşluk hissi |
| ölçeği alt boyutları ile binary lojistik regresyon analizi |
| Tablo 4.18: Deney grubundaki öğrencilerin sanal gerçeklik bilgi ve deneyim durumları |
| ile bilişsel yük ölçeği arasındaki ilişki |
| Tablo 4.19: Sanal gerçeklik uygulamasını deneyimleyen öğrencilerin kalitatif geri |
| hildirimleri 59 |

## ŞEKİLLER LİSTESİ

| Şekil 3.1: G-power analiz sonucu | 22 |
|---------------------------------------------------------|----|
| Şekil 3.2: Araştırma akış diyagramı (CONSORT 2010) | 24 |
| Şekil 3.3: Oculups rift quest 2 sanal gerçeklik gözlüğü | 27 |
| Şekil 3.4: Araştırmanın hazırlık aşaması algoritması | 30 |
| Şekil 3.5:Araştırmanın uygulama aşaması- algoritma | 34 |
| Şekil 3.6: Sanal gerçeklik uygulama anı fotoğrafları | 34 |
| Sekil 3.7: Araştırmanın izlem aşaması | 35 |

### SİMGELER VE KISALTMALAR

**AGNO** : Ağırlıklı Genel Not Ortalaması

CONSORT : Consolidated Standards of Reporting Trials (Çalışmaların

Raporlanmasında Birleştirilmiş Standartlar)

FEGBÖ : Fetal Gelişimi Değerlendirme Bilgi Ölçeği

SG : Sanal Gerçeklik

SGT-FEGU : Sanal Gerçeklik Teknolojisi ile Oluşturulan Fetal Gelişim

Uygulaması

## FETAL GELİŞİMİN ÖĞRETİMİNDE SANAL GERÇEKLİK UYGULAMASININ GELİŞTİRİLMESİ VE KULLANILMASI

### ÖZET

Amaç: Bu araştırma, "Sanal Gerçeklik Teknolojisi ile Oluşturulan Fetal Gelişim Uygulaması (SGT-FEGU)" nun geliştirilmesi ve ebelik öğrencilerine verilen fetal gelişimin öğretiminde etkinliğini saptamak amacıyla gerçekleştirildi.

Gereç ve Yöntem: İzlemsel randomize kontrollü olan çalışma, Kasım 2019-Haziran 2021 tarihleri arasında, Karabük Üniversitesi Sağlık Bilimleri Fakültesi Ebelik Bölümünde gerçekleştirildi. Basit randomizasyon yöntemi ile (Deney =42, ve Kontrol =42) toplam 84 öğrenci örnekleme alındı. Araştırma üç aşamada gerçekleştirildi. İlk aşamada deney grubu için literatür doğrultusunda, fetal gelişimin 6. haftasında 40. haftaya kadar olan süreyi kapsayan SGT-FEGU oluşturuldu. Kontrol grubu için müfredat doğrultusunda fetal gelişim teori eğitimi hazırlandı. İkinci aşamada her iki gruba kişisel bilgi formu ve ön test uygulandı. Ön test sonrasında, deney grubuna oluşturulan SGT-FEGU, kontrol grubuna ise 2 saat süren teori eğitimi verildi. Verilerin toplanmasında, her iki gruba 12 sorundan oluşan soru formu ile ön-son test için araştırmadan bağımsız olarak, araştırma başlamadan önce araştırmacılar tarafından geliştirilen, "Fetal Gelişimi Değerlendirme Bilgi Ölçeği" kullanıldı. Deney grubuna ayrıca tek sorudan oluşan "Bilişsel Yük Ölçeği" ve "Bulunuşluk Hissi Ölçeği" uygulandı. Üçüncü aşama; ilk aşamadan 6 hafta sonra her iki gruba da son test uygulandı.

**Bulgular:** Deney ve kontrol grubundaki öğrencilerin yaş ortalaması sırasıyla, 22,38±0,88 ve 22,54±0,88 olarak saptandı. Deney grubunun son test puanı kontrol grubuna göre istatistiksel olarak anlamlı bulundu (p<0,05). Deney grubunun bilişsel yük puan ortalaması 1,09±0,29 olduğu, uygulamanın yük oluşturmadığı saptandı.

**Sonuç**: Fetal gelişimin öğretiminde geliştirilen SGT-FEGU'nun etkin ve ebelik eğitiminde uygulanabilir bir yöntem olduğu saptandı.

Anahtar Kelimeler: Ebelik, fetal gelişim, sanal gerçeklik

# DEVELOPMENT AND USAGE OF VIRTUAL REALITY APPLICATION IN TEACHING FETAL DEVELOPMENT

#### **ABSTRACT**

**Aim:** This research was carried out to develop the "Fetal Development Application Created with Virtual Reality Technology (SGT-FEGU)" and to determine its effectiveness in teaching fetal development given to midwifery students.

Materials and Methods: The follow-up randomized controlled study was carried out between November 2019 and June 2021 in the Department of Midwifery, Faculty of Health Sciences, Karabuk University. Eighty-four students were included in the sample using the simple randomization method (Experiment =42, and Control =42). The research was carried out in three stages. In the first stage, SGT-FEGU was created for the experimental group following the literature, covering the 6th week of fetal development to the 40th week. Fetal development theory training was prepared in line with the curriculum for the control group. In the second stage, a personal information form and a pre-test were applied to both groups. After the pre-test, the experimental group received SGT-FEGU, and the control group received 2 hours of theory training. In data collection, a questionnaire consisting of 12 questions was used for both groups. The researchers developed the "Fetal Development Evaluation Information Scale" before the research began, independently of the research, for the pre-post test. The "Cognitive Load Scale" and "Sense of Presence Scale" consisting of a single question were also administered to the experimental group. The third stage; Post-test, was applied to both groups six weeks after the first stage.

**Results:** The mean age of the students in the experimental and control groups was  $22.38\pm0.88$  and  $22.54\pm0.88$ , respectively. The post-test score of the experimental group was statistically significant compared to the control group (p<0.05). It was determined that the mean cognitive load score of the experimental group was  $1.09\pm0.29$ , and the application did not create a load.

**Conclusion:** SGT-FEGU, which was developed in fetal development teaching, was an effective and applicable method in midwifery education.

**Keywords:** Fetal development, midwifery, virtual reality

### 1. GİRİŞ VE AMAÇ

İnsan gelişimi ardı ardına gelişimsel süreçleri içeren bir döngüdür. Bu döngü erkek gameti olan sperm ile kadın gameti olan ovumun döllenmesi ile başlar. Döllenme sonucunda oluşan insan gelişiminin tüm genlerini taşıyan zigot benzersiz tüm oluşumların başlangıcıdır. Zigot, defalarca bölünür, farklılaşır, büyür ve tek hücreli halden çok hücreli insan yapısına dönüşür (1–3). Bu bölünmelerle birlikte embriyonel dönemde fetüs ve ekleri gelişir. Sürecin sağlıklı devam edebilmesi fetüsün ve plasentanın normal gelişimsel sürecinde devam etmesi ile mümkündür. Fetal gelişim süreci üç aşamada gerçekleşir. İlk aşama, fertilizasyondan ikinci haftaya kadar olan "preembriyonel" dönem, ikinci aşama fertilizasyondan sonraki on beş gün ile sekizinci hafta arasında geçen "embriyonel gelişim" dönemidir (1, 2, 4). Bu dönemde embriyo ve fetüs dışı oluşumlarda gerçekleşmektedir. Son aşama ise, sekizinci gebelik haftasının sonundan doğuma kadar olan "fetal dönemdir". Tüm bu aşamalarda normal büyüme, gelişme ve olgunlaşmanın bilinmesi maternal ve fetal komplikasyonları saptamada büyük önem taşımaktadır. Ebelik eğitiminde normal doğum ve riskli doğum eğitimlerinin gebelik ve fetal gelişim süreçlerinin öğretilmesinden sonra verildiği göz önünde bulundurulursa bu konuların ebelik öğrencileri tarafından iyi anlaşılması ve öğrenilmesinin gerekliliği ortaya çıkmaktadır.

Fetal gelişimin öğretiminde kullanılacak yöntemler gün geçtikçe gelişmektedir. Bu yöntemler, simülasyon eğitimleri, sanal gerçeklik, 3D görüntüleme ya da video destekli eğitimler olarak sıralanabilir (5). Literatür incelendiğinde ebelikte simülasyon eğitiminin, gebelik, doğum ya da doğum sonu dönemde daha fazla kullanıldığı görülmektedir (6, 7).

Ebelik eğitiminin temelini oluşturan gebeliğin, farklı eğitim teknikleri ile öğretilmesi, klinik uygulama hatalarını en aza indirecek, gebelik ve doğumda yaşanabilecek fetal prezantasyon ve plasental anomalilerinin erken teşhis edilmesin, sağlayacaktır. Bu teknikerlerle, özellikle sanal gerçeklik uygulamalarıyla öğrenciler, gebeliğin ilerleyen haftalarında oluşan farklılıkları ve maternal-fetal yanıtı etkin dönemde gözlemleyebilme fırsatını elde edecektir. Simülasyon eğitiminin ebeliğin, gebelik, doğum ya da doğum sonu dönemde etkin bir şekilde kullanıldığı görülmektedir (7–11).

Ebelikte simülasyon eğitimine sanal gerçeklik bakış açısının kazandırılması öğrencilerin klinik uygulamaya çıkmadan önce ebelik uygulamalarını etkin bir şekilde kullanmasını sağlayacaktır (12, 13). Ebelik eğitiminin temelini oluşturan gebeliğin sanal gerçeklik uygulaması ile öğretilmesi klinik uygulama hatalarını en aza indirerek, gebelik ve doğum yaşana bilecek fetal prezantasyon ve plasental anomalilerinin erken teşhisini sağlayacaktır. Gebelik ilerledikçe oluşan farklılıkları ve bu farklılıklara karşı maternalfetal yanıtı etkin bir şekilde görebileceklerdir. Sanal gebelik uygulaması ile ebelik eğitiminde herhangi bir engel olmadan gebelik sürecini, maternal- fetal gelişimi, plasental farklılıkları ve annenin dolaşımsal yanıtı üç boyutlu bir şekilde görmelerine olanak sağlayacak olan güncel ve önemli bir konudur (7–11).

Araştırma kapsamında, literatür ışığında haftalık gelişimler doğrultusunda hazırlanan "Sanal Gerçeklik Teknolojisi ile Oluşturulan Fetal Gelişim Uygulaması (SGT-FEGU) oluşturuldu. Oluşturulan program randomize kontrollü olarak seçilen ebelik öğrencilerine uygulandı.

Araştırma oluşturulan SGT-FEGU'nun ebelik eğitim müfredatı kapsamında verilen fetal gelişim teori dersinin etkisini saptamak amacıyla yapıldı. Bu doğrultuda araştırmanın hedefleri;

- Araştırmaya özgü tasarlanacak olan SGT-FEGU uygulamasının geliştirilmesi,
- Ebelik eğitiminde SGT-FEGU uygulamasının etkin bir şekilde kullanılmasının sağlanması,
- Ebelik eğitimine temel oluşturacak olan SGT-FEGU uygulaması ile fetal gelişimin görsel hale getirilmesi,
- Gebelik oluşumunun görselleştirilerek eğitim etkinliğinin klinik ve akademik başarıyı arttırmasıdır.

### 2. GENEL BİLGİLER

### 2.1. ÜREME ORGANLARININ ANATOMİSİ

Üreme organları insan neslinin devamını sağlayan ve üreme fonksiyonlarını yerine getiren oranlardır. İnsan neslinin sürdürülmesi için hem dişi hem de erkek üreme organlarının fonksiyonlarını sağlıklı bir biçimde sürdürmeleri gereklidir. Kadın anatomisinin üreme fonksiyonu erkek anatomisine göre daha karmaşık yapıdadır. Kadın anatomisi döllenmeyle başlayıp, gebelik süreci ile devam ederek doğumu gerçekleştirmektedir. Erkek anatomisinin üremedi rolü cinsel ilişki ile sınırlanmaktadır. Bu bölümde üreme anatomisi kadın üreme organları anatomisi ve erkek üreme organları anatomisi olmak üzere iki başlık altında incelenmiştir.

### 2.1.1. Kadın Üreme Organlarının Anatomisi

Kadın üreme organları fetal gelişimde büyük önem taşımaktadır. Kadın üreme sistem, fetal hayatın başlaması için gerekli olan ovumu üretmekle başlar, oluşan ovumu ampullada döller, dölleniş zigotu uterusa iletir ve uterusa gelen döllenmiş zigotun implantasyonunu sağlayarak fetüsün gelişim sürecini başlatır. Kadın üreme organları iç ve dış olmak üzere iki gruba ayrılır. Kadın dış genital organları perinede yer alırken iç üreme organları pelvis içerisinde yer almaktadır (14–20).

# **2.1.1.1. Dış üreme organları:** Kadın üreme sisteminde dış üreme organlarına vulva yada pudenta adı verilir (14, 15).

Dış Üreme Organları;

- Mons Pubis,
- Labia Major (Büyük dudaklar)
- Labia Minör (Küçük Dudaklar),
- Klitoris,
- Vestibül.
- Bulbus Vestibülleri
- Bartholin Bezleri
- Himen (Kızlık Zarı).

Mons pubis: Simfizis pubisin önünde kalan kabarık alana verilen addır. Simfiz pubisin önünde uzanan yuvarlak bir yağ yastığı olarak da tanımlanmaktadır (15). Puberte döneminden önce kılsız olan bu bölge ergenlik döneminden itibaren, normal deri kıllarına göre daha kadın olan kasık kıllarıyla kaplanır. Menopoz döneminden sonra bu kıllanma azalır (14–17, 19, 20).

Labia Major (Büyük dudaklar): Dış yüzeyi deri ve kasık kıllarıyla kaplı ve pembe, pürüzsüz bir iç yüzeye sahip mons pubisten aşağı doğru uzanan iki deri kıvrımıdır. Sinir ve damar yönünde zengin, ön kısmı kalın aşağıya doğru indiğinde incelen, 7-8 cm uzunluğundaki dokulardır. Labia majörlerin alt kışında birleştiği yer ile anüs arasında kalan bölge de **perine** olarak adlandırılır (14, 15, 17, 18, 20).

Labia Minör (Küçük Dudaklar): Labia majorler arasında uzanan, yağ içermeyen iki küçük deri altı kıvrımdır. Erkek üreme sistemindeki karşılığı penis derisidir. Üzerinde kıl bulunmayan, kırmızı pembe renge sahip, 3-3,5 cm. uzunluğunda olan iki küçük deri plakası şeklindedir. İç yüzünde bol miktarda duyu reseptör bulunmakta ve mukozası vajinaya benzerdir. Labia minörler klitoris yakınında ili kola ayrılır. Üst kola prepisyum adı verilir ve bu kol klitorisi üstten sarar. Alt kol ise klitorisi alttan sararak frenulum klitorisi oluşturur. (14, 15, 17, 18, 20, 21)

Klitoris, erkek penisine karşılık gelen küçük, ilkel bir cinsel organdır. Görünümü topuza benzeri kapartı şeklindedir. Üretra ve vajinanın açıklığının üzerinde, labia minorlerin ön birleşim yerinin yakınında yer alır. Penisin aksine, klitoris üretranın distal kısmını içermez ve yalnızca cinsel ilişki sırasında orgazmı sağlamak için işlev görür. Çok sayıda sinir uçları içerir ve uyarılınca ereksiyona uğrar. Herhangi bir darbe aldığında ya da yırtıldığında çok fazla kanamaya neden olur. (14–17, 20, 21).

Vestibül: Üretra ve vajina açıklıklar yer edildiği küçük dudak tarafından çevrelenen bir alandır. Ayrıca labia minörler aralandığında görülen bulbus vestibulleri ile çevrelenmiş üçgen bölge şeklinde de tanımlanmaktadır. Bu üçgen bölgenin tepesini klitoris, yanlarını labia minörler, alt kısmını ise labia minörlerin birleşme kısmı oluşturmaktadır. Vestibüler bölgede himen ve kalıntıları da yer almaktadır (14, 15, 21).

**Bulbus Vestibülleri:** Vajinal açıklığı çevreleyen iki uzun erektil oluşumdur. Arka kısmı kalın, öne doğru incelen bir yapısı vardır. Kalınğı 0,5 cm., uzunluğu 3,5 cm.'dir. Erkekte karşılığı korpus spongiosum dur. (14, 15, 17, 19–21).

Bartholin Bezleri/ Büyük vestibüler bezler: Vajina ağzının her iki tarafında açılan ve labia majorlerin arka kısmında yer alan iki adat nohut büyüklüğünde olan küçük bezlerdir. Erkek cinsel organında karşılığı cowper bezleridir. Cinsel ilişki ya da uyarılma sırsında salgıladıkları müköz salgı ile vajinal kayganlığı sağlarlar. Kanal bazen tıkanabilir, bu da bezden gelen salgıların içine birikmesine ve bir kist oluşturmasına neden olabilir. Bu iltihaplı kiste" bartolinitis" adı verilir. (14, 15, 17, 19–21).

Himen (Kızlık Zarı): Perde anlamına gelen yunanca bir kelimedir. Vajina ile vestibulum vajina arasında yer alan, mukoza plikası şeklinde esnek bir zardır. Tamamen kapalı olmayan bu zarın, adet kanını dışarıya atmasını sağlayan bir veya daha fazla deliği vardır. Himen tipleri bu deliklerin şekillerine göre adlandırılır. İntrauterin 6. Aya kadar himen deliksiz perde şeklindedir. Himen şekil ve farklılık olarak bireysel değişiklikler göstermektedir. Genellikle ilk cinsel birleşme sırasında yırtılır ve bir miktar kanama olur (14, 15, 17, 21, 22).

# **2.1.1.2. İç üreme organları:** Kadın iç üreme organları kemik pelvis içinde yer alan organlardır.

İç üreme organları;

- Vajina,
- Uterus,
- Fallop tüpleri,
- Overler.

Vajina: Vestibulumdan uterusa kadar uzanan 8-10 cm. uzunluğunda olan organdır. Kanal şeklinde bir organ olup, kaslardan oluşmakta ve genişleyip daralma özelliğine sahiptir. Vajinanın önünde mesane ve üretra, arkasında rektum, üstünde ise uterus ile komşudur. Vajina girişinin 1-2 cm ilerisinde himen vardır. Vajinanın üst bölümü halka şeklinde serviksi çevreler. Serviksin vajina içinde kalan bu bölümüne porsio denir. Vajina duvarı ile porsio arasında forniks adı verilen girintiler yer alır. Bu girintilerden en derini olan arka forniks ilişki sırasında spermlerin biriktiği alandır. Vajinanın pH'sı asidiktir. Bu özelliği sayesinde iç üreme organlarını enfeksiyonlardan korur. Vajinanı fonksiyonları arasında, doğumda doğum kanalının son bölümü oluşturmasının yanı sıra, menstürasyon sırasında kanı dışarı akmasını ve cinsel birleşmeyi sağlaması yer alır (14, 16–20).

İç yüzeyi çok katlı yassı epitel hücrelerden oluşan vajina, salgı bezi olmamasına rağmen, dökülmüş epitel hücreleri, bakteri salgıları ve servikal akıntı nedeniyle mukozası her zaman nemli ve ıslaktır. Vajina epiteli hormonların etkisi altında kalır ve vajinal akıntının incelenmesi kadının hormonal durumu ile ilgili bilgi sahibi olmamızı sağlar (14, 15, 21–23).

Uterus: Pelvis boşluğunda rektum ile mesane arasında yer alan, kalın duvarlı, içi boş, önden arkaya basık, kaslı, ortalama uzunluğu 6-7 cm olan ve vajinanın üstüne yerleşmiş bir organdır. Yanlarında follop tüpleri, arkasında rektum, önünde ise mesane yer alır. Normalde 30-60 gr. ağırlığında olan uterusun, gebelikte hacmi artar, şekil ve pozisyonu değiştirir. Doğumdan sonra da eski halini alır. Uterusun normal pozisyonu anteverisyo ve anteflexiodur. Uterus görevleri; sperimin serviksten tubaya geçmesini, döllenmiş yumurtanın yerleşmesi için uygun ortamın hazırlanmasını, fetüsün korunması ve beslenmesini, doğum eylemininde fetüsün ve eklerinin atılmasını ve mesntürasyon kanamasının oluşmasını sağlamaktır. Uterus fonksiyon ve yapı olarak, korpus, serviks, istmus ve fundus olmak üzere dört bölümde incelenir (14, 15, 21–23).

- Korpus, follop tüplerinin uterusa açıldıkları seviyenin altında kalan bölge ile istmusa kadar uzanan alandır. Genişliği 5cm, uzunluğu ise 4-6 cm'dir. Korpus içinde üçgen şeklinde olan kovum uteri yer almaktadır. Bu üçgen bölgenin alt kısmı servikal kanal ile devam eder (14, 17, 19–21).
- Serviks (Kollum), Uterusun vajinaya açılan üçte birlik alt kısmıdır. Mikroorganizmaların uterusa ulaşmasını önler. Dış kısmına ostium eksternum denir. Bu bölge doğum yapmış kadınlarda çizgi şeklinde (yuvarlağı kaybolmuş), hiç doğum yapmamış kadınlarda da yuvarlak şeklinde görülür. Serviks fetal gelişimde erken doğumu önlemek ve düşükleri önlemede büyük önem taşır (14, 17).
- İstmus, bir santim uzunluğunda korpus ile serviks arasında kalan bölgedir.
- **Fundus,** follop tüplerinin uterusa açıldıkları bölgenin üzerinde kalan uterusun üst bölümüdür. Gebelikte, fetusun boy ve kilo tahmini için yapılan birinci leopold manevrası sırasında ölçülen yerdir. Doğumda ya da erken doğum tehdidinde uterin kontraksiyonlarının ölçüldüğü alandır (14, 16–18, 21).

**Uterusun tabakaları,** dışta perimetrium, ortada miyometriyum ve içte endometriyumdur. Endometriyum gebelikte desidua adını alır. Miyometriyum tabakası

kas tabakasır ve doğumda motor gücü oluşturur. Perimetium ise uterusu örten en dış tabakadır ve bağırsakların uterus üzerindeki kayganlığını sağlar (14, 17, 21–23).

**Uterusun ligamentleri (bağları),** ligamentum latum (broad/geniş bağ), ligamentum rotundum (rount/yuvarlar bağlar), Ligamentum kardinale ve ligamentum sakrouterinedir. Bu bağlar uterusun anatomik yapısını korumasını sağlamanı yanı sıra uterusu yerinde tutan yapılardır (16, 17, 19–23).

Fallop tüpleri: Uterusun her iki yanında yer alan ve broad ligament boyunca uzanan ortalama 8-10 cm olan yapılardır. İnfindibulum, ampulla, istmus ve intramural olmak üzere dört bölümden oluşur. Ampulla kısmı döllenmemin olduğu bölümdür. Bu bölüm fetal sürecin başlangıcı (döllenmenin gerçekleştiği bölge) olması nedeniyle büyük önem taşır. Follop tüplerinin görevleri; döllenmede spremlere bir geçiş yolu oluşturmak, ovumu yakalayıp içine almak, döllenme için uygun ortam oluşturmak, döllenmiş ovumun beslenmesini sağlamak ve uterusa taşımaktır (14, 16–19, 21, 23).

Overler: Uterusun her iki tarafında olan badem şeklideki organlardır. Ligamentum latumun arkasında fossa ovarikaya yerleşmiş pembensi renkte olan ve ortalama 5 gr ağırlığında çift organlardır. Korteks (dış) ve medulla (iç) olarak iki tabakadan oluşur. Kortek kısmı, primordiyal foliküllerin bulunduğu yerdir. Medulla tabakası ise, bağ dokusu, sinir, lenf ve kandan zengindir. Overler, ovumu ve kadınlık hormonları olan progesteron ve östrojeni üretir (14, 16, 17, 19, 22, 23).

### 2.1.2. Erkek Üreme Organlarının Anatomisi

Erkek üreme anatomisi kadında olduğu şekilde iç üreme organları ve dış üreme organları olmak üzere iki başlıkta incelenmektedir (17, 21–23).

# **2.1.2.1. Erkek dış üreme organları**: Erkek dış genital organları penis ve skrotumdan oluşur.

**Penis:** Cinsel birleşme ve idrar boşaltma organıdır. İki adet kovpora kavernosa ve bir adet korpus spongiosum olmak üzere iç silindirik süngerimsi tabakası bulunur. Sünnet derisi ile çevrili kısmına glans penis olarak adlandırılır. Bu bölge sinirlerden zengindir ve oldukça duyarlıdır. Penisin görevleri, cinsel ilişki sırasında ereksiyonlaraka vajinaya ulaşarak erkek semen sıvısını arka fornikse bırakmak, sprem ve idrarı üretraya taşımaktır (17, 21–24).

**Skrotum:** Penisi altında yer alan ve içinde iki testisin yer aldığı torba şeklinde organdır. Spermatik kordları ve testisleri içinde taşır. Şekli ve boyutları yaşa göre farklılık gösterir. Yenidoğan döneminde daha sert ve yukarıda iken, yetişkinlik dönemine geldikçe yumuşak ve büyük hale gelir (17, 22–24).

**2.1.2.2.** Erkek iç üreme organları: Erkek iç genital organları, testisler, epididimis, vas deferens/ductus deferens ve erkek eklenti bezlerinden oluşur.

**Testisler,** oval şekilli olan, skrotumun içinde asılı olarak duran, sperm ve testesteron üreten bir çift organdır. Kadın üreme organlarındaki ovaryumların karşılığıdır. Normal fonksiyonlarını yapabilmeleri için skrotuma yerleşmeleri gereklidir (16–19, 21–25).

**Epididimis:** Spermiumların olgunlaşmaya eriştiği, testisler üzerine yerleşmiş 5-6 cm uzanlığında kıvrımlı kanallar topluluğudur (16–18, 22–24).

Vas deferens/ductus deferens: Epididimisten sonra gelen ve sadece iletim işlevi olan bölümdür. Müsküler duvar yapısı nedeniyle kadın üreme organlarından follop tüplerinin karşılığıdır (17–19, 22–24).

**Erkek eklenti bezleri:** Seminal vezikül bezler, prostat bezi, semen kesecikleri ve cowper bezleridir.

Seminal vezikül, mesanenin arka yüzü ile rektum arasında yer alan iki adet salgı bezidir. Semenin %60-70'ini oluşturur. Bezin salgılama fonksiyonu testesteron hormonu tarafından düzenlenir (16, 17, 19, 23, 24).

Prostat bezi, idrar kesesinin altında yer alan, sert, kıvamlı, kestaneye benzeyen bezdir. İçerisinde, çinko, prostaglandin, fosfat, pıhtılaşma enzimi, prostat spesifik antijeni, kalsiyum ve profibrinolozin içeren alkali süte benzer sıvı salgılar (17, 19, 24).

Semen kesecikleri, cinsel ilişkide orgazm sırasında atılan ejekülat olarak adlandırılır. 1 ml semen içinde 40-120 milyon sperm bulunur. Miktarı ereksiyon sıklığı ile değişiklik gösterir (17, 18, 22–24).

Cowper bezleri, bezelye büyüklüğünde olan ve prostatın altında yer alan bezdir. Salgıladığı alkali sıvı sayesinde üretranın yüzeyin idrarın irritan etkisinden korur (16, 17, 22, 24).

### 2.2. EMBRİYONEL- FETAL GELİŞİM VE FİZYOLOJİSİ

### 2.2.1. Preembriyonel Dönem (Fertilizasyon ve İmplantasyon)

İnsan gelişimi yüzyıllardır açıklanmaya çalışılmış, başta karmaşık gibi görülen bir süreç olarak görülmüştür (17, 25, 26). Sağlıklı ve canlı bir fetüsün dünyaya gelmesi, sağlıklı bir gebeliğin oluşması, sürdürülmesi ve başarılı bir şekilde de sonuçlanması gereklidir (2, 17, 25). Düzenli bir menstürasyon döngüsü olan bir kadının gebe kalma ihtimali yalnızca %30'dur (25, 27). Bu süreci göz önünde bulundurduğumuzda gebeliğin oluşumu ve fetüsün süreç içindeki gelişimi büyük önem taşımaktadır.

**Fertilizasyon:** Yumurta ve spermin follop tüplerinin ampulla kısmına karşılaşıp döllenme aşamasıdır. Follop tüplerindeki fimbrialar oositin over yüzeyinden follop tüplerinin içerisine alınmasını sağlar. Östrojenin etkisi ile follop tüplerinin peristaltik hareketleri arta ve oositi döllenmek için ampullaya hareket eder (2, 17).

Spermin döllenme için taşınması içi farklı fizyolojik süreçlerden etkilenir. Cinsel ilişki ile yaklaşık üç yüz milyon spremium seminal sıvı ile vajinaya boşalır. Spemiumler vajinadan serviks, uterus ve follop tüplerine kendi hareketleri ile ilerlerler. Orgazm durumunda uterus ve vajinanın ritmik kasılmaları spremlerin bu hareketine yardım eder (2, 17, 18, 23, 26).

Follop tüplerinin ampulla kısmında spremium oosit ile karşılaşır. Spremin baş kısmında bulunan tripsiklinize ve hyloranidaz enzimleri oositin zona pellisudasını eriterek, tek bir sprem hücre içerisine penetre olur ve döllenme gerçekleşir. Döllenme sonrası spermin ve oositin nükleusları büyüyerek "erkek ve kadın pronukleus" adını alır. Sprem ve ovumda yarıya inen kromozom sayıları döllenme ile birleşerek 46 kromozomlu yeni bir hücre oluşturur. Oluşan bu yenir hücreye zigot adı verilir (1, 2, 4, 17, 28, 28, 29).

Zigot uterusa ortalama yedi gün içinde ulaşır. Bu sürede zigot hızlı bir şekilde bölünerek önce iki hücreli yapı olan blastomer, sonra da 16 hücreli yapı olan morulaya dönüşür. Zigot uterusa ulaştığında morula halindedir.

Endometrium döllenme sürecinde mukus salgısını arttırır, implante olacak zigotun beslenme ve gebeliğin devamlılığını sağlamak için hazır hale gelir. İmplantasyon gerçekleşene kadar zigotun beslenme sürecini uterusun içindeki endometrium sıvıları gerçekleştirir. Bu süreçte emdometrium sıvıları morula aşamasındaki zigotun içerisine girerek ortasında toplanır ve blastomer hücreleri kenarlara doğru itilir. Blastomerlerin bir

kısmı yassı olarak itilirken diğer bir grup bir noktada kitle halinde kalır. Bu görüntüdeki yapı taşlı yüzüğe benzetilir. Taşlı yüzüğün halkasını trofoblast hücreleri, taşını ise embrioblast hücreleri oluşturur. Traofoblastlardan plasenta ve ekleri, embriyoblastlardan da embriyo oluşur (1, 2, 4, 17, 28).

**İmplantasyon:** Fertilizasyondan sonraki ortalama olarak yedi gün sonra ve blastosist safhasında meydana gelir. Blastosistin etrafını çevreleyen zona pellusida kaybolur ve trofoblast hücreleri endometriuma yerleşir. İmplantasyon süreci fertilizasyonda sonra on günde tamamlanır. Endometrium implantsyon sürecinde, fetüsün gelişimi için damardan zengin hale gelerek desidua adını alır (1–3, 17, 26, 28).

İmplantasyondan sonra trofablast hücreleri enzimler salgılayarak lakuna adı verilen kan gölcüklerini oluşturur. Oluşan lakunalar plasental dolaşım başlayana kadar oluşan embriyoyu besler (1, 2, 17, 26, 28).

Fertilzasyonu takiben iki hafta içerisinde preembriyonel dönem başlar ve fetüsün gelişim süreci de görünür hale gelmiş olur (2, 17).

Preembriyonel dönem, fertilizasyondan başlayıp ikinci haftaya kadar olan dönemdir. Fertilizasyo ile implantasyon dönemlerini kapsar. İnsan yaşamının ilk adımları sperm ile ovumun ampullada birleşmesi ile başlamış olur. Fertilizasyondan sonra zigot ismini alan, 46 kromozomdan oluşan bu hücre, kendi içinde bölünmeler geçirerek, blastomer, morula ve blastosist haline gelerek olgunlaşır. Bu evrede bir yandan trofoblast hücreleri endometriuma yerleşirken, diğer yandan embriyoblast hücreleri, endoderm, ektoderm ve mezoderm olmak üzere üç germ yaprağını oluşturmaya başlar. Bu süreç gastrulasyon olarak tanımlanmaktadır. Bu üç germ yaprağında fetüsü sistem ve organları gelişir. Preembriyonel dönem yerini fertilizasyonun ikinci haftası sonrası embriyonel döneme bırakır (2, 17, 30–33).

#### 2.2.2. Embriyonel Dönem

Embriyonel dönem fertilizasyonun 15. gününde başlayıp sekizinci haftanın sonuna kadar geçen süredir. Bu süreçte zigot embriyo adını alır. Bu dönemde organlar hızlı bir şekilde geliştiğinden organagenezis dönemi olarak da bilinir (2, 17, 31, 34). Organların gelişmesi ile embriyonun şeklide değişir ve gelişir. Bu evre organ gelişim süreci olduğundan fetal gelişimde çok kritik dönemdir. Bu dönemde, ilaçlar, enfeksiyonlar, beslenmeye yetersizliği ya da radyasyona maruz kaldığında embriyoda

organ hasarı meydana gelir. Preembriyonel evrede oluşmaya başlayan üç germ yaprağı bu evrede tamamlanır. Bu germ yaprakları endoderm, ektoderm ve mezodermdir. Endoderm, solunum sisteminin iç tabakasını, sindirim kanalını, karaciğer ve pankreas gibi çok önemli bazı organların bir bölümünü meydana getirir. Ektoderm, beyin, omurga, sinirler, deri tırnaklar ve saçları oluşturur. Mezoderm ise kalp, böbrekleri, kemikleri, kıkırdakları, kasları, kan hücrelerini, ve diğer yapıları oluşturur (25, 31–37).

Embriyonun yaşamındaki ilk gelişmeye başlayan sinir sistemidir. Ektoderm döllenmeden sonraki 3.-4. haftalarında yukarı doğru katlanarak nöral tüpü oluşturur. Bu katlantının üst kısımları beyin hücrelerini oluşturmak için yükselir. Sinir sistemi gelişirken fetal kalp atmaya başlar. Fetal kalp atım hızı 6. gebelik haftasında ultrasonografi ile izlenir ve dışarıdan duyulacak hale gelir. Omurgalar, kaburga, gözler, kulaklar, çene ve boyun şekillerin. Bu evrenin sonunda (8. haftada) embriyo insana özgü görünümünü alır. Embriyonun pozisyonu dikleşmiştir (1–3, 29–31, 34, 37).

#### 2.2.3. Fetal Dönem

Fetal dönem, gebeliğin 8. Haftasından doğuma kadar olan, prenatal gelişimin en uzun olduğu dönemdir. Bu dönemde embriyo fetüs adını alır. Fetal dönem organageneziste oluşmuş olan organların büyümesi ve gelişmesi olarak düşünülebilir. Bu dönemde fetal başın büyüme hızı yavaşlar ve vücudun büyüme hızı artar.

Fetüsün büyüme ve gelişme sürecin, hem üç aylık periyotlar olan tremesterler olarak ele alınır hem de dört haftalık (aylık) olarak ele alınmaktadır (2, 17, 34, 37, 38). Araştırma kapsamında tasarlanan SGT-FEGU'da fetal dönem dört haftalık periyotlar şeklinde ele alınmıştır (2, 34, 36, 38).

- 9-12. hafta: Fetal dönemim başlangıcı olan haftadır. Bu haftada cinsiyet farklılaşması devam eder. Sindirim sistemi hareketlilik gösterir. Fetüsün başı hala vücuduna göre orantısız olarak büyüktür. Yüz genişler, gözler birbirinden ayrılır e göz kapakları kapalıdır. Diş tomurcuklarının 20 tanesi sıralanır. Karaciğerden kırmızı kan hücreleri üretilir. Bu haftalarda boy 2,3- 5,4 cm arasında, kilo 2-14 gram arasındadır (2, 17, 32, 34, 37, 38).
- 13-16. haftalar: Bu haftalarda lonuga tüyleri gelişir. Fetüsün derisi tamamen saydamdır. Kemikler sertleşir. Bağırsakların gelişimi 13. haftada başlar. Fetüs aktif hareket eder. Bu döneminde sonunda anne tarafından bebek hareketleri hissedilebilir. Bu

haftalarda boy 7,4- 11,6 cm arasında, kilo 23-100 gram arasındadır (2, 17, 28, 29, 34, 36, 38).

- **17-20. haftalar:** Bu haftalarda beyin büyümesi hızlanır. İdrar oluşur. Verniks kazeoza fetüsün yüzeyini kaplar. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Fetüsün saçları 19. haftada çıkmaya başlar. Bu haftalarda boy 13- 16,4 cm arasında, kilo 140-300 gram arasındadır (2, 17, 29, 34, 36).
- **21-24. haftalar:** Kaş ve kirpikler şekillenmemiştir. Akciğerlerde alveoller şekillenmiş ve sürfaktam oluşumu başlamıştır. Bu haftalarda boy 25,6- 28,9 cm arasında, kilo 300-501 gram arasındadır.
- **25-28.** haftalar: Sinir sistemi bazı fonksiyonlarını kontrol etmeye devam eder. Kan hücrelerinin yapımı dalaktan kemik iliğine geçer. Beyin hızla gelişmeye devam eder. Bu haftalarda boy 30- 36,6 cm arasında, kilo 600-875 gram arasındadır (2, 17, 29, 34, 36).
- **29-32.** haftalar: Fetal kemikler 29. haftada sertleşmeye başlar. Vücut yağ kitlesi hızlıca artar. Akciğerler tam olarak olgunlaşmamıştır. Bu haftalarda boy 37,6- 41,1 cm arasında, kilo 1005-1502 gram arasındadır (2, 17, 34, 36, 38).
- **33-36. haftalar:** Lonuga tüyleri dökülmeye başlar. Anneden fetüse antikor geçişi olur. Fetus uterusu dolduracak kadar büyümüştür. Vücut yağ kütlesi giderek artmıştır. Bu haftalarda boy 42,4- 46,2 cm arasında, kilo 1702- 2383 gram arasındadır.
- **37-40. haftalar:** Fetüsün tırnakları ve saçları uzamaya devam eder. Dersi pembe ve yumuşaktır. Bu haftalarda boy 47,4- 50,7 cm arasında, kilo 2622- 3288 gram arasındadır. Dış dünyada yaşamak için uygun zaman bu haftalar içerisindedir (2, 17, 34, 36, 38).

### 2.2.4. Embriyo ve Fetüs Dışı Oluşumlar

Fetüs dışı oluşumlar, plasenta, umblikal kord ve fetal membranlar olarak sıralanabilir.

**Plasenta:** Yaklaşık 200 adet koryonik villüsün birleşerek oluşturduğu yapıdır. Bu yapıla birkaç villüs birleşerek kotelodan adı verilen lobları oluşturur. Gelişimi gebeliğin üçüncü ayında tamamlanır. Doğum zamanına geldiğinde kilosu 400-600 gr arası, çapı 15-20 cm ve kalınlığı 2,5-3 cm'ye ulaşır. Fetüs ile anne arasında gaz ve madde değişimi

yapmak başlıca görevidir. Bunun dışında; solunum, beslenme, hormon üretimi, mikroorganizmalardan koruma ve atılım görevleri vardır.

**Umbilikal kord:** Gebeliğin 3-4. Haftalarında plasentanın gelişimi ile birlikte oluşmaya başlar. Embriyo ve plasenta arasında yer alan yaşamsal bir bağdır. Warton jeli adı verilen destek doku ile çevrilidir. Worton jelinin içinde iki arter ve bir venden oluşur. 1-2 cm çapında ve ortalama 55 cm uzunluğundadır. Umblikal kordun uzun ya da kısa olması fetal komplikasyonlara neden olabilir (2, 30, 34, 36–38).

Fetal membranlar: Fetal membranlar implantasyonla şekiilenmeye başlar. İçte amnion dışta da kariyon olmak üzere iki adettir. Amniyon ve koriyon başta birbirinden ayrıdır. Gebelik haftası ilerledikçe amniyotik kavite koriyonik kaviteyi doldurur. Bu iki membran plasentanın fetal yüzüne tutunmuştur.

Koriyon zarı, en dıştaki ilk tabakadan oluşur. Trofoblastik hücrelerden gelişir ve çok sayıda koyonik villüs uzantılarından oluşur. Bu koryonik villüslerden gebeliğin ilk tremesterinde (8-11. taftalarda) genetik tanı testi için yararlanılır.

Amniyon zar ve içerinde bulunan sıvıdan oluşur. Amniyon zarı, fertilizasyonun 7-8. gününden sonra embriyonun dorsal yüzeyinde şekillenir. Başlangıçta koriyonik kese içinde birbirine yakın şekilde yer alırken gebelik ilerledikçe tüm uterin kaviteyi kaplar. Amniyon zarının içerisinde amniyon sıvısı bulunmaktadır.

Amniyon sıvısı, gebelik başlangıcında fetal membranlar ve ciltten trasnsüdasyon yoluyla oluşur. Amniyon sıvısınıj içeriği gebelik ilerledikçe farklılık göstermektedir. Başlangıçta ekstraselüler sıvı iken, gebelik ilerledikçe protein konsantrasyonu düşer. İlk tremeseterde pH 7,22 iken ikinci tremesterde 7.12'ye düşer. Bu değişim fetal idrarın amniyos sıvısına katılmasından kaynaklanmaktadır. Amniyos sıvısının miktarı da gebelik ilerledikçe artış göstermektedir. İlk tremesterde 50 ml iken doğuma yaklaşıldığı son günlerde 800 ml civarına ulaşmış olur. Amniyon sıvısı fetüsün epitel hücreleri, lonuga tüyleri, çeşitli enzimler, üre, ürik asit, albümin, bilirübin, lökosit gibi birçok içerikten oluştur. Amniyon sıvısının fetüs için önemli işlevleri vardır. Bu işlevler; fetüsü travmalardan korumak, fetüsün kolay hareket edebilmesini sağlamak ve olası yapışıklıkları önlemek, fetüsün vücut ısısını korumak, umblikal kordo olan basıyı engellemek, fetüsün akciğer gelişimine katkıda bulunmak, doğumda hidrolik basınç oluşturarak iti güç sağlamak, doğumda doğum kanalını aseptik sıvı ile yıkanmasını

sağlamak ve içinde taşıdığı fetüse ait özellikler ile fetüsün sağlık durumu hakkında bilgi vermektir.

Fetal gelişim ebelik eğitiminde büyük önem taşımaktadır. Bu sürecin sağlıklı bir şekilde bilinmesi, ebelik eğitiminin temelini oluşturan normal ve riskli gebelik derslerinin iyi bir şekilde anlaşılmasını sağlayacaktır.

### 2.3. SANAL GERÇEKLİK KAVRAMI VE UYGULAMALARI

Sanal gerçeklik uygulamaları, bir den fazla kullanıcı ile çalışabilen, online (çevrim içi) platformda erişim sağlanan, kullanan kişilerin içinde bulundukları ortam ve diğer kullanıcılarla etkileşime geçmesini sağlayan, bireysel ya da ekip ile eğitim, oyun, öğrenme gibi bir çok alanda kullanılabilen sistemlerdir (5, 39–44). Sanal gerçeklik (SG) uygulaması 1980'li yıllardan günümüze kadar gelmiştir. Bu teknoloji 1990'lı yıllarda ivme kazanmıştır. Bilgisayar ortamına aktarılan üç boyutlu resimlerin teknoloji SG uygulaması ile birleşmesi insanların zihninde gerçek bir ortamda bulunma hissi oluşturmaktadır (40, 43–46). Tüm bu tanımlar çerçevesinde SG, kullanan kişiye güçlü bir bulunuşluk hissi vererek bulundukları ortamda deneyim yaşama şansı sunar (40, 43, 45– 47). Sanal gerçeklik uygulamalarının, süreklilik, görsel gerçeklik ve etkileşimden oluşan üç temel unsur bulunmaktadır (40, 48, 49). Görsel gerçeklik ve etkileşim unsurları, öğrenme, beceri kazanma ve bilgiyi kalıcı hale getirmede önemli iken, sürekliliğin, kullanıcıyı tamamen çevreleyerek bulunduğu ortama ait hissetme unsurunu oluşturmaktadır (40, 45, 46, 48, 49). Bu üç ana unsurun yanı sıra ayrıca SG uygulamalarında üç ana tanımlayıcı boyuttan da bahsedilmektedir. Bu ana boyuttan birincisi gerçeklikte hassaslıktır. Gerçeklikte hassaslık, ses, görüntü, tat ve koku gibi fiziksel duyarlılıkları kapsar. İkinci ana tanımlayıcı aktif katılımdır. Aktif katılım, SG uygulamaları için büyük önem taşır. Kullanıcıların etkileşim halinde olmasını ve deneyimledikleri ortama aktif olarak katılımlarını kapsar. Üçüncü ve en son temel gösterimin doğruluğudur. Bu süreç katılımcıların gösterimdeki doğrulukları algılamaları ve gerçeklik ile uyumu tanımlar. Bu üç ana temelin SG'de bir arada bulunması kullanıcılardaki olumlu deneyim ve öğrenim sürecini arttırmaktadır (46, 50–52).

Sanal gerçeklik uygulama alanları incelendiğinde, ilk dikkat çeken video oyunları ve eğlence alanları olduğu görülmektedir (53, 54). Doksanlı yıllarda SG teknolojisi ile kurulmuş oyun alanları Japonya ve Amerika'da görülmektedir. Oyun alanlarının yanı sıra çöpçatanlık servisleri olarak kullanıldığı da bildirilmiştir (54). Sanal gerçekliğin turizm

ve inşaat alanında kullanılmıştır (53, 55–58). Örneğin Fransız devrimi sonrası yıkılan 'The abbey of Cluncy' önceki kayıtlar sayesinde SG ortamına aktarılmıştır (55). Aynı zamanda modern yapılanma ve şehir planlama alanlarında da kullanış ve kullanılmaya devam edilmektedir (53, 59–61). Sanal gerçeklik uygulamasının kullanıldığı ticaret servisleri de gün geçtikçe yayınlaşmıştır (62–67). Sanal gerçeklik uygulamasının eğitim ve öğretim alanında kullanımı dikkat çekmiştir. Eğitim alanları Fizik, Fen, Tıp, Astronomi, Hemşirelik, Ebelik, Tarih ve Din eğitimi örnek gösterilebilir (39, 43, 50, 68, 68–76).

### 2.3.1. Sanal Gerçekliğin Eğitimde Kullanımı

Sanal gerçekliğin eğitimde kullanımı 1970'li yıllara dayanmaktadır. Bu dönemde pilot eğitimi için kullanılmaya başlanmıştır. Bu uygulama savaş pilotları için çok yararlı bir eğitim uygulaması alarak değerlendirilmiştir (46, 77). Bu başlangıç süreci ile SG uygulamaları diğer bir değişle sanal ortam eğitim alanında da aktif olarak kullanılmaya başlanmıştır. Sanal gerçeklik uygulamalarında öğrenci sahici bir ortamda birçok obje ya da objelerle etkileşim haline girmektedir. Öğrenciler bu etkileşim ile bulundukları ortamdaki nesneleri her açıdan inceleye bilmekte ve ortam içinde bulunabilmektedir. Bu olumlu durumlar sonucunda öğrencilerin SG alanında öğretilmek istenilen konuyu daha etkili ve daha fazla odaklanarak öğrendiği görülmüştür (45). Aynı zamanda SG alanı öğrenciye simüle edilmiş bir ortamda harekete geçmesini sağlayarak dersi anlamada güçlü bir ortam sağlamaktadır (45, 78). Öğrencilerin yapay olarak müfredatlarına yada eğitim aldıkları alana uygun oluşturulan sanal ortamlarda öğrenmenin oldukça yüksek olduğu görülmüştür (43, 79, 80). Sanal gerçeklik ortamı öğrencinin yada kullanıcının ortama entegre olmasını ve simüle edilmiş senaryolar ile ortamla etkileşim kurmasını sağlar (81, 82). Tuncer ve Taşpınar (83), sanal ortamdaki eğitim ve öğretimin geleceği ve sorunlarını inceledikleri makalelerinde, internetin eğitim ve öğretime katkı sağladığı, SG gibi platformların eğitimde etkili olduğu ve bilgisayar destekli online öğrenmenin öğrencilerin bilgi ve becerilerini bireysel ve bağımsız olarak kazanabileceklerini bildirmişlerdir. Tepe (84) başa takılı SG uygulaması kullanarak, yangın ve acil durumlar dersi için geliştirdiği ders materyalinin teori olan öğrencilere oranla daha yüksek öğrenme başarısı olduğunu saptamıştır. Oluşturduğu SG ders destek materyalinin etkin olduğu görülmüştür.

Eğitim alanında sanal gerçekliğin verimli kullanımı için bazı şartları sağlaması gerekmektedir. Bu şartlar;

- Gerçek hayatta o nesne ya da ortamın sağlanması güç veya imkansız olması,
- Uygulanan sanal gerçeklik ortamında gerçek nesnelerin olmaması gerekir.
  Aksi halde sanal ortam kullanıcı için güvensiz ve riskli hale gelebilir,
- Sanal gerçeklik uygulamasına aktarılacak olan materyalin gerçekte çok maliyetli olmasıdır (81, 82).

Sanal gerçeklik uygulamaları teknik ve ders eğitiminin yanı sıra engelli bireylerde kişisel ihtiyaçlarını karşılama, iletişim sağlama, fiziksel yeteneklerini güçlendirme gibi sosyal alan eğitimlerinde de aktif olarak kullanılmaktadır. Bu alanda ihtiyaç duyulan destek de SG uygulamalarından karşılanarak eğitim alan kişilerin motivasyonlarını ve bilişsel yeteneklerini arttırmaktadır (85–89).

Sanal gerçeklik uygulamalarının bir diğer örneği ve eğitim modeli de ülkemizde ve Fransa'da bulunan online ortamda müze gezme olanağıdır (90, 91). Bu sayede kişisel bulundukları ortamdan istedikleri müzenin sanal ortamına girerek müze ziyareti yapabilmekte ve sanal turizm olanağı kazanmaktadır.

Sağlık alanında da sanal gerçeklik uygulamalarının aktif kullanımı görülmektedir (92–94). Hastalara işlem sırasında uygulanan SG uygulamasının anksiyete, stres ve kaygıyı azalttığı görülmüştür (95, 96). Sezaryen ameliyatı öncesi anksiyeteyi azaltmak için SG ile simüle edilmiş hasta bilgilendirme eğitimleri de SG uygulamalarında dikkat çekmektedir (97). Eğitim alanının yanı sıra hasta güvenliği yada hasta bakımının iyileştirilmesinde de SG eğitimi uygulanmaktadır (98–101).

Çalışmalarda eğitimde SG uygulaması kullanımının, öğrenciler ya da kullanıcılar üzerinde olumlu etki bıraktığı, öğrenme yeteneklerini geliştirdiği ve öğrenme başarısını arttırdığı görülmüştür. Sanal gerçeklik uygulamaları eğitime farkı bakış açıları getirerek bireysel ve yaşam boyu öğrenmeye katkı sağlayacaktır. Öğrenmesi zor ya da uygulaması imkansız olan ortama SG simüle edilerek girilmesi dersin kalitesini, öğrencinin derse olan tutumunu ve ders motivasyonlarını arttıracaktır (45, 79, 84).

### 2.3.2. Sanal Gerçekliğin Ebelik Eğitiminde Kullanımı

Ebelik eğitiminde karma öğrenme metottu olan ve yaygın kullanılan yöntemler simülasyon tabanlı öğrenmedir. Simülasyon tabanlı eğitim, öğrenme eğitimindeki belirgin hedeflere ulaşmak için gerçek dünyaya ile aynı özelliklere benzemeye çalışan bir tekniktir (9, 102-104). Sağlık alanında simülasyon eğitiminin geçmişi 40'lı yıllara dayanmasına rağmen, 2000'li yıllarda spesifik olarak ebelik ve hemşirelik eğitiminin içine entegre edilmiştir (105, 106). Ebelik ve hemşirelik becerilerinin geliştirilmesi için önemli bir eğitim stratejisi olmuştur (102, 107). Simülasyon tabanlı öğrenme yönteminin, 2012 yılında Avustralya'da online platformda yapılan anket sonucunda, Avustralya ebelik müfredatından karma bir öğrenme yöntemi olarak kullanıldığı görülmüştür (9). Ebelik eğitiminde simülasyonun kullanımı öğrencilere teknik bilgilerin yanı sıra teknik olmayan ve klinik şartlarda görülme olasılığı düşük olan uygulamaları da deneyimle olanağı tanımaktadır (9, 102). Cooper ve ark.'ları (107) 2012 yılındaki sistematik derlemelerinde simüle edilmiş öğretim yöntemlerinin geleneksel yöntemlere oranla daha fazla öğrenme becerisi kattığı saptanmıştır. Simülasyon temelli eğitimin; senaryolar eşliğinde uygulama, dokunsal gerçeklik, bilgisayar destekli uygulamalar, mankenler kullanılarak simülasyon uygulamaları ve sanal gerçeklik uygulamaları olmak üzere birçok formu mevcuttur (7, 9, 103–105, 107).

Son yıllarda giderek artan, ebelik ve hemşirelik eğitiminde de kullanılan diğer bir simülasyon formu olan SG son on yıl içerisinde daha fazla tercih edilir ve kullanılabilir hale gelmiştir. Ebelik ve hemşirelik öğrencileri bu alanda bazı çalışmalarda birlikte ele alınırken bazı çalışmalarda da ayrı tutulmuştur (102, 109–112).

Sanal gerçeklik uygulamaları gerçeklik uygulamalarının ebelik eğitiminde kullanıldığı alanların sınırlı olduğu görülmüştür. Literatürde az sayıda çalışmaya rastlanmıştır (110, 113, 114).

Ebelikte SG uygulama alanları, gebelik alanında yeni tasarım aşamasında olan "gebelik yolu (road to birth)" projesi, sanal gerçeklik ortamında yenidoğan resüsitasyon uygulaması, üç boyutlu gözlük ile ebelik eğitimi, sanal doğum kliniği eğitimleri olarak görülmüştür (106, 114–118).

# 2.4. FETAL GELİŞİMİN ÖĞRETİMİNDE SANAL GERÇEKLİĞİN KULLANIMI

Fetal gelişimin öğretimi ebelik eğitiminde büyük önem taşımaktadır. Ebelik eğitiminde fetal gelişim, fizyoloji ve embriyoloji dersi müfredatından başlayıp, sağlıklı gebelik ve doğum, riskli gebelik ve doğum, yenidoğan ve çocuk sağlığı hastalıkları olmak üzere neredeyse tüm müfredatında yer almaktadır. Fetal gelişimin öğrenimi öğrencinin her dönemde faydalanacağı bilginin de öğrenimini etkilemektedir. Fetal gelişim öğretiminde arttırılmış gerçeklik uygulamalarının olduğu görülmüştür (118, 119). Literatür incelendiğinde İspanya'da aileler ve gebeler için arttırılmış gerçeklik ile oluşturulmuş fetal gelişim uygulamasının olduğu görülmüştür. Bu uygulama ebelik öğrencilerin değil sadece annelerin kullanabileceği bir uygulamadır. Uygulamada anne karnına bağlanabilen bir kemer üzerine konumlandırılmış arttırılmış gerçeklik ile çalışan hafta hafta fetal gelişim yer almaktadır. Anne karnına kemeri takıp haftasına uygun kartları yerleştirdiğinde bilgisayar ekranına bebeğin o hafta ile uyumlu görselleri gelmektedir. Ebelik öğrencilerinin eğitimi dışında olan bu uygulama, gebelerin ve yakınlarının fetal izlem ile ilgili bilgi gereksinimlerini karşıladığı görülmüştür (120). Fetal gelişimin öğretiminde literatür incelendiği çok az sayıda çalışmaya rastlanmıştır (114, 116). Fetal gelişimin öğretiminin gösterildiği var olan uygulama sadece sanal gerçeklik uygulaması değil aynı zamanda karma ve arttırılmış gerçeklik ile aplikasyon uygulamaların da olduğu görülmüştür (114, 118). İsmail'in, öğrencilerin, ergenlerin, yetişkinlerin ve annelerin fetal gelişimin öğretimi için geliştirildiği uygulamada, fetüsün hafta hafta gelişimi 3 boyutlu resimlerle görselleştirilmiştir. Uygulamanın etkin ve kullanılabilir olduğu görülmüştür (118). Literatüre ışık tutacak nitelikte hazırlanan bu araştırma hem literatürdeki boşluğu kapatacak hem de ebelik öğrencilerinin hafta hafta fetal gelişim öğretiminde yenilikçi bir uygulama olacaktır. Aynı zamanda elde edilen veriler ışığında diğer çalışmalara ışık tutacağı düşünülmektedir.

### 3. GEREÇ VE YÖNTEM

#### 3.1. ARAŞTIRMANIN AMACI

Bu araştırmada, sanal gerçeklik ortamında, fetal gelişim ve plasental gelişim için sanal gebeliğin tasarlanması ve tasarlanan "Sanal Gerçeklik Teknolojisi ile Oluşturulan Fetal Gelişim Uygulaması (SGT-FEGU)"nın ebelik eğitimi üzerine etkililiğinin değerlendirilmesi amaçlanmıştır.

### 3.2. ARAŞTIRMANI HİPOTEZLERİ

Sanal gerçeklik teknolojisi ile oluşturulan hafta hafta fetal gelişim Programı'nın uygulandığı deney/girişim grubunda yer alan ebelik öğrencilerin, kontrol grubunda yer alan öğrencilere göre;

Hipotez (H0): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının etkisi yoktur.

Hipotez (H1): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının etkisi vardır.

Hipotez (H0): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilere bilişsel yükü yoktur.

Hipotez (H1): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilere bilişsel yükü vardır.

Hipotez (H0): Fetal gelişimin öğretiminde SGT-FEGU uygulaması deneyiminde kontrol ve görsel ara yüzlerin etkisi yoktur.

Hipotez (H1): Fetal gelişimin öğretiminde SGT-FEGU uygulaması deneyiminde kontrol ve görsel ara yüzlerin etkisi vardır.

Hipotez (H0): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin görsel, işitsel ve dokunsal olarak algılamasına etkisi yoktur.

Hipotez (H1): Fetal Gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin görsel, işitsel ve dokunsal olarak algılamasına etkisi vardır.

Hipotez (H0): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin çevrelenmişlik duygusu ile sürekli bir deneyim ve uyaran akışı içerisine dahil edilip bunlarla etkileşim kurmasına etkisi yoktur.

Hipotez (H1): Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin çevrelenmişlik duygusu ile sürekli bir deneyim ve uyaran akışı içerisine dahil edilip bunlarla etkileşim kurmasına etkisi vardır.

### 3.3. ARAŞTIRMANIN ŞEKLİ

Bu araştırma ön-test son-test ölçümlü, izlemsel, randomize kontrollü bir çalışmadır.

### 3.4. ARAŞTIRMANIN DEĞİŞKENLERİ

Araştırmanın bağımlı değişkenini eğitim sonrası öğrencilerin FEGBÖ son test puanlarında değişiklik olma durumu oluşturmuştur.

Araştırmanın bağımsız değişkenleri; araştırmaya dahile dilen öğrencilerin sosyodemografik özellikleri, Bilişsel Yük Ölçeği (BYÖ) ve Bulunuşluk Hissi Ölçeği (BHÖ) alt boyut puanları.

### 3.5. ARAŞTIRMANIN YERİ VE ZAMANI

Araştırma Kasım 2019- Haziran 2021 tarihleri arasında gerçekleştirildi. Etik kurul aşaması Aralık 2019- Haziran 2020, Bilimsel Araştırma Projeleri Koordinatörlüğü (BAP) proje onay işlemleri aşaması Haziran 2020- Aralık 2020, Sanal gerçeklik teknolojisi ile hafta hafta fetal gelişimi oluşturma aşaması Aralık 2020- Mart 2021 tarihleri arasında gerçekleştirilmiştir. Araştırmanın veri toplama aşaması Nisan 2021- Mayıs 2021 tarihleri arasında Karabük Üniversitesi Sağlık Bilimleri Fakültesi Ebelik Bölümünde gerçekleştirildi.

### 3.6. ARAŞTIRMANIN EVREN VE ÖRNEKLEMİ

Araştırmanın evrenini; Karabük Üniversitesi Sağlık Bilimleri Fakültesi, Ebelik Bölümünde 2019-2020 eğitim öğretim yılında okuyan 404 öğrenci oluşturmuştur.

Araştırmanın örneklemini; dördüncü sınıf ders uygulaması kapsamında Karabük Üniversitesi Ebelik Bölümü laboratuvarına gelen çalışmaya katılmayı kabul eden 118 öğrenciden uygunluk kriterlerini sağlayan 84 öğrenci oluşturdu.

Araştırmanın örneklem büyüklüğünü belirlemek için güç analizi program olan G-Power 3.1.9.2 programı kullanıldı. Araştırmanın veri tipinde kategorik değişkenlerin bulunması, deney ve kontrol olmak üzere iki farklı örneklem grubunun olması nedeniyle güç analizinde kullanılacak test Independent t testi olarak belirlendi.

Araştırmada, gerçekte olmayan bir etki, fark ya da ilişkiyi varmış gibi bulabilme ihtimalini ifade eden, yalancı pozitiflik olarak da bilinen ve genellikle α hatası olarak adlandırılan I. tip hata düzeyi %5 olarak kabul edildi. Diğer taraftan gerçekte olan bir etki, fark ya da ilişkiyi araştırma sonuçlarında yokmuş gibi gösterme ihtimali olarak ifade edilen, yalancı negatiflik olarak bilinen ve genellikle ß hatası olarak adlandırılan II. tip hata düzeyi %5 olarak kabul edildi. Bu durumda bu araştırma %95 güç ile gerçekleştirildi. Araştırmada gruplara dağılım oranı, yani her bir grupta yer alacak olan örneklemlerin sayısının birbirine oranının bir (1) olacağı ve araştırma hipotezinin de çift taraflı hipotez olduğu durumu göz önüne alınarak güç analizi gerçekleştirildi. %95 güven (1-α), %95 test gücü (1-β), d=0.80 (large-büyük) etki büyüklüğü dikkate alındığında her bir grupta 42 vaka olmak üzere toplamda 84 vaka alınması gerektiği belirlendi (165) (Şekil 3.1, Tablo 3.1). Gruplar arasındaki gerçek farkın daha iyi saptanması için %95 güven aralığı alındı ve araştırmaya her grup için 42 olmak üzere 84 öğrenci alındı. Araştırma deney ve kontrol olmak üzere iki grupta gerçekleştirilmiştir. Sanal gerçeklik ortamında hafta hafta fetal gelişim eğitimini alan grup deney grubunu, yüksek öğretim ebelik çekirdek müfredatı içeriğine uygun olarak hazırlanan müfredat kapsamında anlatılan fetal gelişim teori eğitimini alan grup kontrol grubunu oluşturdu.



Şekil 3.1: G-power analiz sonucu

Tablo 3.1: G-powers analizi sonuç protokolü

| t tests - Means: Difference between two independent means (two groups) | | |
|---|---|---|
| Analysis: | A priori: Compute required sample s | size |
| Input: | Tail(s): Two | |
| | Effect size d | = 0.80 |
| | α err prob | = 0.05 |
| | Power (1-β err prob) | = 0.95 |
| | Allocation ratio N2/N1 | = 1 |
| Output: | Noncentrality parameter $\delta$ | = 3,6660606 |
| | Critical t | = 1,9893186 |
| | Df | = 82 |
| | Sample size group 1 | = 42 |
| | Sample size group 2 | = 42 |
| | Total sample size | = 84 |
| | Actual power | = 0.9518269 |

Araştırmaya dahil edilme kriterleri;

- Karabük Üniversitesi Ebelik Bölümü 4. Sınıf öğrencisi olmak,
- Araştırmaya katılmaya gönüllü olmak

Araştırmaya dahil edilmeme kriterleri;

- Birinci, ikinci ve üçüncü sınıf öğrencisi olmak.
- Araştırmaya katılmaya gönüllü olmamak.

### 3.6.1. Randomizasyon

Araştırmaya dahil edilme kriterleri belirlendikten sonra öğrenciler basit rastgele randomizasyon yöntemiyle deney ve kontrol gruplarına ayrıldı. Basit randomizasyonda rastgele sayılar üreten bir program (random.org) kullanıldı (121). Bu randomizasyon programı sayesinde öğrencilerin sırasıyla hangi gruba dahil edileceği sayıların gruplara dağılımı belirlendi (grup 1 (deney) ve grup 2 (kontrol)). Örnekleme ait basit rastgele randomizasyon sayıları Tablo 3.2'de verilmiştir. Randomizasyon sonrası grupların hangisinin deney hangisinin kontrol olduğunu saptamak için kura çekme yöntemi kullanıldı. Kura sonrası grupların dağılımı tablo 3.3'te verilmiştir.

**Tablo 3.2:** Randomizasyon ile belirlenen deney ve kontrol grupları

| GRUPLAR | |
|---|---|
| Deney Grubu (Grup 1) | Kontrol Grubu (Grup 2) |
| 21, 64, 11, 32, 78, 49, 74, 47, 14, 29, 5, 44, 8, 15, 69, 66, 60, 77, 70, 54, 84, 76, 18, 41, 25, 59, 51, 65, 82, 4, 30, 42, 63, 17, 26, 52, 67, 3, 28, 22, 80, 81 | 75, 71, 43, 36, 45, 20, 50, 58, 57, 38, 16, 79, 83, 23, 24, 7, 2, 61, 56, 33, 31, 1, 55, 13, 19, 48, 34, 53, 39, 27, 46, 73, 72, 68, 35, 37, 10, 40, 62,6, 12, 9 |

**Tablo 3.3:** Örnekleme ait grupların atanması

| Grup adı | Grupların İçeriği |
|----------|-------------------------------------------------|
| Grup 1 | Sanal gerçeklik uygulaması kullanan deney grubu |
| Grup 2 | Müfredata uygun teori alan Kontrol grubu |

Araştırma verilerinin toplanma sürecinde uygunluk için 118 öğrencinin 34'ü çalışmanın uygulama kısmına pandemi sürecindeki ulaşım nedenlerinden, birkaç öğrencinin de COVİD-19 pozitif ya da temaslı olmasından dolayı çalışmaya dahil edilmemiştir. Araştırmanın veri toplama süreci deney grubunda 42 kontrol grubunda da 42 öğrenciye ulaşılmasıyla sonlandırılmıştır. Araştırmaya ait CONSORT (Consolidated Standarts of Reporting Trials) akış diyagramı Şekil 3.2 de yer almaktadır.

Araştırma uluslararası alanda tanınır ve tüm dünya literatüründe geçerli kılmak amacıyla Uluslararası Klinik Araştırmalar Kayıt Platformu'nda (International Clinical Trials Registry Platform) 2020/263 ID ve NCT04444258 ID numarasıyla kayıt altına alındı. Bunun yanı sıra araştırmanın yayınlanması aşamasında bazı dergiler tarafından talep edildiği için World Health Organization (WHO) internet sitesi üzerinden The Universal Trial Number (UTN) is U1111-1246-0530 alındı.



Şekil 3.2: Araştırma akış diyagramı (CONSORT 2010)
#### 3.7. VERİ TOPLAMA ARAÇLARI VE GEREÇLERİ

#### 3.7.1. Veri Toplama Araçları

Araştırmada,

- 1. Kişisel Bilgi Formu (Ek:1)
- 2. Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ) (Ek: 2)
- 3. Bilişsel Yük Ölçeği (BYÖ) (Ek:3)
- 4. Bulunuşluk Hissi Ölçeği (BHÖ) (Ek:4) veri toplamada kullanıldı.

Veri toplama araçlarından Kişisel Bilgi Formu ile Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ) her iki gruba ön test ve son test takipleri boyunca üniversitenin lisansının olduğu platform olan Microsoft Teams programı aracılığı ile doldurulmuştur. Bilişsel Yük Ölçeği (BYÖ) ve Bulunuşluk Hissi Ölçeği (BHÖ) sanal gerçeklik gözlüğünü deneyimleyen deney grubuna uygulama sonrası yüz yüze görüşme yöntemi ile dolduruldu.

- **3.7.1.1. Kişisel bilgi formu (EK 1):** Bu form araştırmaya katılan öğrencilerin sosyodemografik özellikleri, bölüm tercihi ile ilgili bilgileri ve daha önce sanal gerçeklik uygulamasını deneyimleme durumlarını içeren 14 soruyu oluşmuştur.
- 3.7.1.2. Fetal gelişimi değerlendirme bilgi ölçeği (FEGBÖ) (EK: 2): Öğrencilerin fetal gelişimi değerlendirme bilgilerini ölçen literatürde bir ölçüm aracına rastlanmamıştır. Öğrencilerin fetal gelişimlerini değerlendirmek için araştırmacılar tarafından Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ) geliştirilmiştir. Ölçeğin geliştirilmesi tez sürecinden bağımsız olarak devam etmiş ve ayrı bir etik kurul onayı alınmıştır (Sağlık Bilimleri Üniversitesi, Hamidiye Bilimsel Araştırmalar Etik Kurulu, Tarih: 12.03.2021 Karar No: 18875) (EK: 5). Ölçeğin geliştirilmesi sürecinde ölçek geliştirme basamaklarından geçmiştir. On dört uzman görüşü alınmıştır. Uzman görüşü sonrasında 410 öğrenciye uygulanmıştır. Açımlayıcı Faktör Analizi (AFA) ve Doğrulayıcı Faktör Analizi (DFA) sonrasında 23 maddelik tek alt boyuttan oluşan ölçek oluşturulmuştur. Ölçeğin güvenilirlik kat sayısının (Cronbach Alpha) 0,89, Kaiser-Meyer-Olkin (KMO) katsayısının 0,927 ve Bartlett Küresellik Testinin ise anlamlı olduğu belirlenmiştir (χ2(253) =2648,074 p= 0,000). Analizler sonucunda Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ)'nin Türkiye'de lisans ebelik öğrencileri için geçerli ve güvenilir bir ölçme aracı olduğu ve çalışmalarda kullanılabileceği saptanmıştır.

Geçerlik güvenilirliği yapılan ölçek araştırmada ön test ve son test olarak deney ve kontrol grubu olmak üzere tüm gruplara uygulanmıştır. Ön test her iki gruba randomizasyon yapıldıktan sonra ve uygulamaya başlamadan önce Google formlar aracılığıyla online ortamda tüm öğrencilere uygulanmıştır. Son test olarak da 6 hafta sonra online olarak her iki gruba da uygulanmıştır.

3.7.1.3. Bilişsel yük ölçeği (BYÖ) (EK:3): Ölçek, Paas ve Van Merrienboer (1993) tarafından geliştirilmiştir (122). Ölçeğin Türkçe 'ye uyarlanması Kılıç ve Karadeniz tarafından (2004) yapılmıştır (123). Ölçek tek maddeden oluşmakta ve ölçekte 9'lu derecelendirme kullanılmaktadır. Ölçekten alınabilecek en yüksek puan 9, en düşük puan ise 1'dir. Ölçeğin puanlanmasında orta nokta 5'tir. 5'in altındaki puanlar öğrencinin bilişsel olarak aşırı yüklenmediğini, 5'in üstündeki puanlar ise aşırı yüklendiğini göstermektedir. Tek maddeden oluşan ölçek, bir görev/ işi yapan öğrenenlerin bu görev ya da işi yaparken harcadıkları çabayı ölçmektedir. Ölçek deney grubundaki öğrencilere sanal gerçeklik gözlüğünü deneyimledikten sonra uygulandı.

3.7.1.4. Bulunuşluk hissi ölçeği (BHÖ) (EK: 4): Ölçek Witmer, Jerome ve Singer tarafından, davranışsal ve sosyal ordu araştırma enstitüsü simülatör sistemleri araştırma birimindeki öğrencilerin, sürükleyici sanal ortamlara maruz kaldıktan sonra katılımcıların Bulunuşluk hislerini saptamak amacıyla 2005 yılında geliştirilmiştir (124). Ölçeğin Türkçe geçerlik güvenilirliği Gökoğlu ve arkadaşları tarafından 2018'de yapılmıştır (125). Orijinali 7 likert tipte olan ölçek Türkçe geçerliliğinde 5'li likert tipte indirgenmiştir. Ölçeğin orijinalindeki Cronbach's Alpha güvenirlik katsayısı 0,91, Türkçe uyarlama çalışmasında ise 0.844 olarak bulunmuştur. Ölçek sanal gerçeklik temelli öğrenme ortamlarında bulunuşluk hissini ölçmektedir. Ölçeğin, Katılım (Faktör 1), Uyum/Çevreleme (Faktör 2), Duyusal Bağlılık (Faktör 3), Etkileşim (Faktör 4) ve Ara yüz Kalitesi (Faktör 5) olmak üzere 5 faktörü (alt boyu) vardır ve 29 sorudan oluşmaktadır (EK 4).

#### 3.7.2. Veri Toplama Gereçleri

**3.7.2.1.** Oculus rift quest 2 sanal gerçeklik gözlüğü: Donanım özellikleri Oculus Rift Quest 2 (Güncel Sürümü) olarak geliştirilmiş ikinci nesil sanal gerçeklik gözlüğüdür. Bilgisayar destekli ve bağımsız olmak üzere iki özelliği ile oculus işletim sistemine sahiptir. Bunlardan birkaçı; bağımsız bir işletim sistemi ve işlemciye sahip olması, hızlı

bir işlemci ve en yüksek çözünürlüklü ekranı ile her hareketin hızlı olmasını sağlaması, göz başına 1832 x 1920, piksel toplam 3664x1920 piksel çözünürlüğe sahip olması, ekran yenileme hızının 90 Hz. **ve** iki adet kollarının olmasıdır.



Şekil 3.3: Oculups rift quest 2 sanal gerçeklik gözlüğü

İşletim sistemine içeriği ve görselleri araştırmacı tarafından oluşturulan "Hafta hafta fetal gelişim" ile her hafta fetüsün boy, kilo ve gelişim özelliklerinin değiştiği "Hologramik saat" entegre edildi.

Hizmet alımı yapılan firma tarafından, araştırmacıların hazırladığı özellikleri kapsayan "Fetal Gelişim" formatı sanal gerçeklik gözlüğüne entegre edildi. Yazılım ve görselleştirmelerinin yapılmasının ardından SGT-FEGU deney grubundaki öğrencilere uygulandı.

Sanal gerçeklik ortamında oluşturulan SGT-FEGU'nun detayları "Araştırma Hazırlık Aşamasında ele alındı.

### 3.8. ARAŞTIRMANIN AŞAMALARI

Araştırma "Hazırlık", "Uygulama" ve "İzlem" olmak üzere üç aşamada gerçekleştirildi (Tablo 3.4).

**Tablo 3.4:** Araştırmanın uygulama ve veri toplama aşamaları

| | Deney Grubu | Kontrol Grubu |
|---|---|---|
| Hazırlık Aşaması | Deney grubuna uygulanacak olan hafta hafta fetal gelişimin geliştirilmesi için; • Veri toplama araç ve gereçlerinin hazırlanması, • Hafta hafta fetal gelişimin oluşturulması, • Oluşturulan SGT-FEGU uygulamasının incelenmesi, • SGT-FEGU uygulamasının sanal gerçeklik ortamına aktarılması, • Sanal gerçeklik ortamına aktarılan uygulamanın son şeklinin verilmesi. | Kontrol grubuna verilecek teori eğitimi için; • Literatür doğrultusunda, Ebelik çekirdek müfredatı ve ebelik bölüm müfredatı doğrultusunda hafta hafta fetal gelişimi anlatan sunum hazırlanması. |
| | Araştırmanın Ran | domizasyonu |
| Ön test | Deney ve kontrol gruplarınd<br>Her iki gruba da; • Kişisel bilgi formu • Fetal gelişimi Değerlendirme Bilgi Ölçeğ | |
| Uygulama<br>Aşaması | Sanal gerçeklik ortamında geliştirilen hafta hafta fetal gelişimin uygulanması | Müfredat doğrultusunda oluşturulan Fetal gelişim teori eğitimin uygulanması |
| Son Test Uygulama Sonrası | Sanal gerçeklik uygulamasından hemen sonra; Bilişsel Yük Ölçeğinin (BYÖ), Bulunuşluk Hissi Ölçeği (BHÖ) | Uygulama sonrası herhangi bir ölçek uygulanmadı. |
| Son Test | Sanal gerçeklik eğitiminden 6 hafta sonra, • Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ) uygulandı. | Teori eğitiminden 6 hafta sonra, • Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ) uygulandı. |
| Son Test<br>Sonrası | Deney grubu için araştırma tamamlandı. | Araştırmanın son test uygulanması<br>bittikten sonra Kontrol grubundaki<br>öğrencilere Sanal gerçeklik ortamında<br>hazırlanan SGT-FEGU uygulandı. |

#### 3.8.1. Araştırmanın Hazırlık Aşaması

Sanal gerçeklik teknolojisi ile oluşturulmuş fetal gelişim uygulaması (SGT-FEGU)'nun oluşturulması tümüyle bu aşamada yapıldı. Geliştirilen SGT-FEGU'nun işlem basamakları ve hazırlık aşaması adım adım aşağıdaki maddelerde anlatıldı (Şekil 3.4).

- 1. Sanal gerçeklik teknolojisi ile hazırlanan fetal gelişim eğitim programında hafta hafta fetal gelişim aşamaları (boy, kilo ve fetal oluşumlar) literatür doğrultusunda yazıldı ve oluşturuldu (2, 29) (Ek: 6)
- SGT-FEGU'nun görselleri literatür doğrultusunda hazırlandı, hizmet alımı yapılacak firmaya gönderildi, firma tarafından teze özel modellendi (2, 29, 124). Modelleme işlemi yapıldıktan sonra tüm görseller tek tek incelendi ve son hali verildi.
- 3. Görselleştirme işlemi tamamlandıktan sonra literatür doğrultusunda hazırlanan fetal gelişimin haftaları, fetüsün boy ve kilo gelişimi ile her haftadaki gelişimini içeren bilgiler hologramik görsel bir saate aktarıldı.
- 4. Uygulamanın son güncellemeleri bittikten sonra beş akademisyenden uzman görüşü alındı. Uzmanlar, 1 Profesör, 1 Doçent, 2 Araştırma Görevlisi ve 1 Öğretim Görevlisinden oluşmuştur.
- 5. Uygulama oluştuktan sonra ön test için kişisel bilgi formu ve FEGBÖ online ortamda oluşturuldu.
- 6. Araştırma için uygunluk kriterlerini karşılayan öğrenciler arasında randomizasyon yapıldı deney ve kontrol grubu oluşturuldu.



Şekil 3.4: Araştırmanın hazırlık aşaması algoritması

#### 3.8.1.1. Sanal gerçeklik teknolojisi ile fetal gelişim uygulamasının geliştirilmesi:

Sanal gerçeklik teknolojisi ile oluşturulan hafta hafta fetal gelişim eğitim programının (SGT-FEGU) geliştirilmesi araştırmanın temelini oluşturdu. Bu aşamada araştırmacılar tarafından literatür doğrultusunda hafta hafta fetal gelişim yazıldı (EK 6). Oluşturulan SGT-FEGU'nun içeriği 6. gebelik haftasından başlayarak (embriyonel dönemin son iki haftası ile fetal gelişim dönemin başlangıcı) 40. gebelik haftası ile sonlandırıldı. Oluşturulan bu içerikte; fetal hafta, fetüsün boy ve kilosu, haftalardaki gelişimsel süreç anlatılmıştır. Oluşturulan sanal gerçeklik ortamında aynı zamanda fetüsün 6. gebelik haftasından sonra abdominal ultrasonografi ile duyulan fetal kalp atımları (FKA) ses olarak eklendi. FKA gebelik haftasına göre 120-160 atım/dakika arasında değişmektedir (2, 29, 124, 125). Uygulamada da FKA haftalara uygun olarak yerleştirildi. Uygulamanın fetal gelişim görselleri literatür referans alınarak hazırlandı ve hafta hafta tanımlandı (1–4, 29). Aynı zamanda görseller için ücretli uygulamalardan da referans alındı. Referans alınan görseller EK 7'de sunuldu. Referans verilen görseller doğrultusunda araştırmaya özgü modellemeler yapıldı. Modellemeler hizmet alımı ile bütçelendirildi.

Uygulamanın sağ kontroller (sağ kol) kısmına hologramik saat eklendi. Bu saatte fetüsün; boy, kilo ve gelişim süreçleri yer aldı. Hologramik saate, uyulmanın tamamı bittikten sonra (fetüs 40. Gebelik haftasına geldiğinde) fetüsün gelişimini hafta hafta geriye döndürmek için üst ve alt ok ile uygulamayı baştan izlemek için yuvarlak bir ok yerleştirildi. Bu hologramik saat uygulamayı kullanan kişinin interaktif bir şekilde tıklaması, uygulamaya aktif katılım sağlanması ve istediği haftayı izlemesi için oluşturuldu (EK 8).

Uygulamadaki modellemeler hizmet alımı yapılan firma ile toplantılar yapılarak güncellendi ve araştırmadaki uygulanabilir son halini oluşturuldu. Oluşturulan SGT-FEGU Ebelik öğretim üyesi (Profesör ve Doçent), Ebelik (Araştırma Görevlisi ve Öğretim Görevlisi) ile Hemşirelik alanındaki bir öğretim elemanı olmak üzere beş uzman görüşüne sunulmuş ve deneyimlenmiştir. Uzmanlardan uygulama ile ilgili geri bildirim alınmış ve uygulamanın son şekli verilmiştir. Uygulama üç buçuk dakika süren ve Araştırma için geliştirilmiş özgün bir uygulamadır.

3.8.1.2. Ebelik çekirdek müfredatı doğrultusunda fetal gelişim teori eğitiminin oluşturulması: Fetal gelişim ebelik müfredatında Normal Gebelik/ Doğum Bilgisi I/ Doğum Öncesi Dönem derslerinin 14 haftalık içeriğinde 4 ya da 8 saat olarak, fetal sağlığın değerlendirilmesi, gebeliğin fizyolojisi ya da fetal gelişim şeklinde verilmektedir. İçerik ve program yeterlilikleri benzer olmasına rağmen isimler kurumsal farklılıklar gösterebilir (128–131). Kontrol grubu için rutin müfredat doğrultusunda hazırlanan fetal gelişim teori eğitimi; hafta hafta fetal gelişim ve oluşum ile fetüsün hafta hafta boy, kilo ve görselleri yer almaktadır (1–4, 130, 131). Fetal gelişim teori eğitim içeriği 55 slayttan oluşmuştur. Sunum içeriği EK 9'da verilmiştir.

#### 3.8.2. Araştırmanın Uygulama Aşaması

Hazırlanan sanal gerçeklik uygulaması ve teori eğitim materyalinden sonra araştırma uygunluk kriterlerini karşılayan öğrenciler arasından Deney (Grup 1= 42) ve Kontrol (Grup 2= 42) grubu ataması yapılmış ve uygulama aşamasına geçilmiştir (Şekil 3.4). Araştırmanın bu aşamasında bu aşamasına randomizasyonu yapılan deney ve kontrol grubundan onam alınmıştır (Ek 10).

- **3.8.2.1. Deney grubu için veri toplama süreci:** Bilgilendirilmiş onam formu alanına deney grubunun uygulama akışı aşağıdaki sıra ile gerçekleştirilmiştir (Şekil 3.5).
  - Deney grubundaki öğrencilere üniversitenin lisansının olduğu platform olan Microsoft Teams programında kişisel bilgi formu ve FEGBÖ ön test olarak uygulandı.
  - Ön test uygulandıktan sonra deney grubu farklı saatlerde SGT-FEGU için Karabük Üniversitesi, Sağlık Bilimleri Fakültesi, Ebelik Bölümü laboratuvarına çağırıldı.
  - 3. Öğrenciler SGT-FEGU için teker teker uygulama alanına alındı ve her öğrenciye uygulama tanıtıldı.
  - 4. Bilgilendirme sonrası sanal gerçeklik gözlüğü takılmıştır. Öğrencilere fetal gelişimi 6. haftadan 40. haftaya kadar izletildi. Uygulama 40. Gebelik haftasına ulaştıktan sonra öğrencilere hologramik saat ile hafta hafta geri giderek ya da tekrar baştan başlayarak her bir haftanın içeriğini adım adım tekrar izlenmesi sağlandı. Gözlük için her bir öğrenciye 25 dakika verildi. Aynı zamanda öğrencilere kendileri bırakmak istediklerinde gözlüğü çıkarıp sanal ortamdan

- ayrılma özerkliği de sunuldu. Her bir öğrencinin uygulamada kalma süresi 20-25 dakika arasında değiştir. Uygulama fotoğrafları Şekil 3.6 da verilmiştir.
- 5. Her bir öğrenciye uygulama yapıldıktan sonra sanal gerçeklik gözlüğü yüzey ve kumaşlar için uygun olan hijyenik sprey ile temizlendi. Uygulamalar arasında laboratuvar havalandırıldı ve 20 dakika aralıklar ile uygulama yapıldı.
- 6. Uygulama sonrası deney grubundaki öğrencilere BYÖ ve BHÖ uygulandı. Aynı zamanda deneyimlediği SGT-FEGU için kalitatif geri bildirim alındı. Uygulama sonrası deney grubun uygulama aşaması bitirildikten sonra izlem aşamasına geçildi.
- **3.8.2.2.** Kontrol grubu için veri toplama süreci: Kontrol grubuna verilecek eğitim öncesi araştırmacı online İstanbul İşletme Enstitüsü'nden 5 gün 10 saatlik Eğitici Eğitimi sertifikası almıştır (EK 11). Bilgilendirilmiş onam formu alanına kontrol grubunun uygulama akışı aşağıdaki sıra ile gerçekleştirildi.
  - Kontrol grubundaki öğrencilere üniversitenin lisansının olduğu platform olan Microsoft Teams programında online ortamda kişisel bilgi formu ve FEGBÖ ön test olarak uygulandı.
  - 2. Ön testi uygulana öğrenciler için Microsoft Teams'de bir sınıf oluşturuldu ve teori eğitimi için öğrenciler tek tek gruba eklendi,
  - 3. Kontrol grubundaki öğrencilere 55 slayttan oluşan hafta hafta fetal gelişimi anlatan, ebelik müfredatına uygun içerik ile hazırlandı ve 2 saat süren teori eğitimi yapıldı.
  - 4. Teori eğimi sonrası kontrol grubun uygulama aşaması bitirildi ve izlem aşamasına geçildi.



Şekil 3.5: Araştırmanın uygulama aşaması- algoritma



Şekil 3.6: Sanal gerçeklik uygulama anı fotoğrafları

#### 3.8.3. Araştırmanın İzlem Aşaması

Oluşturulan SGT-FEGU'nun ve ebelik çekirdek müfredatına uygun hazırlanan teori eğitiminin izlemleri bu aşamada yapıldı (Şekil 3.6). İzlem aşamasında deney ve kontrol grubuna yapılan uygulama aşağıda listelenmiştir.

- 1. Deney ve Kontrol grubuna 6 hafta sonra son test uygulandı.
- 2. Her iki gruba da son test olarak FEGBÖ uygulandı.

Deney ve Kontrol grubuna son test uygulandıktan sonra araştırma sonlandırılmıştır. Kontrol grubundaki tüm öğrencilere araştırma sonunda SGT-FEGU izletildi.



**Şekil 3.7:** Araştırmanın izlem aşaması

#### 3.9. VERİLERİN ANALİZİ

Araştırmadan elde edilen veriler, SPSS for Windows (versiyon 20.0, Statistical Package for Social Sciences) programı ile analiz edildi. Araştırmada kullanılan ölçekler için iç tutarlılık Cronbach's Alfa güvenilirlik katsayısı ile değerlendirildi. Verilerin dağılımı Skewness / Kurtosis (Basıklık/ Çarpıklık) değerlerine göre incelenmiş ve normal dağılıma uygun olduğu saptanmıştır (134). Araştırmadaki sürekli değişkenlere ait istatistikler ortalama, standart sapma, minimum ve maksimum değerler ile gösterilmiştir. Kategorik değişkenlere ait tanımlayıcı istatistikler frekans ve yüzde ile incelenmiştir. Bağımsız grupların karşılaştırılmasında Bağımsız iki örneklem T testi (Independent Sample T testi) kullanılmıştır. Gruplar arasındaki farkın tanımlanmasın poet hoc analiz de Bonferroni testi uygulanmıştır. Bağımlı örneklemlerin ön test- son test karşılaştırılmasında Eşli İki Örnek T testi (Paired Smaple T test) kullanılmıştır. Grupların son test puan karşılaştırılmasında ön testin etkisini ayırmak için Kovaryans Analizi yapıldı. Gruplar üzerine etki eden parametreler Binary Lojistik regresyon modeliyle açıklanmıştır. Ölçekler arası ilişkiyi saptamak için Pearson korelasyon yapılmıştır. Araştırmada anlamlılık düzeyi için p değeri 0,05'ten küçük olarak alındı. Bonferroni poc toc analizi için p değeri 0,01'in altı alındı. Verilerin istatistiksel analizi Tablo 3.5'te verilmiştir.

**Tablo 3.5:** Veri analiz parametre ve istatistik yöntemleri

| İstatistik Uygulamasın Yapıldığı Parametreler | Kullanılan İstatistik Vöntami |
|---|---|
| | Kunaman Istatistik Tontenn |
| Ölçeklerin ve alt boyutlarının güvenilirliği/ iç<br>tutarlılığı | Cronbach' Alfa güvenilirlik kat sayısı |
| Grupların kategorik bakımdan homojenliği | Pearson Ki-kare testi |
| Normallik dağılıma uygunluk, | Skewness / Kurtosis (Basıklık/ Çarpıklık) değerleri |
| Tanımlayıcı istatistikler; | |
| <ul> <li>Sürekli değişkenler için</li> </ul> | Ortalama ve standart sapma |
| <ul> <li>Sayılabilen nitel değişkenler için</li> </ul> | • Sayı ve yüzde |
| Deney ve Kontrol grubunun ön test ve son test puan ölçümleri | Paried Sample T testi (eşit iki örneklem T testi/<br>İki zamanlı ölçümler için) |
| | <ul> <li>Kovaryans Analizi (Ancova Testi)</li> </ul> |
| Deney ve Kontrol grubunun kendi içindeki ön | Independent Sample T testi (Bağımsız Örneklem T |
| test ve son test puanları | testi) |
| <ul> <li>Deney ve Kontrol Gruplarının</li> </ul> | Binary Regresyon Analizi |
| tanımlayıcı istatistikler ile FEGBÖ ön | |
| test ve son test puanları üzerine etkisi, | |
| <ul> <li>Deney grubundaki öğrencilerin sanal</li> </ul> | |
| gerçeklik ve bilgisayar kullanımın | |
| BHÖ üzerine etkisi | |
| Deney grubundaki öğrencilerin BYÖ ve BHÖ arasındaki ilişki | Pearson Korelasyon |

### 3.10. ARAŞTIRMANIN SINIRLILIKLAR VE TAMAMLANMA SÜRECİNDE KARŞILAŞILAN DURUMLAR

Araştırma sürecinde karşılaşılan durumlar olumlu ve olumsuz olmak üzere iki aşamada ele alınmıştır.

#### Olumlu Durumlar;

- Öğrencilerin araştırmaya katılmada gönüllü olması,
- Araştırıma sürecinde uygulama yapılacak öğrencilerin COVID-19 pandemi döneminde olmasına rağmen uygulamasını tamamlamak için araştırmanın yapıldığı kurum olan Karabük Üniversitesinde bulunuyor olmaları,
- Hizmet alımı yapılan firmanın online platforma uygulama basamaklarını aksatmadan sürdürmeleri ve toplantılara devam etmeleri olumlu durum olarak ele alındı.

#### Olumsuz Durumlar;

- Araştırma veri toplama aşamasına başlamadan önce pandemi nedeniyle etik kurul izinlerinin 6 ay sonra çıkması. Benzer şekilde BAP'ın da pandemi süreci nedeniyle 6 ay değerlendirme aşamasında kalması ve bu süreçlerin araştırmaya 12 ay zaman kaybı yaşatması,
- COVID-19 pandemisi nedeniyle bazı öğrencilerin araştırmaya katılmak için seyahat edememeleri,
- Öğrencilerden birkaçının COVID-19 pozitif ya da temaslı olması olumsuz durum olarak ele alındı.

#### Araştırmanın Sınırlılıkları;

- COVID-19 nedeniyle uygulama yapılacak alanda kişi sınırlamasına gidildiğinden uygulamayı yapan ve anket uygulayan kişinin aynı araştırmacı olması,
- Araştırmanın sadece araştırmaya katılan öğrenciler ile sınırlı olmasıdır.

#### 3.11. ARAŞTIRMA SÜRECİNDE ALINAN COVİD-19 TEDBİRLERİ

Araştırma süreci 11 Mart 2019'da ilen edilen COVİD-19 pandemisinden etkilenmiştir. Süreçten etik kurul izinleri ve BAP proje başvurularının yanı sıra araştırmanın uygulama aşaması da etki altında kalmıştır. Araştırmanın uygulama aşamasındaki COVİD-19 tedbirleri aşağıdaki sırasıyla yer almaktadır;

- 1. Araştırma öncesinde YÖK tarafından aşılama kapsamına alınan öğrencilerin COVID-19 aşı yaptırma durumları kontrol edildi. Tüm öğrencilerin aşılarının iki dozunu da tamamlanması beklendikten sonra uygulamaya başlandı.
- 2. Aşı olmayan öğrencilerin klinik uygulamaya ve ikamet edecekleri yurtlara gelmeden önce yaptırdıkları COVİD-19 testleri kontrol edildi.
- 3. Uygulama yapılacak laboratuvar ortamı öğrenciler gelmeden önce havalandırılmıştır,
- 4. Uygulamaya alınacak öğrenciler teker teker laboratuvara alındı.
- 5. Uygulamaya katılan öğrencilerin ve uygulamayı yapan araştırmacının çift maske takması sağlandı.
- 6. Uygulamanın öğrencilere sosyal mesafe kurallarına uygun şekilde anlatılmış ve bireysel olarak gözlüğü takmaları sağlandı.

- 7. Her öğrenciye sanal gerçeklik gözlüğü, uygulama sonrası COVID-19 enfeksiyonu sürecine özel hazırlanan, 90° alkol içeriğine sahip yüzey ve kumaşlar için uygun sprey ile temizlendi.
- 8. Her öğrenci uygulama sonrası laboratuvar ortamı 15 dakika havalandırıldı.
- 9. Uygulama sürecinde ve sonrasında COVID-19 enfeksiyonu hiçbir öğrencide ve araştırmacıda görülmedi.

#### 3.12. ARAŞTIRMANIN YASAL VE ETİK BOYUTU

Araştırmanın yürütülmesinde;

- 1. Etik kurul izni Karabük Üniversitesi Klinik Araştırmalar Etik Kurulu'ndan (09.06.2020 tarihli, 2020/263 sayılı kara numarası) alındı (EK 12). Araştırma süresince İnsan Hakları Helsinki Deklarasyonu'na uyuldu.
- 2. Etik kurul onayı alındıktan sonra Sağlık Bilimleri Üniversitesi Bilimsel Araştırmalar Proje Birimi, Doktora Projesi başvurusunda bulunuldu ve kabul alındı (BAP Proje no: 2020/13).
- 3. Araştırmada kullanılacak olan Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ) için ayrı bir etik kurul alındı (EK 5). FEGBÖ ölçeği araştırmacılar tarafından tez çalışmasından önce geliştirildi (EK 2).
- 4. Araştırmada kullanılan Bulunuşluk Hissi Ölçeği (BHÖ)'nün kullanımı için sorumlu yazardan e-posta ile izin alındı (EK 13).
- 5. Araştırmada kullanılan Bilişsel Yük Ölçeği (BYÖ) için sorumlu yazara iki kez eposta gönderildi fakat geri dönüş alınamadı. Ölçeğin kullanımı, yazarların yayın sürecinde dergi ile yaptıkları Telif Hakkı Devir Formu doğrultusunda, ölçeğin dergide yayımlanması durumu referans alınarak ve ölçeğe atıf yapılarak kullanıldı (EK 14).
- 6. Araştırma yapılacak kurumdan yazılı kurum izni alındı (EK 15).
- 7. Araştırmaya katılan öğrencilere araştırma ile ilgili bilgi verilerek araştırma anlatıldı. Araştırma ile ilgili detaylı bilgi verildikten sonra sözlü ve yazılı onamları alındı (EK 10). Aynı zamanda öğrencilerden uygulama sırasında kullanılacak görseller içinde sözlü ve yazılı onam alındı (EK 16).

#### 4. BULGULAR

Bu bölümde, "Sanal Gerçeklik Teknolojisi ile Oluşturulan Gelişim Uygulaması (SGT-FEGU)" için sanal gebeliğin tasarlanması ve tasarlanan sanal gebeliğin ebelik eğitimi üzerine etkinliğinin değerlendirilmesi amacıyla randomize kontrollü olarak gerçekleştirilen araştırmanın istatistiksel analizleri sonucunda elde edilen bulgular tablolar halinde sunulmuştur. Araştırmadan elde edilen bulgular;

- 1. Deney ve Kontrol grubundaki öğrencilerin sosyo-demografik ve tanımlayıcı özelliklerine ait bulgular,
- 2. Deney ve Kontrol grubundaki öğrencilerin öğretim materyallerine (Teori eğitimi ve VR uygulaması) ilişkin bilgi düzeylerine ait bulgular,
- 3. Deney grubundaki öğrencilerin sanal gerçeklik uygulamasına ait bilişsel yük ve bulunuşluk hissi düzeylerine ait bulgular,
- 4. Deney grubundaki öğrencilerin deneyimledikleri sanal gerçeklik uygulamasındaki kalitatif geri bildirimlerine ait bulgular, başlıkları altında ele alınmıştır.

# 4.1. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN SOSYO-DEMOGRAFİK/TANIMLAYICI ÖZELLİKLERİNE İLİŞKİN BULGULAR

Tablo 4.1: Deney ve kontrol grubunun sosyo-demografik ve tanımlayıcı özellikleri

| Tanımlayıcı Özellikler | D | eney | Kontrol | | Toplam | Toplam is | | p |
|---|---|---|---|---|---|---|---|---|
| | orta<br>sta | tmetik<br>lama ±<br>ndart<br>pma | Aritme<br>ortalam<br>standa<br>sapm | a ±<br>rt | Aritmeti<br>ortalama<br>standar<br>sapma | ± | <u>i</u><br>t* | p |
| Yaş | 22,3 | 8±0,88 | 22,54±0 | ,88 | 22,46±0,8 | 38 | 0,86 | 0,79 |
| Sınıf Ortalama | 2,9 | 4±0,36 | 2,88±0 | ,45 | 2,91±0,4 | 1 | -0,72 | 0,41 |
| Bölüm Tercih Sırası | 8,8 | 0±7,44 | 6,97±6 | ,44 | 7,89±6,8 | 8 | -1,2 | 0,13 |
| | n | % | n | % | n | % | x <sup>2**</sup> | p |
| En Uzun Süre Yaşanıla | n yer | | | | | | | |
| Şehir Merkezi | 20 | 47,6 | 21 | 50 | 41 | 48,8 | | |
| İlçe | 14 | 33,3 | 15 | 36 | 29 | 34,5 | 0,34 | 0,84 |
| Köy | 8 | 19 | 6 | 14 | 14 | 16,7 | | |
| Şu an yaşadığınız yer | | | | | | | | |
| Yurt | 17 | 40,5 | 17 | 40,5 | 34,0 | 40,5 | | |
| Aile Yanı | 5 | 11,9 | 5 | 11,9 | 10,0<br>0 | 11,9 | 0,000 | 1,000 |
| Arkadaşlarla Ev | 20 | 47,6 | 20 | 47,6 | 40,0<br>0 | 47,6 | | |
| Bölümü İsteyerek Terci | h Etme | Durumu | | | | | | |
| Evet | 31 | 74 | 37 | 88 | 68 | 81 | | |
| Hayır | 11 | 26 | 5 | 12 | 16 | 19 | 2,77 | 0,095 |
| Mesleği Tercih Etme No | edenleri | | | | | | | |
| Ekonomik nedenler | 14 | 33 | 12 | 29 | 26 | 31 | | |
| İş bulma kolaylığı | 6 | 14 | 4 | 10 | 10 | 12 | | |
| Aile İsteği | 16 | 38 | 22 | 52 | 38 | 45 | 1,901 | 0,591 |
| Kendi seçimim (ilgi duyuyor olmam) | 6 | 14 | 4 | 10 | 10 | 12 | | |
| Mezuniyet sonrası plan | lar | | | | | | | |
| Devlet ya da özel bir<br>kuruma girip çalışmak | 28 | 67,7 | 32 | 76,2 | 60 | 71,4 | | |
| Akademisyen olarak çalışmak | 10 | 23,8 | 8 | 19 | 18 | 21,4 | 1,156 | 0,561 |
| Çalışmak ve yüksek<br>lisans yapmak | 4 | 9,5 | 2 | 4,8 | 6 | 7,1 | | |

<sup>\*</sup>Independent- Sample T Testi, \*\*Kikare Testi.

Deney ve kontrol grupların sosyo-demografik özellikleri ile tanımlayıcı istatistikleri incelendiğinde her iki grubunda benzer dağılım gösterdiği aralarında anlamlı fark olmadığı görülmüştür (Tablo 4.1). Grupların yaş dağılımları incelendiğinde deney grubunun 22,38±0,88, kontrol grubunun 22,54±0,88 olduğu saptandı. Deney ve Kontrol gruplarının sınıf not ortalamaları sırasıyla 2,94±0,36 ve 2,88±0,45, bölüm tercih sıralarının ise 8,80±7,42 ile 6,97±6,44 olduğu görüldü (Tablo 4.1).

Deney ve kontrol gruplarındaki yer alan öğrencilerin en uzuz yaşadıkları yer incelendiğinde; deney grubunun %47,6'sının şehir merkezi, %33'ünün ilçe ve %19'unun köy, kontrol grubundaki öğrencilerin ise; %50'sinin şehir merkezi, %36'sının ilçe ve %14'ünün de köy olduğu saptadı. Öğrencilerin şu an yaşadığı kişiler/yer sorgulandığında; deney grubunun %40,5'inin yurtta, %11,9'unun aile yanında ve %47,6'sınında arkadaşlarıyla evde, kontrol grubundaki öğrencilerinin de benzer şekilde, %40,5'inin yurtta, %11,9'unun aile yanında ve %47,6'sınında arkadaşlarıyla evde yaşadığı görülmüştür (Tablo 4.1).

Öğrencilerin bölümü isteyerek tercih etme nedenleri incelendiğinde; deney grubunun %74,0'nün, kontrol grubunun ise; %88,0'nin isteyerek tercih ettiği saptanmıştır. Öğrencilerin mesleği tercih etme nedenleri incelendiğinde; deney grubunun %33,0'nün ekonomik nedenler, %14,0'ünün iş bulma kolaylığı, %38'inin aile isteği ve %14,0'nün kendi isteği olduğu, kontrol grubunun ise; %29'unun ekonomik nedenler, %10,0'nun iş bulma kolaylığı, %52,0'sinin aile isteği ve %10,0'unun kendi isteği olduğu görülmüştür. Öğrencilerin mezuniyet sonrası planları incelendiğinde deney grubunun; %67,7'sinin atanıp ya da özel bir kuruma girip çalışmak, %23,8'inin akademisyen olarak çalışmak ve %9,5'inin hem ebe olarak çalışmak hem de yüksek lisans yapmak olduğu, kontrol grubunun ise; %76,2'sinin atanıp ya da özel bir kuruma girip çalışmak, %19'nun akademisyen olarak çalışmak ve%4,8'nin de hem ebe olarak çalışmak hem de yüksek lisans yapmak olduğu saptanmıştır.

Tablo 4.2: Öğrencilerin bilgisayar oyunu oynama ve sanal gerçeklik uygulaması bilgileri

| Bilgisayar Oyunu<br>Oynama ve Sanal<br>gerçeklik bilgileri | D | eney | Ko | ntrol | Toplam | | Test<br>istatistiği<br>t* | p |
|---|---|---|---|---|---|---|---|---|
| Bilgisayar Oyunu Oyn | ama Du | rumları | | | | | | |
| Evet | 18 | 42,9 | 20 | 47,6 | 38 | 45,2 | 1 100 | 0.661 |
| Hayır | 24 | 57,1 | 22 | 52,4 | 46 | 54,8 | 1,192 | 0,661 |
| Bilgisayar Oyunu Oyn | ama Sık | lığı** | | | | | | |
| Ayda bir gün | 7 | 38,9 | 7 | 35 | 14 | 36,8 | | |
| Haftada bir gün | 3 | 16,7 | 4 | 20 | 7 | 18,4 | | |
| Her gün | 1 | 5,6 | 1 | 5 | 2 | 5,3 | 1,050 | 0,645 |
| Çok Nadir | 7 | 38,9 | 8 | 40 | 15 | 39,5 | | |
| Sanal gerçeklik ile ilgi | li bilgi sa | hibi olm | a | | | | | |
| Evet | 13 | 31 | 12 | 29 | 25 | 29,8 | | 0.011 |
| Hayır | 29 | 69 | 30 | 71 | 59 | 70,2 | 0,057 | 0,811 |
| Sanal Gerçeklik (VR) | yöntemi | nin kulla | nıldığı he | rhangi bir | uygular | naya katı | lma durumla | rı |
| Evet | 3 | 7,1 | 2 | 4,8 | 5 | 6 | 0.010 | 0.645 |
| Hayır | 39 | 92,9 | 40 | 95,2 | 79 | 94 | 0,213 | 0,645 |
| Öğrencilerin Deneyim | ledikleri | VR uygu | ılamalar | *** | | | | |
| Gerçek bir ortam | 2 | 66,7 | 0 | 0 | 2 | 40 | | |
| Eğlenceli | 0 | 0 | 1 | 50 | 1 | 20 | 0,540 | 0,950 |
| Etkileyici | 1 | 33,3 | 1 | 50 | 2 | 40 | | , |
| Toplam | 42 | 100 | 42 | 100 | 84 | 100 | | |

<sup>\*</sup>Kikare Testi. \*\*Analiz Deney grubu için 18 öğrenci, kontrol grubu içinse 20 öğrenci üzerinde yapılmıştır.

Öğrencilerin bilgisayar oyunu oynama durumları incelenmiş; deney grubunun %42,9'unun, kontrol grubun ise %47,6'sının bilgisayar oyunu oynadığı saptanmıştır (Tablo 4.2). Bilgisayar oyunu oynayan öğrencilerin oyun oynama sıklığı incelendiğinde; deney grubundaki öğrencilerin (18 öğrenci); %5,6'sının her gün, %16,7'sinin haftada 1 gün, %38,9'unun ayda 1 gün, %38,9'ununda çok nadir, kontrol grubundaki öğrencilerin (20 öğrenci) ise; %5'inin her gün, %20'sinin haftada 1 gün, %35'inin ayda 1 gün, %40'ınında çok nadir olduğu görülmüştür.

Deney ve kontrol grubundaki öğrencilerin sanal gerçeklik ile ilgili bilgi durumları sorulduğunda; deney grubunun %31'inin, kontrol grubunun ise %29'unun bilgi sahibi olduğu görülmüştür. Öğrencilerin VR yöntemin kullanıldığı herhangi bir uygulamaya katılma durumları sorgulandığında; deney grubundaki öğrencilerin %7,1'inin, kontrol grubunda ise %4,8'inin bir uygulamaya katıldığı saptanmıştır.

<sup>\*\*\*</sup>Analiz Deney grubu için 3 öğrenci, kontrol grubu içinse 2 öğrenci üzerinde yapılmıştır.

**Tablo 4.3:** Deney ve kontrol grubunun bağımsız değişkenler ile binary lojistik regresyon analizi

| Bağımsız Değişkenler | β | Standart<br>Hata<br>(S.E.) | Wald | p | Exp(β)<br>Odd<br>Oranı | | Güven<br>alığı |
|---|---|---|---|---|---|---|---|
| Sabit (Constant) | 1,808 | 7,554 | 0,057 | 0,811 | 6,099 | | |
| Yaş | -0,181 | 0,302 | 0,362 | 0,548 | 0,834 | 0,462 | 1,507 |
| Ön test Puanları | -0,107 | 0,061 | 3,058 | 0,080 | 0,899 | 0,797 | 1,013 |
| Son Test Puanları | 0,209 | 0,083 | 6,396 | 0,011 | 1,233 | 1,048 | 1,450 |
| Bölüm tercih sırası | 0,014 | 0,039 | 0,138 | 0,710 | 1,015 | 0,940 | 1,095 |
| Sanal Gerçeklik (VR) | 0,230 | 1,387 | 0,027 | 0,868 | 1,258 | 0,083 | 19,081 |
| yönteminin kullanıldığı | -, | , | - , | - , | , | - , | - , |
| herhangi bir uygulamaya<br>katılma durumları (Ref. Kat:<br>Last kategori olan hayır olarak<br>alınmıştır). | | | | | | | |
| Sanal gerçeklik ile ilgili bilgi<br>sahibi olma (Ref. Kat: Last<br>kategori olan hayır olarak<br>alınmıştır). | 0,255 | 0,575 | 0,196 | 0,658 | 1,290 | 0,418 | 3,985 |
| Bilgisayar oyunu oynama<br>durumları (Ref. Kat: Last<br>kategori olan hayır olarak<br>alınmıştır). | 0,005 | 0,550 | 0,000 | 0,992 | 1,005 | 0,342 | 2,953 |
| Mezuniyet sonrası planlar (Ref<br>Kat: Hem ebe olarak çalışıp<br>hem de yüksek lisans yapmak) | | | 0,919 | 0,632 | | | |
| Atanıp ya da özel bir kuruma<br>girip çalışmak | -0,886 | 1,252 | 0,500 | 0,479 | 0,412 | 0,035 | 4,800 |
| Akademisyen olarak çalışmak | -0,435 | 1,384 | 0,099 | 0,753 | 0,647 | 0,043 | 9,747 |
| Mesleği<br>Tercih Etme Nedenleri (Ref<br>Kat: Kendi seçimim (ilgi<br>duyuyor olmam) | | | 0,454 | 0,929 | | | |
| Ekonomik nedenler | -0,457 | 0,840 | 0,296 | 0,586 | 0,633 | 0,122 | 3,285 |
| İş bulma kolaylığı | -0,182 | 1,059 | 0,030 | 0,863 | 0,833 | 0,105 | 6,642 |
| Aile İsteği | -0,518 | 0,851 | 0,371 | 0,543 | 0,596 | 0,112 | 3,157 |
| Bölümü İsteyerek Tercih Etme<br>Durumu (Ref. Kat: Last<br>kategori olan hayır olarak | -0,295 | 0,777 | 0,144 | 0,704 | 0,745 | 0,162 | 3,416 |
| alınmıştır). | | | | | | | |
| En Uzun Süre Yaşanılan yer<br>(Ref. Kat: Köy)<br>Şehir Merkezi | -0,182 | 0,756 | 0,059 | 0,971<br>0,810 | 0,834 | 0,189 | 3,670 |
| İlçe<br>Şu an Yaşadığınız yer (Ref kat:<br>Arkadaşlarla Ev) | -0,123 | 0,796 | 0,024<br>0,085 | 0,877<br>0,958 | 0,885 | 0,186 | 4,207 |
| Yurt<br>Aile Yanı | -0,162<br>-0,006 | 0,580<br>0,840 | 0,078<br>0,000 | 0,780<br>0,995 | 0,850<br>0,994 | 0,273<br>0,192 | 2,652<br>5,157 |

Model Uyum Chi Square=17,245 p=0,00, Cox&Snell R2=0,186; Nagelkerke R2=0,24; Hosmer and Lemeshow Chi Square=7,002, p=0,536; DS=%67,9

Çalışmamıza katılan öğrencilerin sanal gerçeklik uygulaması kullanma ve kullanmama (Deney ve kontrol) durumları ile; yaş, en uzun yaşanılan yer, bölümü tercih etme sırası, şimdiye kadar ki akademik başarısı (4 üzerinden), okuldan mezun olduktan sonraki planları, Bilgisayar oyunu oynama durumları, Sanal gerçeklik ile ilgili bilgi sahibi olma durumları, Fetal gelişimi değerlendirme ön test ve son test puanları arasındaki ilişki binary lojistik regresyon analizi ile incelenmiştir (Tablo 3). Oluşturulan SGT-FEGU'yu kullanan ve teori eğitimi alan olgularda bu parametrelerin etkilerini binary lojistik regresyon analizi ile değerlendirdiğimizde modelin düzeyde anlamlı (Hosmer and Lemeshow test: 0536) bulunduğu ve doğru sınıflandırma oranının %67,9 ile başarılı olduğu görülmüştür. Modelde VR kullanma (deney grubu) ile kullanmamanın (klasik teori eğitimi- kontrol grubu) son test puanları arasındaki ilişki anlamlı bulunmuştur (p=0,011). Modeldeki diğer parametreler arasında anlamlı ilişki saptanmamıştır (Tablo 3).

# 4.2. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN ÖĞRETİM MATERYALLERİNE (SG UYGULAMASI ve TEORİ EĞİTİMİ) İLİŞKİN BİLGİ DÜZEYLERİNE AİT BULGULAR

Araştırmada kullanılan fetal gelişimi değerlendirme ölçeğinin toplam gruptaki ön test cronbach's alfası 0,79, son test cronbach's alfası ise 0,77 olarak bulunmuştur. Deney ve kontrol grubu ayrı ayrı bakıldığında ise; deney ölçek ön test cronbach's alfası 0,79, son test cronbach's alfası 0,70 olarak saptanmıştır. Kontrol grubunun ön test cronbach's alfası 0,78, son test Cronbach's alfası da 0,81 olarak saptanmıştır. Deney ve Kontrol grubundaki öğrencilerin fetal gelişim ile ilgili uygulanan teori ve VR uygulama materyallerinin ön test ve son test sonuçları, sorulara verdikleri doğru ve yanlış cevapların yüzdesi aşağıda incelenmiştir.

Tablo 4.4: Deney grubundaki öğrencilerin fetal gelişim ölçeğine verdikleri doğru ve yanlış cevaplar

| Feta | Fetal Gelişim Bilgi Ölçeği Soruları | | Γest | | | Son To | est | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | oğru | Yanlış/Bilmiyorum | | Doğru | | Yanlış/E | Bilmiyorum |
| | | n* | %** | n* | %** | n* | %** | n* | %** |
| 1 | Sperm ve ovumun mayoz bölünme sonucu yarıya indirgenen kromozomları fertilizasyonla 46 kromozomlu yeni bir hücre olan "zigotu" meydana getirir | 36 | 85,7 | 6 | 14,3 | 42 | 100 | 0 | 0 |
| 2 | İlk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | 31 | 73,8 | 11 | 26,2 | 39 | 92,9 | 3 | 7,1 |
| 3 | Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir | 24 | 57,1 | 18 | 42,9 | 34 | 81 | 8 | 19 |
| 4 | Trofoblastların dış tabakası sinsityotrofoblastlardır. | 31 | 73,8 | 11 | 26,2 | 37 | 88,7 | 5 | 11,3 |
| 5 | Embriyonel evreye organogenezis evresi de denir. | 23 | 54,8 | 19 | 45,2 | 35 | 83,3 | 7 | 16,7 |
| 6 | Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. | 17 | 40,5 | 25 | 59,6 | 27 | 64,3 | 15 | 35,7 |
| 7 | 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. | 22 | 52,4 | 20 | 47,6 | 34 | 81 | 8 | 19 |
| 8 | Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir | 27 | 64,3 | 15 | 35,7 | 36 | 85,7 | 6 | 14,3 |
| 9 | 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. | 25 | 59,5 | 17 | 40,5 | 33 | 78,6 | 9 | 21,4 |
| 10 | Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. | 20 | 47,6 | 22 | 52,4 | 29 | 69 | 13 | 31 |
| 11 | Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. | 12 | 28,6 | 30 | 71,4 | 26 | 61,9 | 16 | 38,1 |
| 12 | 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. | 23 | 54,8 | 19 | 45,2 | 34 | 81 | 8 | 19 |
| 13 | Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. | 17 | 40,5 | 25 | 59,5 | 36 | 85,7 | 6 | 14,3 |
| 14 | Umblikal kord 12. haftanın sonunda gelişir. | 22 | 52,4 | 20 | 47,6 | 34 | 81 | 8 | 19 |
| 15 | Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. | 21 | 50 | 21 | 50 | 35 | 83,3 | 7 | 16,7 |
| 16 | 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. | 21 | 50 | 21 | 50 | 31 | 73,8 | 11 | 26,2 |
| 17 | Bağırsakların gelişimi 13. haftada gelişmeye başlar. | 14 | 33,3 | 28 | 66,7 | 28 | 73,8 | 14 | 26,2 |
| 18 | Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. | 13 | 31 | 29 | 69 | 33 | 78,6 | 9 | 21,4 |
| 19 | Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. | 13 | 31 | 29 | 69 | 31 | 73,8 | 11 | 26,2 |
| 21 | 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. | 18 | 42,9 | 24 | 57,1 | 24 | 57,1 | 18 | 42,9 |
| 21 | Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. | 23 | 54,8 | 19 | 45,2 | 38 | 90,5 | 4 | 9,5 |
| 22 | 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | 24 | 57,1 | 18 | 42,9 | 36 | 85,7 | 6 | 14,3 |
| 23 | Fetüs 36-40. haftalarda dış ortama artık uyum sağlayabilir. | 38 | 90,5 | 4 | 9,5 | 41 | 97,6 | 1 | 2,4 |

<sup>\*</sup>n: Öğrenci sayısı %: Yüz.

**Tablo 4.5:** Deney grubundaki öğrencilerin ön test ve son test sonrası doğru cevap veren kişi sayısı

| Feta | l Gelişim Bilgi Ölçeği Soruları | Ön<br>Test | Son<br>Test |
|---|---|---|---|
| | | n* | n* |
| 1 | Sperm ve ovumun mayoz bölünme sonucu yarıya indirgenen kromozomları | 36 | 42 |
| | fertilizasyonla 46 kromozomlu yeni bir hücre olan "zigotu" meydana getirir | | |
| 2 | İlk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | 31 | 39 |
| 3 | Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir | 24 | 34 |
| 4 | Trofoblastların dış tabakası sinsityotrofoblastlardır. | 31 | 37 |
| 5 | Embriyonel evreye organogenezis evresi de denir. | 23 | 35 |
| 6 | Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. | 17 | 27 |
| 7 | 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. | 22 | 34 |
| 8 | Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir | 27 | 36 |
| 9 | 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. | 25 | 33 |
| 10 | Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. | 20 | 29 |
| 11 | Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. | 12 | 26 |
| 12 | 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. | 23 | 34 |
| 13 | Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. | 17 | 36 |
| 14 | Umblikal kord 12. haftanın sonunda gelişir. | 22 | 34 |
| 15 | Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. | 21 | 35 |
| 16 | 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. | 21 | 31 |
| 17 | Bağırsakların gelişimi 13. haftada gelişmeye başlar. | 14 | 28 |
| 18 | Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. | 13 | 33 |
| 19 | Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. | 13 | 31 |
| 20 | 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. | 18 | 24 |
| 21 | Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. | 23 | 38 |
| 22 | 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | 24 | 36 |
| 23 | Fetüs 36-40. haftalarda dış ortama artık uyum sağlayabilir. | 38 | 41 |

<sup>\*</sup>Doğru cevap veren öğrenci sayısı

Deney grubundaki öğrencilerin FEGBÖ'ye verdikleri ön test ve son test sonuçları Tablo 4.4 ve 4.5'te verilmiştir. Öğrencilerin ölçekteki her maddeyi verdikleri doğru ve yanlış cevapların dağılımı yüzde ve sayı olarak incelenmiştir.

Deney grubundaki öğrencilerin ön testte en yüksek doğru cevap verdikleri sorular sırasıyla, 1 (%85,7), 2 (%73,8), 4 (%73,5) ve 23 (%90,5) olarak saptanmıştır. Bunun yanı sıra en fazla yanış verilen cevaplar ise sırasıyla; 6 (%59,6), 10 (%52,4), 11 (%71,4), 13 (%59,6), 17 (%66,7), 18 (%69), 19 (%69), 20 (%57,1), 21 (%45,2), ve 22 (%42,9) olarak bulunmuştur (Tablo 4.4).

Deney grubundaki öğrencilerin son test cevapları incelendiğinde, doğru cevaplayan öğrenci sayısının %53,3'ün üzerinde olduğu görülmüştür. Öğrencilerin yanlış cevapları incelendiğinde, 6 (%35,7), 11 (%38,1) ve 20 (%42,9) yüksek oranda yanlış

cevaplandığı görülmüştür (Tablo 4.4). Deney grubundaki öğrencilerin ön test ve son testteki doğru cevapları tablo 5'te incelenmiştir. Ön testteki doğru cevap veren öğrenci sayısının ortalama 22 olarak saptanırken, son testi doğru cevaplayan öğrenci sayısı ortalamasının 33 olduğu görülmüştür. Son teste doğru cevap veren öğrenci sayısının ön teste doğru cevap veren öğrenci sayısına oranla daha yüksel saptanmıştır (Tablo 4.5).

Deney grubundaki öğrencilerin ön test ve son test ölçümleri arasındaki ilişki Tablo 4.6'da görülmektedir.

**Tablo 4.6:** Deney grubundaki öğrencilerin ön test ve son test cevaplarının karşılaştırılması

| Fetal | Gelişim Bilgi Ölçeği Soruları | Ön Te<br>Son T | |
|---|---|---|---|
| Soru<br>No | | Test<br>İstatistiği<br>t* | p |
| 1 | Sperm ve ovumun mayoz bölünme sonucu yarıya indirgenen kromozomları fertilizasyonla 46 kromozomlu yeni bir hücre olan "zigotu" meydana getirir | -2,614 | 0,012 |
| 2 | İlk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | -2,442 | 0,019 |
| 3 | Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir | -2,354 | 0,023 |
| 4 | Trofoblastların dış tabakası sinsityotrofoblastlardır. | -1,776 | 0,083 |
| 5 | Embriyonel evreye organogenezis evresi de denir. | -3,106 | 0,003 |
| 6 | Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. | -2,354 | 0,023 |
| 7 | 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. | -2,751 | 0,009 |
| 8 | Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir | -2,291 | 0,027 |
| 9 | 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. | -1,947 | 0,058 |
| 10 | Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. | -2,036 | 0,048 |
| 11 | Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. | -3,788 | 0,000 |
| 12 | 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. | -2,892 | 0,006 |
| 13 | Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. | -4,376 | 0,000 |
| 14 | Umblikal kord 12. haftanın sonunda gelişir. | -2,751 | 0,009 |
| 15 | Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. | -3,146 | 0,003 |
| 16 | 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. | -2,125 | 0,040 |
| 17 | Bağırsakların gelişimi 13. haftada gelişmeye başlar. | -3,532 | 0,001 |
| 18 | Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. | -4,367 | 0,000 |
| 19 | Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. | -4,705 | 0,000 |
| 20 | 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. | -1,289 | 0,205 |
| 21 | Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. | -3,747 | 0,001 |
| 22 | 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | -2,751 | 0,009 |
| 23 | Fetüs 36-40. haftalarda dış ortama artık uyum sağlayabilir. | -1,355 | 0,183 |

<sup>\*</sup> Paired- Sample T testi

Deney grubundaki öğrencilerin ön test ve son test sonrası FEGBÖ'ye verdiği cevaplar arasındaki fark Paired- Sample T testi ile karşılaştırılmıştır. Anlamlılık düzeyi

p<0,05 olarak alınmıştır. Deney grubundaki öğrencilerin 4, 9, 20. ve 23. Sorular hariç diğer tüm sorularda ön test- son test cevapları arasında anlamlı fark saptanmıştır (Tablo 4.6). Anlamlı bulunmayan bu soruların hem ön testte hem de son testte doğru olarak yanıtlandığı görülmüştür (Tablo 4.6).

Kontrol grubundaki öğrencilerin FEGBÖ'ye verdikleri ön test ve son test sonuçları Tablo 4.7 ve 4.8'de verilmiştir. Öğrencilerin ölçekteki her maddeyi verdikleri doğru ve yanlış cevapların dağılımı yüzde ve sayı olarak incelenmiştir.

**Tablo 4.7:** Kontrol grubundaki öğrencilerin fetal gelişim ölçeğine verdikleri doğru ve yanlış cevaplar (n:42)

| Fetal Gelişim Bilgi Ölçeği Soruları | | | | Ön Test | | Son Test | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Doğru Yanlış/Bilm | | | iyorum Doğru | | Bilmiyorum |
| | | n* | %** | n* | 0/0** | n* | %** | n* | %** |
| 1 | Sperm ve ovumun mayoz bölünme sonucu yarıya indirgenen kromozomları | 40 | 95,2 | 2 | 4,8 | 41 | 97,6 | 1 | 2,4 |
| | fertilizasyonla 46 kromozomlu yeni bir hücre olan "zigotu" meydana getirir | | | | | | | | |
| 2 | İlk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | 35 | 83,3 | 7 | 16,7 | 35 | 83,3 | 7 | 16,7 |
| 3 | Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir | 27 | 64,3 | 15 | 35,7 | 28 | 66,7 | 14 | 33,3 |
| 4 | Trofoblastların dış tabakası sinsityotrofoblastlardır. | 34 | 81,0 | 8 | 19,0 | 35 | 83,3 | 7 | 16,7 |
| 5 | Embriyonel evreye organogenezis evresi de denir. | 23 | 54,8 | 19 | 45,2 | 26 | 61,9 | 16 | 38,1 |
| 6 | Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. | 16 | 38,1 | 26 | 61,9 | 26 | 61,9 | 16 | 38,1 |
| 7 | 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. | 26 | 61,9 | 16 | 38,1 | 29 | 69,0 | 13 | 31,0 |
| 8 | Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir | 30 | 71,4 | 12 | 28,6 | 33 | 78,6 | 9 | 21,4 |
| 9 | 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. | 26 | 61,9 | 16 | 38,1 | 29 | 69,0 | 13 | 31,0 |
| 10 | Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. | 22 | 52,4 | 20 | 47,6 | 27 | 64,3 | 15 | 35,7 |
| 11 | Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. | 16 | 38,1 | 26 | 61,9 | 23 | 54,8 | 19 | 45,2 |
| 12 | 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. | 33 | 78,6 | 9 | 21,4 | 32 | 76,2 | 10 | 23,8 |
| 13 | Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. | 27 | 64,3 | 15 | 35,7 | 32 | 76,2 | 10 | 23,8 |
| 14 | Umblikal kord 12. haftanın sonunda gelişir. | 27 | 64,3 | 15 | 35,7 | 25 | 59,5 | 17 | 40,5 |
| 15 | Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. | 24 | 57,1 | 18 | 42,9 | 30 | 71,4 | 12 | 28,6 |
| 16 | 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. | 29 | 69,0 | 13 | 31,0 | 34 | 81,0 | 8 | 19,0 |
| 17 | Bağırsakların gelişimi 13. haftada gelişmeye başlar. | 21 | 50,0 | 21 | 50,0 | 25 | 59,5 | 17 | 40,5 |
| 18 | Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. | 20 | 47,6 | 22 | 52,4 | 23 | 54,8 | 19 | 45,2 |
| 19 | Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. | 15 | 35,7 | 27 | 64,3 | 22 | 52,4 | 20 | 47,6 |
| 21 | 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. | 20 | 47,6 | 22 | 52,4 | 24 | 57,1 | 18 | 42,9 |
| 21 | Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. | 26 | 61,9 | 16 | 38,1 | 32 | 76,2 | 10 | 23,8 |
| 22 | 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | 20 | 47,6 | 22 | 52,4 | 28 | 66,7 | 14 | 33,3 |
| 23 | Fetüs 36-40. haftalarda dış ortama artık uyum sağlayabilir. | 35 | 83,3 | 7 | 16,7 | 34 | 81,0 | 8 | 19,0 |

<sup>\*</sup>n= 42 n: Öğrenci sayısı%: Yüzde

**Tablo 4.8:** Kontrol grubundaki öğrencilerin ön test ve son test sonrası doğru cevap veren kişi sayısı

| Sıra<br>No | Fetal Gelişim Bilgi Ölçeği Soruları | Ön<br>Test | Son<br>Test |
|---|---|---|---|
| INO | | Test | Test |
| | | n | n |
| 1 | Sperm ve ovumun mayoz bölünme sonucu yarıya indirgenen kromozomları fertilizasyonla 46 kromozomlu yeni bir hücre olan "zigotu" meydana getirir | 40 | 41 |
| 2 | İlk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | 35 | 35 |
| 3 | Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir | 27 | 28 |
| 4 | Trofoblastların dış tabakası sinsityotrofoblastlardır. | 34 | 35 |
| 5 | Embriyonel evreye organogenezis evresi de denir. | 23 | 26 |
| 6 | Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. | 16 | 26 |
| 7 | 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. | 26 | 29 |
| 8 | Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir | 30 | 33 |
| 9 | 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. | 26 | 29 |
| 10 | Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. | 22 | 27 |
| 11 | Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. | 16 | 23 |
| 12 | 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. | 33 | 32 |
| 13 | Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. | 27 | 32 |
| 14 | Umblikal kord 12. haftanın sonunda gelişir. | 27 | 25 |
| 15 | Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. | 24 | 30 |
| 16 | 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. | 29 | 34 |
| 17 | Bağırsakların gelişimi 13. haftada gelişmeye başlar. | 21 | 25 |
| 18 | Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. | 20 | 23 |
| 19 | Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. | 15 | 22 |
| 20 | 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. | 20 | 24 |
| 21 | Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. | 26 | 32 |
| 22 | 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | 20 | 28 |
| 23 | Fetüs 36-40. haftalarda dış ortama artık uyum sağlayabilir. | 35 | 34 |

<sup>\*\*</sup>Doğru cevap veren öğrenci sayısı

Kontrol grubundaki öğrencilerin ön testte en yüksek doğru cevap verdikleri sorular sırasıyla, 1 (%95,2), 2 (%83,3), 4 (%81), 8 (%71,4), 12 (%78,6) ve 23 (%90,5) olarak saptanmıştır. Bunun yanı sıra en fazla yanış verilen cevaplar ise sırasıyla; 6 (%61,9), 11 (%71,4), 19 (%64,3) ve 22 (%42,9) olarak bulunmuştur (Tablo 4.7).

Kontrol grubundaki öğrencilerin son test cevapları incelendiğinde, doğru cevaplayan öğrenci sayısının %61'nin üzerinde olduğu görülmüştür. Öğrencilerin yanlış cevapları incelendiğinde, 6 (%35,7), 11 (%38,1) ve 20 (%42,9) yüksek oranda yanlış cevaplandığı görülmüştür (Tablo 4.7). Kontrol grubundaki öğrencilerin ön test ve son testteki doğru cevapları tablo 8'de incelenmiştir. Ön testteki doğru cevap veren öğrenci sayısının

ortalama 25 olarak saptanırken, son testi doğru cevaplayan öğrenci sayısı ortalamasının 29 olduğu görülmüştür. Son teste doğru cevap veren öğrenci sayısının ön teste doğru cevap veren öğrenci sayısına oranla daha yüksel saptanmıştır (Tablo 4.8).

Kontrol grubundaki öğrencilerin ön test ve son test ölçümleri arasındaki ilişki Tablo 4.9'da karşılaştırılmıştır.

**Tablo 4.9:** Kontrol grubundaki öğrencilerin ön test ve son test cevaplarının karşılaştırılması

| Sıra | Fetal Gelişim Bilgi Ölçeği Soruları | Ön Te | |
|---|---|---|---|
| No | | Son T<br>Test | |
| | | İstatistiği | p |
| | | t* | |
| 1 | Sperm ve ovumun mayoz bölünme sonucu yarıya indirgenen kromozomları | -0,573 | 0,570 |
| | fertilizasyonla 46 kromozomlu yeni bir hücre olan "zigotu" meydana getirir | | |
| 2 | İlk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | 0,000 | 1,000 |
| 3 | Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir | -0,198 | 0,844 |
| 4 | Trofoblastların dış tabakası sinsityotrofoblastlardır. | -0,274 | 0,785 |
| 5 | Embriyonel evreye organogenezis evresi de denir. | -0,771 | 0,445 |
| 6 | Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. | -2,354 | 0,023 |
| 7 | 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. | -0,684 | 0,498 |
| 8 | Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir | -0,903 | 0,372 |
| 9 | 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun | -0,650 | 0,519 |
| | ve kulaklar belirmeye başlar. | | |
| 10 | Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. | -1,152 | 0,256 |
| 11 | Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. | -1,553 | 0,128 |
| 12 | 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen | 0,255 | 0,800 |
| | perdeler ile birbirine bağlıdır. | | |
| 13 | Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. | -1,152 | 0,256 |
| 14 | Umblikal kord 12. haftanın sonunda gelişir. | 0,467 | 0,643 |
| 15 | Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. | -1,289 | 0,205 |
| 16 | 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. | -1,403 | 0,168 |
| 17 | Bağırsakların gelişimi 13. haftada gelişmeye başlar. | -0,850 | 0,400 |
| 18 | Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. | -0,650 | 0,519 |
| 19 | Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. | -1,480 | 0,146 |
| 20 | 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. | -0,813 | 0,421 |
| 21 | Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. | -1,635 | 0,110 |
| 22 | 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | -1,839 | 0,073 |
| 23 | Fetüs 36-40. haftalarda dış ortama artık uyum sağlayabilir. | 0,298 | 0,767 |
| *Doi: | rad Sample T testi | | |

<sup>\*</sup>Paired-Sample T testi

Kontrol grubundaki öğrencilerin ön test ve son test sonrası FEGBÖ'ye verdiği cevaplar arasındaki fark Paired- Sample T testi ile karşılaştırılmıştır. Anlamlılık düzeyi p<0,05 olarak alınmıştır. Kontrol grubundaki öğrencilerinin yalnızca 6. soruya verdiği ön test- son test cevapları arasında anlamlı fark saptanmıştır p<0,05 (Tablo 4.9). Anlamlı

bulunmayan bu soruların hem ön testte hem de son testte doğru olarak yanıtlandığı görülmüştür (Tablo 4.9).

**Tablo 4.10:** Deney ve kontrol gruplarının ölçek toplam puanlarının ön test ve son testlerinin karşılaştırılması

| - | Deney | Kontrol | Test İstatsitiği | p |
|----------|----------------|----------------|------------------|-------|
| | $x\pm ss$ | x±ss | t* | p |
| Ön test | 12,26±4,70 | 14,09±4,49 | 1,826 | 0,071 |
| Son Test | $18,40\pm2,79$ | $16,02\pm4,63$ | -2,853 | 0,006 |

<sup>\*</sup> Independent- Samples T test

Deney ve Kontrol gruplarının ön test son test toplam puanları Independent-Samples T testi ile karşılaştırılmış ve tablo 4.10'da sunulmuştur

Deney grubun FEGBÖ toplam puanları incelendiğinde, ön test puanının  $12,26\pm4,70$ , son test puanının ise  $18,40\pm2,79$  olduğu görülmüştür. Kontrol grubun ölçek puanları karşılaştırıldığında ise; ön test puanlarının  $14,09\pm4,49$ , son test puanlarının da  $16,02\pm4,63$  olduğu saptanmıştır. Deney ve kontrol grubun ön test puanları arasında anlamlı fark saptanmazken (p=0,071), son test puanları arasında anlamlı fark görülmüştür (p=0,006) (Tablo 4.10).

Deney ve kontrol grupların FEGBÖ'nün ön test ve son test toplam puanları, deney ve kontrol rubu kendi arasında öncesi ve sonrası olmak üzere iki zamanlı olarak Paired-Sample T testi ile karşılaştırılmıştır. Aynı zamanda araştırmaya katılan tüm öğrencilerin (deney ve kontrol grubu toplam) toplam puanları öncesi ve sonrası iki zamanlı olarak Paired-Sample T testi ile karşılaştırılmıştır (Tablo 4.11).

**Tablo 4.11:** Deney, kontrol ve tüm grupların ön test ve son test puanlarının karşılaştırılması

| Grup | Zaman | Ön Test | Son Test | Fark | р |
|---|---|---|---|---|---|
| Deney Grubu | Ölçek Toplam Puan | $12,26 \pm 4,75$ | $18,40 \pm 2,79$ | 6,15 | 0,000* |
| Kontrol Grubu | Ölçek Toplam Puan | $14,\!09 \pm 4,\!49$ | $16,02 \pm 4,63$ | 1,93 | 0,043* |
| Toplam | Ölçek Toplam Puan | $13,17\pm4,66$ | $17,\!21\pm3,\!98$ | 4,04 | 0,000* |

<sup>\*</sup>Paired samples t test

Deney grubunun fetal gelişim ölçeği toplam puanları incelendiğinde, ön test toplam puanının  $12,26 \pm 4,75$ , son test puanının da  $18,40 \pm 2,79$  olduğu ve aralarında istatistiksel olarak anlamlı fark bulunduğu saptanmıştır (p=0,000). Kontrol grubun ölçek toplam puanları incelendiğinde, ön test puanının  $14,09 \pm 4,49$ , son test puanının da  $16,02 \pm 4,63$  olduğu, aralarında istatistiksel olarak sınırda anlamlı olduğu görülmüştür (p=0,043). Tüm öğrencilerin ön test ve son test ölçek puanları incelendiğinde, ölçek toplam ön test puanlarının  $13,17 \pm 4,66$ , son test puanlarının da  $17,21 \pm 3,98$  olduğu saptanmıştır. Tüm öğrencilerin ölçek toplam ön test ve son test puanları arasında anlamlı ilişki saptanmıştır (p=0,000) (Tablo 4.11).

**Tablo 4.12:** Deney ve kontrol gruplarında yer alan öğrencilerin fetal gelişimi değerlendirme son test toplam puanlarının kovaryans analizi sonuçları

| Varyansın<br>Kaynağı | Kareler<br>(KT) | Toplamı | Sd | Kareler<br>(KO) | Ortalaması | F* | p |
|---|---|---|---|---|---|---|---|
| Kontrol Edilen<br>Değişken (Öntest) | 17,735 | | 1 | 17,735 | | 1,216 | 0,273 |
| Yöntem | 132,896 | | 1 | 132,896 | | 9,112 | 0,003 |
| Hata | 1181,360 | | 81 | 14,585 | | | |
| Toplam | 26210,000 | | 84 | | | | |

<sup>\*</sup>Ancova Testi

Deney ve kontrol gruplarında yer alan öğrencilerin FEGBÖ son test toplam puanlarının kovaryans analizi sonuçları Tablo 4.12'de verilmiştir.

Kovaryans analizi sonuçları incelendiğinde, deney ve kontrol gruplarının on testtten arındırılmış/düzeltilmiş son test puanları arasında anlamlı fark saptanmıştır (F (5,80)=9,112; p=0,003). Öğrencilere fetal gelişimi öğretiminde kullanılan sanal gerçeklik öğretim yöntemi olan SGT-FEGU'nun teori eğitimine oranla farklılık gösterdiği görülmüştür (Tablo 4.12).

## 4.3. DENEY GRUBUNDAKİ ÖĞRENCİLERİN SANAL GERÇEKLİK UYGULAMASINA AİT BİLİŞSEL YÜK VE BULUNUŞLUK HİSSİ DÜZEYLERİNE AİT BULGULAR

Deney grubundaki öğrencilerin BYÖ puanları Tablo 13'te incelenmiştir.

Tablo 4.13: Deney grubundaki öğrencilerin bilişsel yük puanları

| Grup | n | Ortalama puan | sd | t* | p |
|---|---|---|---|---|---|
| Bilişsel Yük Puan ortalaması | 42 | 1,09±0,29 | | | |
| Bilişsel Olarak Aşırı Yüklenmeyenler | 38 | $1,47\pm0,35$ | 1.63 | -12.26 | 0.000 |
| Bilişsel Olarak Aşırı Yüklenenler | 4 | $6\pm 5,\!27$ | 1,05 | -12,20 | 0,000 |

<sup>\*</sup>One Sample T testi

Öğrencilerin bilişsem yük puan ortalaması 1,09±0,29 olarak bulunmuştur. Öğrencilerin %90,5'nin bilişsel olarak aşırı yüklenmediği, bilişsel yük puanlarının 1-5 arasında değiştiği, %9,5'inin ise bilişsel olarak aşırı yüklendiği, puanlarının 5-9 puan arasında olduğu saptanmıştır (Tablo 4.13). Öğrencilerin bilişsel yük puanları Bilişsel yük ölçeğinin kesme noktası olan 5'e göre One Sample T testi ile karşılaştırılmıştır. 42 öğrencinin BYÖ puan ortalamaları arasında anlamlı fark görülmüştür (p=0,000).

Öğrencilerin bilişsel yük kesme noktası olan 5 puandan daha düşük bir ortalamaya sahip oldukları görülmüştür.

**Tablo 4.14:** Sanal gerçeklik deneyimleyen öğrencilerin bulunuşluk hissi ölçek alt boyutları puan ortalamaları

| Bulunuşluk Hissi Ölçeği Alt | x±ss* | Referans Alına | Test | р |
|---|---|---|---|---|
| Boyutları | | Puan | İstatistiği** | |
| Katılım | $4,67\pm0,44$ | 5 | -4,699 | 0,000 |
| Uyum/Çevreleme | $4,44\pm0,54$ | 5 | -6,595 | 0,000 |
| Duygusal Bağlılık | $4,66\pm0,42$ | 5 | -5,186 | 0,000 |
| Etkileşim | $4,23\pm0,56$ | 5 | -8,803 | 0,000 |
| Ara yüz Kalitesi | $1,65\pm0,82$ | 5 | -26,166 | 0,000 |

<sup>\*</sup>Ortalama ve standart sapma, \*\*One Sample T test

Deney grubuna uygulanan sanal gerçeklik gözlüğünün öğrencilerin sanal ortama ilişkin durumlarını ölçmek için BHÖ uygulanmıştır. Ölçeğin tüm maddelerinin ve alt boyutlarının cronbach's alfa değerleri incelenmiştir. BHÖ' nün tüm maddelerinin (29 madde) cronbach's alfası 0,88, katılım alt boyutunun cronbach's alfası 0,90, uyum/çevreleme alt boyutunun cronbach's alfası 0,84, duygusal bağlılık alt boyutunun cronbach's alfası 0,67, etkileşim alt boyutunun cronbach's alfası 0,68 ve ara yüz kalitesi alt boyutunun cronbach's alfası 0,80 olarak saptanmıştır.

Deney grubundaki öğrencilerin BHÖ'nün alt boyutlarından aldığı puan ortalamaları Tablo 4.14'de verilmiştir. Öğrencilerin katılım alt boyut puanı 4,67±0,44, uyum/çevreleme alt boyut puanı 4,44±0,54, duygusal bağlılık alt boyutu puanı 4,66±0,42, etkileşim alt boyut puanı 4,23±0,56 ve ara yüz kalitesi alt boyut puanı 1,65±0,82 olarak bulunmuştur (Tablo 4.14). Ölçek alt boyutları ile referans puanları one sample T testi ile karşılaştırılmıştır. Her alt boyuttaki alınan puan ortalaması ile referans puan ortalaması arasında anlamlı ilişki görülmüştür. Öğrencilerin aldıkları puan ortalamalarının ölçek alt boyut referansa puanından düşük olduğu görülmüştür (Tablo 4.14).

**Tablo 4.15:** Bilişsel yük ölçeği ile bulunuşluk hissi ölçeğinin alt boyutları arasındaki ilişki

| | BHÖ Ölçeğinin alt boyutları | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| n: 42 | Kat | • | | yum/Çevrel Duygusal<br>eme Bağlılık | | , | Etkileşim | | Ara yüz<br>Kalitesi | |
| Bilişsel Yüke<br>Ölçeği | r<br>-0,24 | p<br>0,116 | r<br>-0,22 | p<br>0,147 | r<br>-0,07 | p<br>0,63 | r<br>-0,36 | p*<br><b>0,01</b> | r<br>-0,10 | p<br>0,51 |

<sup>\*</sup>Korelasyon 0,05 düzeyinde anlamlıdır.

Deney grubundaki öğrencilerin BYÖ ve BHÖ arasındaki ilişki pearson kolerasyon ile incelenmiştir. Deney grubundaki öğrencilerin, BYÖ ve BHÖ'ğinin alt boyutları arasından sadece etkileşim alt boyutu ile negatif yönde orta düzeyde kolerasyon görülmüştür (Tablo 4.15).

**Tablo 4.16:**Sanal gerçeklik ile ilgili bilgi durumunun bulunuşluk hissi ölçeğinin alt boyutları ile binary lojistik regresyon analizi

| | β | Standart<br>Hata (S.E.) | Wald | p | Exp(β)<br>Odd Oranı | %95 Güven<br>Aralığı | |
|---|---|---|---|---|---|---|---|
| | | | | | | Düşük | Yüksek |
| Sabit (Constant) | 0,524 | 4,469 | 0,014 | 1 | 0,907 | | |
| Katılım | -0,078 | 0,153 | 0,262 | 1 | 0,609 | 0,925 | 0,685 |
| Uyum/Çevreleme | -0,027 | 0,141 | 0,036 | 1 | 0,849 | 0,974 | 0,738 |
| Duygusal Bağlılık | -0,067 | 0,244 | 0,076 | 1 | 0,782 | 0,935 | 0,580 |
| Etkileşim | 0,277 | 0,205 | 1,825 | 1 | 0,177 | 1,320 | 0,882 |
| Ara yüz Kalitesi | 0,028 | 0,149 | 0,037 | 1 | 0,848 | 1,029 | 0,769 |

Model Uyum Chi Square=1,987 p=0,016, Cox&Snell R2=0,046; Nagelkerke R2=0,065; Hosmer and Lemeshow Chi Square=5,745 p=0,676; DS=%69

Deney grubundaki öğrencilerin sanal gerçeklik ile ilgili bilgi sahibi olma durumları ile BHÖ'nin alt boyutları arasındaki ilişki binary lojistik regresyon modeli ile açıklanmıştır (Tablo 4.16). Çalışmamıza katılan öğrencilerin sanal gerçeklik uygulaması ile ilgili bilgi durumunun BHÖ alt boyutları olan; Katılım, Uyum/Çevreleme, Duygusal Bağlılık, Etkileşim ve Ara yüz Kalitesi parametreleri arasındaki ilişki binary lojistik regresyon analizi ile incelenmiştir (Tablo 4.16). Oluşturulan modelin sanal gerçeklik uygulaması bilgisi olma durumu ve bu parametrelerin etkilerini binary lojistik regresyon analizi ile değerlendirdiğimizde modelin düzeyde anlamlı (p=0,016) bulunduğu ve doğru sınıflandırma oranının %69 ile başarılı olduğu görülmüştür. Modelde sanal gerçeklik ile ilgili bilgi sahibi, olma durumu ile BHÖ ölçeğinin tüm alt boyutları arasında anlamlı ilişki saptanmamıştır (Tablo 4.16).

**Tablo 4.17:** Sanal gerçeklik ile ilgili uygulamaya katılma durumunun bulunuşluk hissi ölçeği alt boyutları ile binary lojistik regresyon analizi

| | β | Standart<br>Hata (S.E.) | Wald | p | Exp(β)<br>Odd<br>Oranı | | Güven<br>alığı |
|---|---|---|---|---|---|---|---|
| Sabit (Constant) | -3,919 | 8,783 | 0,199 | 1 | 0,655 | | |
| Katılım | -0,112 | 0,222 | 0,255 | 1 | 0,614 | 0,894 | 0,579 |
| Uyum/Çevreleme | -0,107 | 0,259 | 0,172 | 1 | 0,679 | 0,898 | 0,541 |
| Duygusal Bağlılık | 0,794 | 0,419 | 3,582 | 1 | 0,058 | 2,211 | 0,972 |
| Etkileşim | -0,150 | 0,491 | 0,094 | 1 | 0,759 | 0,861 | 0,329 |
| Ara yüz Kalitesi | -0,035 | 0,289 | 0,014 | 1 | 0,904 | 0,966 | 0,549 |

Model Uyum Chi Square=5,105 p=0,000, Cox&Snell R2=0,114; Nagelkerke R2=0,284; Hosmer and Lemeshow Chi Square=11,045 p=0,199; DS=%95,2

Çalışmamıza katılan öğrencilerin sanal gerçekliğin kullanıldığı bir uygulamaya katılma durumlarının BHÖ alt boyutları olan; Katılım, Uyum/Çevreleme, Duygusal Bağlılık, Etkileşim ve Ara yüz Kalitesi parametreleri arasındaki ilişki binary lojistik regresyon analizi ile incelenmiştir (Tablo 4.17). Oluşturulan modelin sanal gerçeklik uygulaması bilgisi olma durumu ve bu parametrelerin etkilerini binary lojistik regresyon analizi ile değerlendirdiğimizde modelin düzeyde anlamlı (p=0,000) bulunduğu ve doğru sınıflandırma oranının %92,9 ile başarılı olduğu görülmüştür. Modelde sanal gerçeklik ile ilgili bilgi sahibi, olma durumu ile BHÖ ölçeğinin tüm alt boyutları arasında anlamlı ilişki saptanmamıştır (Tablo 4.17).

**Tablo 4.18:** Deney grubundaki öğrencilerin sanal gerçeklik bilgi ve deneyim durumları ile bilişsel yük ölçeği arasındaki ilişki

| Parametre | | BYÖ* | Test İstatistiği** | р |
|---|---|---|---|---|
| Sanal Gerçeklik ile ilgili bilgi | Evet | $2,46\pm1,50$ | 1.500 | 0.140 |
| sahibi olma | Hayır | $1,65\pm1,65$ | 1,500 | 0,142 |
| Sanal gerçeklik ile ilgili | Evet | $2,66\pm2,08$ | 0.024 | 0.400 |
| uygulamaya katılma durumu | Hayır | $1,84\pm1,61$ | 0,834 | 0,409 |

<sup>\*</sup>mean±sd, \*\*Independent Sample T testi

Deney grubundaki öğrencilerin sanal gerçeklik ile ilgili bilgi durumları ve sanal gerçeklik uygulmasına katılma durumları ile BYÖ puanları arasındaki ilişki Independent-Sample T testi ile karşılaştırılmıştır. BYÖ puanları ile her bir parametre arasındaki ilişki saptanmamıştır (p=0,142, p=0,409) (Tablo 4.18).

# 4.4. DENEY GRUBUNDAKİ ÖĞRENCİLERİN DENEYİMLEDİKLERİ SANAL GERÇEKLİK UYGULAMASINDAKİ KALİTATİF GERİ BİLDİRİMLERİ

Sanal gerçeklik gözlüğünü uygulayan öğrencilere uygulama sonrası deneyimlerinin sorulduğu "Sanala gerçek uygulaması ile yaşadığınız deneyimi birkaç cümle ile tanımlayınız?" sorusu sorulmuştur. Öğrencilerin yanıtları Tablo 4.19'da gösterilmektedir.

**Tablo 4.19:** Sanal gerçeklik uygulamasını deneyimleyen öğrencilerin kalitatif geri bildirimleri

| Öğrenci<br>Kodları* | Sanal gerçek uygulaması ile yaşadığınız deneyimin geri bildirimleri |
|---|---|
| K1 | Fetal gelişimi yakından görmek bebeğin hareketlerini gözlemlemek çok çok güzeldi anlatılmaz yaşanır dedikleri bu olsa gerek 🕄 |
| K2 | Muhteşem ve çok farklı bir deneyimdi. |
| K3 | Çok güzel bir deneyimdi. Bebeğin hareketleri (tekme, gülümseme vb.) görebildik. |
| K4 | Umblikal kordu görebildik. Fetüsün hafta hafta gelişimini en yakından izleyerek deneyimlemeyi sağlayan mucizevi bir uygulama. Özellikle embriyoloji derslerinden sonra fetus gelişimini pekiştirmek adına uygulana bilinecek bir uygulamadır. |
| K5 | Bebeğin gelişimini hafta hafta izlemek gerçekten çok güzel ve heyecan vericiydi. |
| K6 | Gerçekçi bir bebek oluşumu izledim |
| K7<br>K8 | Çok gerçekçi ve bilgilendiriciydi. Daha fazla geliştirilebilecek bir uygulama. Her alanda yapılabilir ve öğretici. Teorik bilgilerin gerçekçi görsel ile pekiştirilmesini sağlıyor. Görsel olduğundan daha fazla akılda kalıcı ve eğitici |
| K9 | Sanal gerçeklik uygulamasını daha önce keşfetmemiştim. Gözlüğü taktığımda kendimi olayın merkezinde hissettim. Bu keyifli anları bize yaşattığınız için teşekkür ederim hocam. |
| K10 | Güzel bir deneyimdi görsel olarak kalıcı bir etkinliktir. |
| K11 | Anne karnında bebeğin oluşumu tam bir mucize. Bu uygulama sayesinde bizde en yakından bir mucizenin oluşumuna tanık olmuş olduk. Teşekkürler :) |
| K12 | Gözlüğü taktığım andan itibaren büyülendim diyebilirim. Fetal gelişimi ilk haftalardan itibaren anne karnında gözlemleyebilmek ve istediğimiz haftaya dönüp tekrar izleyebilmek çok güzeldi ve çok gerçekçiydi. Muhteşem bir çalışma olmuş |
| K13 | Farklı ve etkili bir deneyimdi. |
| K14 | Çok güzel bir duygu ve histi. Sanki gerçekten o an fetüsle birlikte büyüyüp küçüldüğünü hissediyorsun. Bence kesinlikle her ebelik öğrencisinin yaşaması gereken bir an. Derste tabi ki bu evreleri teorik olarak öğreniyoruz ama sanki canlıymış gibi görmek mükemmeldi. |
| K15<br>K16 | Anne karnındaki bebeğin haftalara göre gelişimini çok yakından izlemek beni oldukça mutlu etti. Çok şaşırtıcı ve büyüleyiciydi. Bu duyguyu hiçbir zaman unutmayacağım. Çok güzeldi ve herkesin deneyimlemesi gerekli |
| K17 | Sanal gerçekliği ilk kez deneyimledim çok etkileyiciydi. Gözlüğü taktığım andan itibaren kendimi olayın tamamen içerisinde hissettim. Her şey çok gerçekçiydi ve çok güzel bir deneyimdi. Bu güzel deneyimi bize yaşattığınız için teşekkür ederim hocam. |
| K18 | İlk kez böyle bir deneyim yaşadım, etkileyiciydi. |
| K19 | Çok etkileyici bir deneyimdi |
| K20 | Harika, sanki o anı kendim yaşıyor gibi hissettim. |
| K21 | Güzel ve gerçeğe yakın bir deneyimdi Teşekkürler reyhan hocamıza |
| K22<br>K23 | Muhteşem bir deneyimdi. Gerçeğe en yakın bu kadar başarılabilirdi. Çok güzel bir tecrübeydi benim için. Çok teşekkürler Muhteşem bir deneyimdi. Çok güzel bir tecrübeydi benim için. |
| K24 | Bize bu güzel deneyimi yaşattığınız için teşekkür ederim hocam çok güzel bir deneyimdi |
| K25 | Sanal gerçeklik uygulaması çok güzeldi. Gerçekliğin yanı sıra duygusal bir anı olarak kaldı. Fetüse bu kadar yakın hissetmek çok güzel bir duyguydu |
| K26 | Uygulama çok gerçekçiydi ve kolay kontrol edilebilirdi. Hafta hafta bilgilerin geçmesi ve duyulan seslerin gerçekliği güzeldi. Sanal ortam kolay uyum sağlanabilirdi ve rahatsız |
| K27 | edici bir özellik yoktu. Deneyimlememizi sağladığınız için teşekkürler. Sanal gerçeklik uygulaması ile gerçekten anne karnındaymışım gibi hissettim. Bebeğin gelişim aşamalarını en yakından yanı yanından takip edebildim. Çok güzel bir uygulama olmuş hocamızın ellerine sağlık |

Tablo 4.19 (devam)

| K28 | Her şey gerçek gibiydi bebeğin gelişimine bu kadar yakından şahit olmak harikaydı. |
|---|---|
| K29 | Gerçekten çok güzel bir deneyimdi sanki bebekle birlikte bizde anne karnındaydık. |
| K30 | Tek kelimeyle mükemmeldi. Sanki bebek anne karnında değil de benim hemen yanımda büyüyor gibiydi. Bütün organları hafta ilerledikçe daha da belirginleşiyor ve her şey net oluyordu. Yüzündeki hareketlere kadar her şey çok netti. Gelişimle birlikte kalp seslerini dinlemek de çok güzeldi. Kesinlikle bütün ebelik öğrencilerinin, anne ve babalarında deneyimlemesi gerekiyor. Reyhan hocamızda bize böyle bir fırsat sunduğu için ona da çok teşekkür ederim. Gerçekçi bir deneyimdi |
| K32 | Çok güzel ve etkileyici bir deneyim oldu sanki gerçek gibi annenin karnında bebeği ile büyümüş gibi oldum |
| K33 | Anne karnında fetüsün gelişimine canlı şahit olmak mükemmel bir şey |
| K34 | Fetal gelişmesini canlı öğrenmiş oldum Reyhan hocamıza çok teşekkür ediyorum |
| K35 | Yani anne ve baba adayları ön bilgilendirmede için çok güzel bir uygulama |
| K36 | Çok güzel deneyimdi benim için yaratıcı gerçek gibiydi |
| K37 | Çok gerçekçi ve bilgilendiriciydi. Teorik bilgilerin pekişmesini sağladı. |
| K38 | Çok farklı ve yararlı bir deneyimdi. Çok mutlu oldum teşekkürler hocam 😉 |
| K39 | Güzel deneyimdi hocama teşekkür ederim |
| K40 | Çok güzel bir uygulamaydı. İlk defa böyle bir deneyim yaşadım o yüzden çok teşekkür ederim \iint |
| K41 | Mükemmel bir çalışma olmuş. Gerçekten anne karnında bebeğin gelişimini izliyor gibi hissettim. Haftalar arasında geçiş yaparak izleyebilmekte oldukça iyiydi. |
| K42 | Çok yararlı ve faydalı herkesin izlemesi gerekli teşekkürler hocam 🤤 |

<sup>\*</sup>K harfi katılımcıyı temsil etmektedir.

Sanal gerçeklik teknolojisi ile oluşturulmuş fetal gelişim uygulamasını deneyimleyen öğrencilerin olumlu geri bildirim verdikleri görülmüştür. Öğrencilerin geri bildirimleri arasında, diğer derslerde de SG uygulaması kullanmanın dersi anlamalarına olumlu katkı sağlayacağı ifadeleri yer almıştır. Fetal gelişimi SG uygulaması ile yakından izlemenin öğrenciler üzerinde olumlu bir etki bıraktığı görülmüştür.
### 5. TARTIŞMA

Sanal gerçeklik teknolojisi ile fetal gelişim uygulaması (SGT-FEGU)'nun etkinliğinin değerlendirildiği çalışmada, bulgular literatür bilgileri ışığında;

- 1. Deney ve kontrol grubundaki öğrencilerin sosyo-demografik özelliklerinin tartışılması,
- 2. Deney ve Kontrol grubundaki öğrencilerin öğretim materyallerine (Teori eğitimi ve SG uygulaması) ilişkin bilgi düzeylerine ait bulguların tartışılması,
- 3. Deney grubundaki öğrencilerin sanal gerçeklik uygulamasına ait bilişsel yük ve bulunuşluk hissi düzeylerine ait bulguların tartışılması,
- 4. Deney grubundaki öğrencilerin deneyimledikleri sanal gerçeklik uygulamasındaki kalitatif geri bildirimlerine ait bulguların tartışılması olmak üzere dört alt başlık altında sunulmuştur.

## 5.1. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN SOSYO-DEMOGRAFİK ÖZELLİKLERİNİN KARŞILAŞTIRILMASI

Öğretimde öğrenme stilleri yada yeni tip öğrenme modelinden etkileyen faktörlerin arasında yaş, öğrenim görülen bölüm ve sınıf değişkeni yer almaktadır (135–140). Benzer şekilde de ebelik simülasyon eğitimi etkinliğinin incelendiği çalışmalarda da bu değişkenler yer almış ve değişkenlerin homojenliği sağlanmıştır (117, 141–143). Hemşirelik ve Tıp eğitiminde sanal gerçeklik uygulamalarının etkinlerinin araştırıldığı çalışmalarda da yaşın homojen dağıldığı görülmüştür (144–151). Araştırmada uygulanan yeni öğretim tekniği olan SGT-FEGU'nun uygulandığı öğrenci grubunda bu parametrelerin homojenliği sağlanmıştır. Araştırmada deney grubundaki öğrencilerin yaş ortalaması 22,38±0,88, kontrol grubundaki öğrencilerin yaş ortalaması 22,54±0,88 olarak saptanmıştır. Araştırmada grupların yaş değişkeni arasında benzer dağılım gösterdiği ve aralarında anlamlı fark olmadığı görülmüştür (p>0,05). Literatür ebelik öğrencilerinin simülasyon etkinliğinin incelendiği çalışmalarda da öğrencilerin yaş ortalamasının, araştırma ile benzer olduğu görülmüştür (117, 141–143, 152, 153).

Eğitimde öğrenme stillerine etki eden diğer parametrelerden biri de öğrencinin akademik başarısı olduğu görülmüştür (135–140). Öğrenme stillerinin farklı olması akademik başarıyı, akademik başarıda öğrenme stillerini etkilemektedir. Araştırmada öğrencilerin akademik başarıları okudukları yıldaki Ağırlıklı Genel Not Ortalaması (AGNO) puanları incelenerek değerlendirilmiştir. Deney grubundaki öğrencilerin AGNO puanları 2,94±0,36, kontrol grubundaki öğrencilerin ise 2,88±0,45 olarak saptanmıştır. Literatür incelendiğinde öğrencilerin akademik başarı değişkeninin homojen dağılım gösterdiği saptanmıştır (145, 154, 155). Araştırmada benzer şekilde öğrencilerin AGNO puanları arasında homojen dağılım görülmüş ve anlamlı fark saptanmamıştır (p>0,05).

Araştırmada öğrencilerin yaşadığı yer, ebelik mesleğini tercih etme sırası ve mezun olduktan sonraki planları incelenmiştir. Öğrencilerin bu parametreleri arasında anlamlı ilişki saptanmamıştır (p>0,05). Öğrencilerin bu parametrelerinin homojen dağılım gösterdiği, deney ve kontrol gruplarında eşit dağılım gösterdiği görülmüştür.

Öğrencilerin bilgisayar kullanımı ile daha önce SG uygulaması deneyimleme durumları kullanılacak SG uygulaması kullanımı etkilemektedir. Bu değişkenlerin deney ve kontrol grubunda homojen olarak dağılması çalışmayı deneyimleyenlerin sonuçları üzerinde etkilidir. Literatürde bu değişkenlerin homojenliğinin sağlandığı görülmüştür (154, 156) Butt ve ark. (154), hemşirelik öğrencilerinin hasta güvenliğini sağlarken temel becerileri geliştirmelerinde SG uygulamasının etkinliğini inceledikleri çalışmalarında öğrencilerin bilgisayar kullanımlarının ve SG deneyimlerinin gruplar arasında homojen dağılım gösterdiği görülmüştür. Stepan ve ark. (156) tıp öğrencilerinde SG'nin nöroanatomi eğitimi üzerindeki etkinliğini saptamak amacıyla yaptıkları randomize kontrollü çalışmalarında, öğrencilerin bilgisayar kullanımı sıklığının ve SG uygulama deneyimlerinin homojen olduğu görülmüştür. Araştırmada deney ve kontrol grubundaki öğrencilerin bilgisayar oyunu oynama durumları ve sıklığı, SG ile ilgili bilgi sahibi olma durumları ve daha önce SG uygulaması deneyimlerinin homojen dağılım gösterdiği, aralarında anlamlı fark saptanmadığı görülmüştür (p>0,05). Araştırma literatür ile benzerlik göstermektedir.

Araştırmada deney ve kontrol gruplarının bağımsız değişkenleri binary lojistik regresyon puanları incelenmiştir. Modelde bu değişkenler arasında anlamlı ilişki görülmemiştir. Bu durumun deney ve kontrol grubundaki homojenliğin sağlandığından kaynaklanmıştır. Literatürle uyumluluk göstermiştir (144–148, 154, 156, 157).

## 5.2. DENEY VE KONTROL GRUBUNDAKİ ÖĞRENCİLERİN ÖĞRETİM MATERYALLERİNE (TEORİ EĞİTİMİ VE VR UYGULAMASI) İLİŞKİN BİLGİ DÜZEYLERİNE AİT BULGULARIN TARTIŞILMASI

Araştırmada ebelik öğrenci için oluşturulmuş, fetal gelişimin öğretimi için tasarlanmış sanal gerçeklik platformu olan SGT-FEGU kullanılmıştır. Ebelik alanından fetal gelişim öğretiminde benzer sanal gerçeklik uygulaması sadece Jones ve ark.'ları tarafından oluşturulmuş "road to birth" uygulaması olduğu görülmüştür (114, 158). Literatürde fetal gelişim öğretimi için arttırılmış gerçeklik ve 3D modelleme gibi uygulamaların kullanıldığı görülmüştür (34, 133). Fetal gelişimi öğretiminde sanal gerçekliğin SG uygulamalarının literatürde kısıtlı olması nedeniyle geliştirilen SGT-FEGU hemşirelik ve tıp fakültesi alanlarında geliştirilen ve uygulanan diğer eğitim modelleri ile tartışılmıştır (42, 144–151, 154–157, 159–167).

Tsai ve ark. (144), hemşirelerin port katater yerleştirme becerilerini iyileştirmek için geliştirdikleri, 43 deney ve 49 kontrol grubunun bulunduğu randomize kontrollü çalışmalarında, SG ortamından port katater eğitiminin hemşirelerin post katater becerini geliştirilmesinde etkili olduğu görülmüştür. Çalışmada deney grubuna 40 dakika süren SG uygulaması ile port katater eğitimi verilmiştir. Kontrol grubundaki katılımcılara da geleneksel hemşirelik eğitimi verilmiştir. Uygulama sonrasında ve uygulamadan üç hafta sonra son test puanları incelenmiştir. Uygulama sonrası SG destekli simülasyon eğitimin post katater takımında uygulanabilir yöntem olduğu görülmüştür.

Gu ve ark. (145), lisans hemşirelik öğrencileri için hemşirelik esasları dersi kapsamında geliştirdikleri SG destekli eğitim programlarını 14 deney ve 14 kontrol olmak üzere 28 öğrenci ile randomize kontrollü bir şekilde uyguladıkları çalışmalarında, SG destekli uygulamanın standart ders prosedürüne oranla daha etkili olduğu görülmüştür. Çalışmada öğrencilere meslek esasları kapsamında kateter bakımı, asepsi antisepsi teknikleri ile ilaç tedavisi içeren vaka uygulamaları öğretilmiştir. Uygulama sonrası 100 puan üzerinden son test bilgi testi ile değerlendirilmiştir. Deney ve Kontrol grubunun son test puanları sırasıyla, 73,31±9,27 ve 55,36±8,93 olarak saptanmıştır. Deney grubunun kontrol grubuna oranla daha yüksek puan aldığı ve vaka yönetiminde daha başarılı oldukları görülmüştür.

Liaw ve ark. (146), sanal hasta simülasyonunun gelişimini tanımlamak ve etkinliğini değerlendirmek, hemşirelik öğrencilerinin değerlendirmedeki

performanslarını iyileştirmek için geleneksel bir manken tabanlı simülasyon ile karşılaştırdıkları randomize kontrollü çalışmalarında, SG temelli hasta simülasyonunun geleneksel manken simülasyonuna oranla daha etkili olduğu saptanmıştır. Çalışma 31 deney 26 kontrol olmak üzere 57 lisans öğrencisi ile yapılmıştır. Eğitim 2 saat süre ile uygulanmış, eğitim sonrası ve eğitimden 8 hafta sonra son test ile etkinlik değerlendirilmiştir. Çalışmada etkinlik 19 sorundan oluşan ölçek ile değerlendirilmiştir. Deney ve kontrol grubunun ön test puanları sırasıyla, 31,52 ve 29,46; 8 hafta sonrası son test puanları ise, 33,58 ve 33,38 olarak saptanmıştır.

Jung ve ark. (147), intavenöz (IV) kateter hemşirelik uygulamasında SG ile geleneksel kol simülatörünün etkinliğini değerlendirdikleri, geleneksel kol simülatörü (Grup A, n=41), SG uygulamalı kol simülatörü (Grup B, n=40) ve hem geleneksel hem de SG uygulamalı kol simülatörünün (Grup C, n=38) kullanıldığı çalışmalarında, geleneksel kol ile SG uygulamasının birlikte kullanıldığı grubun diğer gruplara oranla daha başarılı olduğu görülmüştür. Ayrıca çalışmada sadece SG simülasyonunu kullanan grubun geleneksel gruba oranla daha başarılı olduğu görülmüştür. Öğrencilerin kaygı değerlendirilmesi görsel analog kaygı ölçeği olan VAS ile değerlendirilmiştir. Grupların VAS değerleri ön test punları Grup A 4,84±2,42, Grup B 4.14±2,22 ve Grup C 4,99±2,58 olarak görülmüştür. Grupların son test puanları ise sırasıyla, 3,38±2,60; 2,80±2,32; 2,58,2,11 olara saptanmıştır. Çalışmada grupların kendi içlerinde anksiyete puanlarının azalma göstermesine rağmen gruplar arası fark saptanmamıştır.

Cobbett ve ark. (148), anne- yenidoğan hemşireliği öğrencilerinde, sanal klinik simülasyonun yüz yüze yüksek kaliteli manken simülasyonuna göre etkinliğini inceledikleri, 42 deney ve 42 kontrol grubundan oluşan çalışmamalarında, iki uygulama arasında fark görülmemiştir. Araştırma değerlendirilmesinde öğrencilerin kaygı ve kendine güve seviyelerini ölçen anket kullnılmıştır. Deney ve kontrol grubunun eğitim sonrası kaygı puanları sırasıyla, 57,75±15,25 ve 73,26±19,95 olarak saptanmıştır. Öğrencilerin kendine güven puanalrı ise, deney grubunun 115,25±21,95, kontrol grubunda 104,89±17,52 olarak saptanmıştır. Öğrencilerin kazanım ve öz güven seviyeleri arasında fark saptanmamıştır.

İsmailoğlu ve Zaybak (149), hemşirelik öğrencilerin IV kateter takma becerilerini geleneksel model ve SG modelin etkinliğini inceledikleri, 33 deney ve 33 kontrol grubunda oluşan, randomize kontrollü çalışmalarından, doyum puanlarının ve psikomotor

becerilerinin deney grubunda daha yüksel olduğu görülmüştür. Eğitim öncesi ve sonrası bilgi puanlarının eşit olduğu ve aralarında fark olmadığı saptanmıştır. Çalışmada öğrencilerin değerlendirmesi 15 gün sonra laboratuvar ortamında maket üzerinde yapılan tek kör izlem ile değerlendirilmiştir. Ayrıca öğrencilere memnuniyet anketi uygulanmıştır. Deney grubundaki öğrencilerin memnuniyet puanları 43.89±8.70, kontrol grubunun ise 21.77±5.28 olduğu saptanmıştır.

Smith ve ark. (150), dekontaminasyon becerisini öğretmek için iki seviyeli sürükleyici sanal gerçeklik simülasyonunu (VRS) hemşirelik öğrencilerindeki etkisini saptamak amacıyla tasarladıkları, sürükleyici SG, bilgisayar destekli SG ve geleneksel eğitim olmak üzere üç gruptan oluşan yarı deneysel çalışmalarında, gruplar arası fark saptanmamıştır. Buna karşın sürükleyici SG grubunun diğer gruba oranla daha fazla etkileşimde bulunduğu ve daha fazla aktif olduğu görülmüştür. Çalışmada iki grup arsında fark 20 sorudan oluşan ve araştırmacılar tarafından hazırlanan maksimum puanı 20 olan anket formu ile ön test ve 6 ay sonra son test olarak değerlendirilmiştir. Sürükleyici SG, bilgisayar destekli SG ve geleneksel gruplarının ön test puanları sırasıyla, 8,78±0,39, 9,47±0,29 ve 9,38±0,29 olarak, son test puanları ise, sırasıyla, 14,19±0,33, 14,24±0,34 ve 14,25±0,33 olarak saptanmıştır.

LeFlore ve ark. (151), hemşirelik öğrencilerinde SG ile pediatrik solunum bakımının etkinliğini inceledikleri, 46 deney 47 kontrol grubunda oluşan randomize kontrollü çalışmalarında, SG uygulaması ile verilen eğitimin teori dersine oranla daha iyi bir öğrenme yöntemi olduğu saptanmıştır. Çalışmada değerlendirme araştırmacılar tarafından geliştirilen pediatrik solunum bakımının parametrelerini içeren değerlendirme aracı ile ölçülmüştür. Ölçüm süre olarak yapılmıştır. Test sonrası deney be kontrol grubunun işlem süreleri karşılaştırılmıştır. Deney grubu müdahaleyi 7,0±1,5, kontrol grubunun ise 10,3± 5,4 saniyede tamamladığı görülmüştür. İki ölçüm arasında anlamlı fark saptanmıştır.

Healing (155), kronik akciğerli bir hastanın bakımının SG ve manken tabanlı simülasyonda maliyet etkinliğini incelediği randomize kontrollü çalışmada, SG temelli simülasyonun maket tabanlı simülasyona oranla daha az maliyetli olduğu saptanmıştır. Araştırmada maliyet; okuldaki kişi sayısı, fakültede bulunma zamanları, laboratuvarda bulunan kişi sayı ve senaryo giderleri ele alınarak hesaplanmıştır. Çalışmada öğrencilerin

eğitim sonrası nicel ölçümlerinde bir farklılık olmazken, nitel geri dönüşlerde SG temelli eğitimin daha yaralı olduğu görülmüştür.

Butt ve ark. (154), hemşirelik öğrencilerinde, üriner kateterizasyon uygulamak için tasarlanmış oyun tabanlı bir SG sisteminin kullanılabilirliğini inceledikleri, 10 deney, 10 kontrol grubundan oluşan randomize kontrollü çalışmalarında, uygulamanın etkin olduğunu ve hemşirelik eğitiminde kullanılabileceğini saptamışlardır. Araştırma deney ve kontrol grubu ürüner kateter takma sürelerine ve prosedürleri tamamlama durumlarına göre değerlendirilmiştir. Çalışmada SG grubunun (25,3 saniye) kontrol grubuna (14,9 saniye) oranla daha uzun sürede kateter taktığı saptanmıştır. Buna rağmen SG grubun 3,9'unun, kontrol grubunda ise 1,8'inin prosedürü tamamladığı görülmüştür.

Bryant ve ark. (159), hemşirelik öğrencilerinde, SG klinik ortamının etkinliğini inceledikleri, 22 deney, 38 kontrol grubundan oluşan randomize kontrollü çalışmalarında, hazırlana SG klinik ortamı ile geleneksel öğrenme yöntemi arasında anlamlı fark olmadığı görülmüştür. Çalışmada deney grubundaki öğrencilere 7 hafta süren eğitim verilmiştir. Eğitimin etkinliği dönem sonu müfredat dahilinde yapılan, vaka çözümlemeyi içeren genel sınav ile değerlendirilmiştir. Sınavdan 100 üzerinden 80 puan alan öğrenciler başarılı olarak görülmüştür. Deney grubunun dönem sonu puanları 46,96±12,11, kontrol grubunun puanları 52,63±14,27 olarak saptanmıştır. Çalışmada SG klinik ortamı öğrenci memnuniyetinden dolayı ek bir eğitim aracı olarak önerilmiştir.

Stepan ve ark. (156), Tıp öğrencilerinde 3D modelleme ile interaktif SG anatomi modelinin etkinliğini karşılaştırdıkları, 33 deney, 33 kontrol grubunda oluşan randomize kontrollü çalışmalarında, iki grup arasında anlamlı fark görülmemiştir. Her iki modelinde aynı ölçüde etkin olduğu saptanmıştır. Araştırmada ölçme aracı olarak araştırmacılar tarafından hazırlana 40 sorudan oluşan analog skala kullanılmıştır. Soru formundan alınacak en düşük puan 0, en yüksek puanınsa 100 olarak alınmıştır. Deney ve kontrol grubuna 8 hafta sonra son test uygulanmıştır. Deney ve kontrol grubunun uygulamadan memnun kalma ve eğlenceli bulma durumlarına ilişkin punaları sırasıyla, 72,35±19,68 ve 15,67±14,19 olarak saptanmıştır. Çalışmada SG grubundaki öğrencilerin daha olumlu deneyim ve motivasyona sahip oldukları görülmüştür.

Soylar ve ark. (160) tarafından, tıp fakültesi öğrencilerinde, Lockheed Martin (168) tarafından geliştirilen bir sanal gerçeklik cihazı olan Endoskopik Sinüs Cerrahisi Simülatörü (ES3)'nün eğitim ve öğretimde etkinliğini inceledikleri çalışmalarında, ES3

grubu ile ders kitabı eğitim grubunun kendi içlerinde ön test ve son test puanların anlamlı ilişki görülmüştür. Araştırmada gruplar arası fark araştırmacılara tarafından hazırlana 5'li likerttipte olan 10 soru ile değerlendirilmiş ve ortama puanlar alınarak hesaplanmıştır. Deney ve kontrol grubunun ön test puanları sırasıyla, 6,9±1,2 ve 6,7±1,5 son test puanları ise 9,4±0,5 ve 5,1±3,0 olarak saptanmıştır. Gruplar arası fark incelendiğin de ilişkinin anlamsız olduğu görülmüştür. Buna rağmen ES3 grubundaki öğrencilerin olumlu geri dönüşleri olduğu bildirilmiştir. ES3'ün sinonazal eğitimde etkin bir eğitim aracı olarak kullanılabilir olduğu saptanmıştır.

Mikelus ve ark. (161), tıp fakültesi öğrencileri ve asistanları için, anatomide sanal gerçeklik robotik cerrahi simülatörünün (RoSS)'nün etkinliğini inceledikleri çalışmalarında, RoSS'un teori eğitime oranla daha etkin bir öğrenme aracı olduğu görülmüştür. Çalışmada eğitimin etkinliği süre olarak ölçülmüştür. RoSS üzerinde eğitim alan grup cerrahi işlemi 118 saniye tamamlarken, sadece müfredata uygun eğitim alan grup 143 saniyede tamamlamıştır. İki grup arasında anlamlı ilişki görülmüştür.

Moro ve ark. (162), Tıp fakültesi öğrencilerinde, SG, AR ve 3D tablet uygulamalarının etkinliğini inceledikleri, randomize kontrollü çalışmalarında, AR ve SG uygulamaları ile verilen anatomi eğitiminin mevcut eğitimden daha fazla etkili olduğu görülmüştür. Çalışmada her grupta 59 öğrenci alınmıştır. Öğrencilerin değerlendirilmesi araştırmacılara tarafından hazırlanan 20 soruluk çoktan seçmeli anket ile yapılmıştır. Puanlama 100 puan üzerinden yapılmıştır. SG, AR ve 3D tablet uygulama grubunun son test puanları sırasıyla; %64,5, %62,5 ve %66,5 olarak saptanmıştır. Öğrencilerin değerlendirmeleri son test puanları üzerinden yapılmıştır. Sanal gerçeklik grubundaki öğrencilerde baş dönmesi ve baş ağrısı yaşandığı görülmüştür.

Khot ve ark. (163), anatomi öğretiminde temel eğitim, manken model ve SG uygulamasının etkinliğini incelediği, her bir grupta 20 tıp öğrencisinin yer aldığı randomize kontrollü çalışmalarında, SG eğitimi temel eğitim ve maket model ağitimi arasında anlamlı fark görülmemiştir. Araştırmada eğitimin etkinliği araştırmacılar tarafından hazırlana 15 çoktan seçmeli, 10 fonksiyonel olmak üzere 25 soru ile değerlendirilmiştir. Öğrencilerin test performans değerleri %95 güven aralığı üzerinden verilmiştir. Maket model, klasik öğretim ve SG grubunun çoktan seçmeli son test puanları sırasıyla; %65, %40 ve %45 oranında, fonksiyonel son test cevapları ise, %25, %20 ve

%25 olarak bulunmuştur. Çalışmada anatomik modellerin diğer modellere oranla daha etkili olduğu görülmüştür.

Codd ve Choudhury (164) Önkol Kas-İskelet Sistemi öğretiminde SG (model grubu) eğitimi etkinliğini inceledikleri çalışmalarında SG tekniğinin mevcut teori eğitimine oranla daha etkin olduğu görülmüştür. Çalışmada deney grubuna (n=12) 3D modelleme ile hazırlanmış SG eğitimi 30-50 dakika arasında uygulanmıştır, geleneksel eğitim grubuna (n=13) ise yalnızca e-kaynak olarak teori eğitimi verilmiş ve kontrol (n=14) grubuna hiçbir eğitim verilmemiştir. Araştırmanın etkinliği 10 sorudan oluşan, araştırmacılara tarafından hazırlanmış ve 0-10 arasında puanlanan soru formu ile değerlendirilmiştir. Eğitim sonrası kontrol grubunun puanı 1-2 puan arasında, SG ile eğitim alan grubun puanı 7-8 puan arasında ve geleneksel eğitim alan grubun ise 6-7 puan arasında olduğu görülmüştür. Araştırmada SG eğitimi etkili bulunmasına rağmen araştırmacılar SG uygulamasını teori eğitimine ek olarak verilmesi görüşünü önermiştir.

Ellington ve ark. (165), kadın kemik pelvis kemiği eğitiminin öğretiminde SG ve müfredat eğitiminin karşılaştırıldığı, deney grubunda 15 kontrol grubunda 16 tıp fakültesi öğrencisinin yer aldığı randomize kontrollü çalışmasında, iki eğitim karşılığında anlamlı fark görülmemiştir. Çalışmada deney grubuna 10 dakika SG modelli kadın pelvis kemiği eğitimi verilirken, kontrol grubuna müfredat eğitimine uygun bir eğitim uygulanmıştır. Eğitim etkinliği ön test ve son testte, araştırmacılar tarafından hazırlanan, çoktan seçmeli 28 sorudan oluşan anket ile değerlendirilmiştir. Ankette alınacak en düşük puan 0 en yüksek puan ise 100 olarak belirlenmiştir. Deney ve kontrol grunundaki öğrencilerin ön test puanları sırasıyla; 74,3±8,8 ve 70,5±13,5, son test puanları ise 83,0±7,8 ve 78,6±13,3 olarak saptanmıştır. SG eğitimindeki deney grubunun eğitim puanlarında önemli bir artış görülmemesine rağmen uygulamanın öğrenciler tarafından olumlu algılandığı görülmüştür.

Chang ve ark. (42), sezaryen ve normal doğumun hemşirelik öğrencilerine video tabanlı sanal gerçeklik eğitimi (VTSG) ile müfredat uygun video eğitimin etkinliğini inceledikleri çalışmalarında, VTSG ile öğrenen öğrencilerin kontrol grubuna oranla daha başarılı oldukları görülmüştür. Çalışma 32 deney 32 kontrol grubu olmak üzere yarı deneysel olarak tasarlanmıştır. VTSG ve rutin müfredata uygun videolar eğitim öğrencilere 16 hafta boyunca haftada 3 saat toplamda 48 saatlik bir eğitim platformu oluşturulmuştur. Eğitim sonrası her iki gruptaki öğrencilere ön ve son test değerlendirme

yapılmıştır. Yapılan değerlendirme için 20 çoktan seçmeli soru kullanılmıştır. Öğrencilerin en çok 100 en az 0 puan alabilecekleri puanlama sistemi kullanılmıştır. Deney ve kontrol grubundaki öğrencilerin etkinliği ancova analiziyle değerlendirilmiştir. Ancova sonuçlarına göre öğrencilerin ön test etkinliğinden arındırılmış son test puanları, deney grubu 85,57, kontrol grubunun ise 79,02 olarak saptanmıştır. Öğrencilerin son test puanları arasında anlamlı ilişki görülmüştür. Çalışmada VTSG ile öğrenen öğrencilerin daha iyi olduğu, hemşirelik öğrencilerini geliştirmek için bu güçlü ortamın potansiyelinin doğum eğitimi bağlamında öğrenme performansını arttırdığı görülmüştür.

Pratiwi ve ark. (169), ebelerin rahim içi araç (RİA) uygulamalarında SG etkinliğini inceledikleri, 30 deney, 30 kontrol grubunun olduğu yarı deneysel çalışmalarında, RİA uygulamasında SG uygulamasının geleneksel eğitime oranla etkin oldu görülmüştür. Çalışmada deney grubundaki ebelere uygulanan SG uygulaması 11 dakika sürmüştür. Eğitim öncesi ve sonrası, araştırmacılara tarafından hazırlanan, puan aralığı 0-100 arasında değişen test uygulanmıştır. Deney ve kontrol grubundaki ebelerin ön test puanları sırasıyla; 48,24±6,03 ve 55,93±15,77, son test puanları ise 73,27±7,87 ve 84,93±7,57 olduğu görülmüştür. Kullanılan SG uygulamasının ebelerin ve ebelik öğrencilerin aile planlaması eğitiminde kullanılabilecek bir yöntem olduğu görülmüştür. Ayrıca uygulamanın pandemi durumlarında da etkin kullanılabilecek bir yöntem olduğu vurgulanmıştır.

Araştırmanın bulguları literatür ile uyumlu görülmüştür. Çalışmamızda deney grubundaki öğrencilerin ön test ve son test puanları arasında anlamlı fark görülmüştür. Kontrol grubun ön test ve son test puanları arasında ise anlamlı fark saptanmamıştır. Grupların ön test puanları benzer olduğu görüldüğünden, yapılan ancova analizinde gruplar arası fark anlamlı bulunmuştur. Fetal gelişim öğretiminde araştırma kapsamında geliştirilen SGT-FEGU'nun etkin bir araç olduğu ve güvenli bir şekilde müfredat eğitimine ek olarak kullanılabileceği görülmüştür.

Bu sonuçlar doğrultusunda araştırmada "Fetal gelişimin öğretiminde SGT-FEGU uygulamasının etkisi vardır." hipotezinin doğrulanmıştır.

## 5.3. DENEY GRUBUNDAKİ ÖĞRENCİLERİN SANAL GERÇEKLİK UYGULAMASINA AİT BİLİŞSEL YÜK VE BULUNUŞLUK HİSSİ DÜZEYLERİNE AİT BULGULARIN TARTIŞILMASI

Bilişsel yük kavramı ilk olarak Sweller (170) tarafından çoklu öğrenme ortamlarında dikkat edilmesi gereken önemli bir kavram olarak tanımlanmıştır. İyi geliştirilmiş bir sanal öğretim materyali kullanıcının bilişsel yükünü yönetebilmeli, öğrenme performansını da arttırmaya yardımcı olmalıdır (74, 171, 172). İnsan beyni kısa ve uzun süreli olmak üzere iki bellek kullanır. Bilişsel yük kuruma uzun süreli bellek ile ilişkili bir kavramdır. Öğretimde oluşturulan işitsel ve görsel bilgiler uzun süreli bellek ile iletişime girdiğinden bilişsel yük ortaya çıkar. Eğitim için geliştirilin modellerde kısa süreli bellek ile uzun süreli bellek eş zamanlı işlenmeli, bu sayede de çalışma belleğine düşen yük azaltılmalıdır (74, 173). Bilişsel yükte yük oluşturan unsurlar uygulamayı kullanan kişinin önemsemeyi gerektiği nesnelerin sayısıdır. Nesnelerin sayısı arttıkça öğrenen tarafından işlenmesi gereken bilgi sayısı da artacak ve böylece bilişsel yük de artacaktır (74).

Çalışan bellek kapasitesi sınırlıdır. Belleğe yüklenen bilginin ve örüntülerin artması bilişsel yükü arttırarak öğrenme ve hatırlama süreçlerini olmuşuz etkileyecektir. Bu sebeple bilişsel yük kapasitesini arttırmayacak öğretim metotlarının geliştirmesi gerekmektedir. Öğrenme metodundaki bilişsel yük düzeyi tekniğin başarısı üzerinde ilişkilidir. Sunulan bilgi miktarının da fazla olması bilişsel yükü arttıracak, böylece öğrenme sürecini de etkileyecektir (74, 174).

Bilişsel yükü arttıran bu faktörlere rağmen, özellikle öğrencilerde bilgisayar kullanımının yaygın olması, video oyun oynama sıklığının fazla olması ve bir çok işi aynı anda yapabiliyor olması azaltan faktörler arasında görülmektedir (74). Literatürdeki güncel çalışmalarda da bu azaltan faktörlerin etkileri doğrultusunda, AR ve SG gibi çoklu ortam kullanıcılarının eğitim sonrası bilişsel yüklerinin oluşmağı görülmüştür (74, 175–180).

Du ve ark. (181) optik başa monte ekranlı (OHMD) öğrenme simülasyonunun etkinliğini saptamak amacıyla, 15 öğrenciyi kapsayan ve beş senaryodan oluşan uygulamalarından, öğrencilerin bilişsel yük puanlarının düşük olduğu ve senaryolar ile bilişsel yük puanların arasında ilişki saptanmadığı görülmüştür. Öğrencilerin 5 senaryo

için bilişsel yük puanlarının sırasıyla;  $5,47\pm1,55$ ;  $5,20\pm1,55$ ;  $5,20\pm1,46$ ;  $4,73\pm1,43$ ;  $4,53\pm1,30$  olarak saptanmıştır.

Timar (182), duygusal tasarımlı çoklu ortam değerlendirme materyalinin öğrencilerin üzerindeki bilişsel yük ve motivasyon durumunu incelediği, 159 deney, 147 kontrol grubunun yer aldığı, doktora tezinde, öğrencilerin BYÖ puanları arasında anlamlı fark saptanmamıştır.

Park ve ark. (183), çoklu ortam öğrenmenin bilişsel ve duygusal etkilerini inceledikleri, iki modelden ve altı yapıdan oluşan, 123 öğrenciyi kapsayan çalışmamalarında, öğrencilerin altı yapı arasındaki BYÖ puanlarının ilişkili olmadığı görülmüştür. Öğrencilere uygulanan çoklu ortamın modellerinin bilişsel yük oluşturmadığı saptanmıştır. Öğrencilerin altı alt boyuttan aldıkları BYÖ puanları sırasıyla; 4,75±0,96; 4,26±0,89; 4,35±0,73; 4,03±1,15 ve 4,06±0,75 olarak bulunmuştur.

Plass ve ark. (184) çoklu ortam öğrenmede duygusal tasarı modelinin etkinliğini inceledikleri, 121 öğrenciyi kapsayan çalışmamalarında, BYÖ puanları ile model anlamlı ilişki saptanmamıştır. Katılımcıların BYÖ puan ortalamasının 5,46 olduğu görülmüştür.

Um ve ark. (185), multimedya öğrenmesinin bilişsel yük durumunu inceledikleri, 118 kişiyi inceledikleri çalışmalarında, oluşturdukları çoklu ortamda duygusal öğrenme modelinin katılımcılarda bilişsel yük oluşturmadığını saptanmıştır. Katılımcıların bilişsel yük ortalama puanlarının 7,52 olduğu görülmüştür. Modelde olumlu ruh hali olan öğrencilerin BYÖ puanlarının nötr ruh hali olan öğrencilere oranla daha yüksek olduğu görülmüştür.

Araştırmada deney grubundaki öğrencilerin BYÖ ortalama puanları 1,09±0,29 olarak bulunmuştur. Bu sonuç literatür ile uyum göstermektedir. Ölçek puanın düşük olma nedenlerinin, öğrencilerin ilk defa SG gözlüğü ile fetal gelişimi izlemeleri, heyecanlı olmaları ve merak duymaları olduğu düşünülmektedir.

Bu sonuçlar doğrultusunda SGT-FEGU'nun kullanan öğrencilerinde bilişsel yük oluşturmadığı saptanmıştır. Araştırmada belirlenen "Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilere bilişsel yükü yoktur." hipotezi kabul edilmiştir.

Araştırmada öğrencilerin uygulama içerisine entegre edilen hologramik saati sorunsuz kullandığı gözlemlenmiştir. Bu gözlem sonucunda araştırma hipotezlerinden, "Fetal gelişimin öğretiminde SGT-FEGU uygulaması deneyiminde kontrol ve görsel ara

yüzlerin etkisi yoktur." ve "Fetal Gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin görsel, işitsel ve dokunsal olarak algılamasına etkisi yoktur." Hipotezleri kabul edilmiştir. Öğrencilerin uygulamayı aktif kullanmasının, sürekli bilgisayar kullanıyor olmaları ve online derste aktif birçok platformu kullanmalarından kaynaklandığı düşünülmüştür.

Bulunuşluk hissi, sanal ortamda gerçek dünyaymış gibi zamansız olarak yaşanma hissi olarak tanımlanabilir (186–188). Bir başka ifade ile bulunuşluk hissi, sanal gerçeklik ortamında bulunan kişinin kendisini içinde olduğu ortamda hissetmesini ve o ortama inanmasıdır.

Bulunuşluk hissi ile oluşan çevrenlenme ya da çevreleyen hissinde, kişiler SG'de içinde bulunduğu ortamda yoğun duygular yaşamakta ve kedilerini o ortamın içerisinde bulunuyormuş gibi hissedebilirler (189, 190).

Bulunuşluk hissi ile oluşan çevrelenme duygusu SG kullanan kişilere bulundukları ortamın bir parçasıymış hissiyatı sağlar. Bu şekilde de kişi içinde bulunduğu SG ortamını gerçek dünyaymış gibi algılar (191). Bu süreçte de bulunuşluk hissi ile çevrelenmiş duygusunu arttırarak deneyimleyenlerin öğrenme çıktılarını arttırmaktadır. Literatür incelendiğinde SG kullanıcıların ortam katılımı arttırıldıkça oluşan uygulamanın çevrelenme özelliği artarak öğrenmeyi motive ettiği ve arttırdığı görülmüştür (188, 192–194).

Öğrenme sürecinde kullanıcı SG ortamında kendini ne kadar var olmuş hissederse bilginin o kadar kalıcı olduğu görülmüştür(121, 192, 193, 195–198).

Servotte ve ark. (199) lisans sağlık eğitimi alan öğrenci (n:42) ile lisans üstü öğrencilerin (n:19) buradalık duygusunu etkileyen unsurları saptamayı amaçlayan, toplu kazazede olayı-kapsayıcı simülasyona çalışmasında, bulunuşluk hissi yüksek olan katılımcıların eğitim çıktılarının daha yüksek olduğu saptanmıştır.

De leo ve ark.(197), 29 üyeden oluşan 3 Hava Kuvvetleri Ulusal Muhafız Sağlık Hizmeti seferi tıbbi destek ekibiyle gerçekleştirdikleri, katılımcıların kullanıcı özellikleri ve varlık duygusu derecesine ilişkin geriye dönük bir araştırma sonrası gözlemsel bir çalışmada, SG ortamının etkisini arttırmak için bulunuşluk hissinin ve varlık duygusunun yüksek olması gerektiğini saptamıştır. Çalışmada bulunuşluk hissisinin öğrenme üzerinde olumlu etkisi olduğu vurgulanmıştır.

Kılıç (187), SG ortamında içmimarlık eğitim modelini oluşturduğu doktora tezinde, katılımcıların genel bulunuşluk puan ortalaması 5 üzerinden 4,29 olarak bulunmuştur. Bu sonuç doğrultusunda uygulamaya katılan kişilerin yüksek oranda bulunuşuk hissine sahip olduğu görülmüştür. Bununla beraber uygulamaya katılan öğrencilerin genel BHÖ ile SG uygulaması kullanma durumları arasında ilişki görülmemiştir.

Araştırmamızda uygulamaya katılan öğrencilerin genel BHÖ ortalaması puanları ile alt boyut puanları literatür ile uyum göstermiştir (Tablo 4.14). Araştırmamızda öğrencilerin yüksek oranda bulunuşluk hissine sahip olduğu görülmüştür. Aynı zamanda öğrencilerin uyum ve çevreleme alt boyut puanları da literatür ile uyumluluk göstermiştir (Tablo 4.14).

Bu sonuç doğrultusunda araştırmanın hipotezleri olan, "Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin görsel, işitsel ve dokunsal olarak algılamasına etkisi vardır." ve "Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin çevrelenmişlik duygusu ile sürekli bir deneyim ve uyaran akışı içerisine dahil edilip bunlarla etkileşim kurmasına etkisi vardır." hipotezleri kabul edilmiştir.

## 5.4. DENEY GRUBUNDAKİ ÖĞRENCİLERİN DENEYİMLEDİKLERİ SANAL GERÇEKLİK UYGULAMASINDAKİ KALİTATİF GERİ BİLDİRİMLERİNE AİT BULGULARIN TARTIŞILMASI

Literatür incelendiğinde SG uygulamalarının kullanıldığı çalışmalarda kalitatif geri bildirim çok az sayıda makale de incelendiği görülmüştür. Kalitatif geri bildirim alınan çalışmalarda uygulanan SG tekniği mevcut eğitime göre anmalı fark oluşturmamış olsa da, öğrencilerden alınan sözel geri bildirimlerin olumlu olduğu ve uygulamayı kullanmaya pozitif baktıkları görülmüştür (162, 200, 201).

Moro ve ark. (162), medikal anatomide SG ve AR gerçeklik modelinin etkinliği inceledikleri çalışmalarında öğrencilerin uygulama ile ilgili sözel bildirimlerinin aşağıdaki şekilde olduğu görülmüştür.

"Oculus (SG gözlüğü), kafatasının tüm kısımlarını istediğiniz açıda görmenizi sağladığı için iyi bir öğrenme aracı olarak kullanılabilir. Öğrendiklerimizi herhangi bir şekilde görselleştirebilmek yardımcı oluyor",

"Gerçekten iyi! Kemikleri görselleştirmek ve hangi kemiklere bakılacağını görebilmek/seçebilmek için son derece yararlıdır. Ses bilgilendiriciydi. Bu aktiviteyi yaparak çok şey öğrendim- kesinlikle bunu yaparken bir derste öğrenmekten çok daha fazlasını öğrendiğimi hissediyorum."

"Ses akışına gerçekten dikkat etmiyordum. Biraz başımı döndürebilse de teknoloji daha çok ilgimi çekti"

"Programın ne kadar havalı olduğu konusunda çok dikkatimin dağıldığını fark ettim ve programın öğrenme yönüne odaklanmadığımı fark ettim! Bunun dışında çok havalı ve bunun anatomi öğrencileri için faydalı bir araç olduğunu görebiliyorum."

Saab ve ark. (200), hemşirelik öğrencilerinde (n=26), SG uygulaması ile ilgili görüşlerini inceledikleri kalitatif çalışmalarında, SG'nin büyüleyici, yenilikçi ve güçlendirici doğası, bağlamsal aktarım ve Gerçekleştirmeye yönelik zorluklar ve tehditler temaları belirlenmiştir. Çalışmada öğrencilerin SG ile ilgili geri bildirimleri aşağıda yer almaktadır.

"...İnternet'te veya TV'de herkes posterler ve videolar görür ve yoluna devam eder. Ama SG'de bir başkasına 'Aa ben bunu yaptım, bunu öğrendim 'diyeceksiniz ve bunu aktaracaksınız."

"Gerçekte, dördüncü derece bir bası yarasını asla görmeyebilirim , fakat o zaman başka biri görebilir. Bu beni dezavantajlı bir duruma sokuyor olabilir, oysa bunu SG'de görebilseydim, herkesi aynı oyun alanına sokardı."

"SG, bu 'Sadece sen ve gözlük var. Kimse seni izlemeyecek. Hata yapmaktan çekinmeden kendinize olan güveninizi artırabilirsiniz. Başarısız olabilirsin, yanlış şeyler yapabilirsin, hatalardan ders alabilirsin."

" Slaytlarda ne olduğunu tam olarak anlamadıysanız, bir derste soru sormak isteyebilirsiniz. Ama bence VR ile soru sorma fırsatınız olmazdı."

Araştırmaya katılan öğrencilerin kalitatif geri bildirim Tablo 4.19'da verilmiştir. Öğrencilerin SG kullanım geri bildirimleri literatürle uyum göstermektedir. Araştırmada öğrencilerin, uygulamayı müthiş, etkileyici ve harika bir deneyim olarak gördüğü ve fetal gelişim için etkili bir uygulama olduğunu bildirmişlerdir. Araştırmada SGT-FEGU ile ilgili negatif bir geri bildirim alınmamıştır. Katımcılardan birkaçının SGT-FEGU geri dönüşleri aşağıdaki ifadeleri içeriyordu:

Öğrenci 1 (K1) "Fetal gelişimi yakından görmek bebeğin hareketlerini gözlemlemek çok çok güzeldi anlatılmaz yaşanır dedikleri bu olsa gerek 🔞"

K3 "Çok güzel bir deneyimdi. Bebeğin hareketleri (tekme, gülümseme vb.) görebildik. Umblikal kordu görebildik."

K12 "Gözlüğü taktığım andan itibaren büyülendim diyebilirim. Fetal gelişimi ilk haftalardan itibaren anne karnında gözlemleyebilmek ve istediğimiz haftaya dönüp tekrar izleyebilmek çok güzeldi ve çok gerçekçiydi. Muhteşem bir çalışma olmuş"

K21" Güzel ve gerçeğe yakın bir deneyimdi Teşekkürler reyhan hocamıza 🕄"

K26 "Uygulama çok gerçekçiydi ve kolay kontrol edilebilirdi. Hafta hafta bilgilerin geçmesi ve duyulan seslerin gerçekliği güzeldi. Sanal ortam kolay uyum sağlanabilirdi ve rahatsız edici bir özellik yoktu. Deneyimlememizi sağladığınız için teşekkürler."

K30 "Tek kelimeyle mükemmeldi. Sanki bebek anne karnında değil de benim hemen yanımda büyüyor gibiydi. Bütün organları hafta ilerledikçe daha da belirginleşiyor ve her şey net oluyordu. Yüzündeki hareketlere kadar her şey çok netti. Gelişimle birlikte kalp seslerini dinlemek de çok güzeldi. Kesinlikle bütün ebelik öğrencilerinin, anne ve babalarında deneyimlemesi gerekiyor. Reyhan hocamızda bize böyle bir fırsat sunduğu için ona da çok teşekkür ederim."

K33 "Anne karnında fetüsün gelişimine canlı şahit olmak mükemmel bir şey"

K41 "Mükemmel bir çalışma olmuş. Gerçekten anne karnında bebeğin gelişimini izliyor gibi hissettim. Haftalar arasında geçiş yaparak izleyebilmekte oldukça iyiydi."

Araştırmada, öğrencilerin kendilerini anne karnında gibi hissetmeleri, bebeğin hareketlerini yakından gözlememeleri ve ortamda hareket ederek bebeğe yaklaşmaları SGT-FEGU ile etkileşim kurmalarını sağlamıştır. Bu eylemlerde öğrencilerden olumlu geri bildirim alınmış ve kalitatif olarak da bu durum doğrulanmıştır. Bu sonuçlar doğrultusunda araştırmanın "Fetal gelişimin öğretiminde SGT-FEGU uygulamasının öğrencilerin çevrelenmişlik duygusu ile sürekli bir deneyim ve uyaran akışı içerisine dahil edilip bunlarla etkileşim kurmasına etkisi vardır." Hipotezi kabul edilmiştir.

## 6. SONUÇLAR VE ÖNERİLER

#### 6.1. SONUÇLAR

Fetal gelişimin öğretiminde SGT-FEGU'nun geliştirilmesi ve kullanılması amacıyla randomize kontrollü deneysel olarak tasarlanan araştırmada H<sub>1</sub> hipotezleri kabul edildi. Kabul edilen hipotezler doğrultusunda;

- Araştırmadaki deney ve kontrol grubundaki öğrencilerin, yaş, AGNO puanları, yaşadıkları yer, bölümü tercih etme sıraları, mezuniyet sonrası planları, bilgisayar kullanım durumları, SG bilgi düzeyleri ile SG uygulamasını deneyimleri durumları arasında homojen dağılım saptandı (Tablo 4.1).
- Deney ve kontrol grubunun FEGBÖ ön test ve son test puanları incelendiğinde; deney grubun kendi içindeki puanları arasında fark saptandı, kontrol grubunun puanları arasında fark görülmedi (Tablo 4.11).
- Deney ve kontrol grubunun ön test puanları arasında fark saptanmadı (Tablo 4.10).
- Grupların son test puanları arasında istatistiksel olarak anlamlı fark görüldü (Tablo 4.11).
- Araştırmada geliştirilen SGT-FEGU'yu kullanan deney grubu öğrencilerin BYÖ puanları düşük bulundu (Tablo 4.13).
- Deney grubundaki öğrencilerin uygulama sonrası BHÖ puan alt boyutları ölçek referans değerlerine yakın, literatüre oranla da olarak saptandı (Tablo 4.14).
- Araştırmada deney grubunda BYÖ ile BHÖ'nün etkileşim alt boyutu arasında düşün düzeyde negatif yönde anlamlı ilişki saptandı (Tablo 5.15).
- Deney grubunda SGT-FEGU'yu deneyimleryen öğrencilerin olumlu kalitatif geri bildirimler alındı. Uygulama öğrenciler tarafından "muhteşem, güzel, gerçekçi ve harika" olarak tanımlandı (Tablo 4.19).

### 6.2. ÖNERİLER

- Fetal gelişim öğretimi için geliştirilen SGT-FEGU'nun alternatif bir öğretim aracı olarak kullanılması,
- Öğrencilerin fetal gelişim gibi gerçek hayatta gözlemlenmesinin zor olacağı uygulamalar için sanal gerçeklik modellemesinin eğitim materyali olarak kullanılması,
- Geliştirilen uygulamanın farklı örneklem gruplarında uygulanıp sonuçlarının değerlendirilmesi ve ebelik eğitiminde kullanılması,
- Ebelik eğitiminde sanal gerçeklik alanının daha farklı ve daha fazla çalışmalarla desteklenmesi önerilebilir.

#### KAYNAKLAR

- 1. Cochard, L. R. (2012) Netter's Atlas of Human Embryology E-Book: Updated Edition (Elsevier Health Sciences)
- 2. Gür, E. Y., Apay, S. E. (2018) *Embriyonel ve Fetal Gelişim ve Fizyolojisi* (İstanbul Tıp Kitapevleri, İstanbul). 1st Ed.
- 3. Smith, R. P. (2017) Netter's Obstetrics and Gynecology E-Book (Elsevier Health Sciences)
- 4. Carlson, B. M. (2018) *Human Embryology and Developmental Biology E-Book: With Student Consult Online Access* (Elsevier Health Sciences)
- 5. Cooper, S., Cant, R., Porter, J., Bogossian, F., McKenna, L., Brady, S., Fox-Young, S. (2012) Simulation based learning in midwifery education: a systematic review. *Women and Birth* 25, 64–78
- 6. Hazar, H. U., Gültekin, S. (2019) Ebelik Eğitiminde Simülasyon Kullanımı. Life Sciences 14, 74–83
- 7. Williams, J., Jones, D., Walker, R. (2018) Consideration of using virtual reality for teaching neonatal resuscitation to midwifery students. *Nurse education in practice* 31, 126–129
- 8. Becker, J., Zankl, M., Fill, U., Hoeschen, C. (2008) Katja—the 24th week of virtual pregnancy for dosimetric calculations. *Polish Journal of Medical Physics and Engineering* 14, 13–20
- 9. Bogossian, F., McKenna, L., Higgins, M., Benefer, C., Brady, S., Fox-Young, S., and Cooper, S. (2012) Simulation based learning in Australian midwifery curricula: Results of a national electronic survey. *Women and Birth* 25, 86–97
- 10. Ohmaru, T., Fujita, Y., Sugitani, M., Shimokawa, M., Fukushima, K., Kato, K. (2015) Placental elasticity evaluation using virtual touch tissue quantification during pregnancy. *Placenta* 36, 915–920
- 11. Verwoerd-Dikkeboom, C. M., Koning, A. H. J., Hop, W. C., Rousian, M., Van Der Spek, P. J., Exalto, N., Steegers, E. A. P. (2008) Reliability of three-dimensional sonographic measurements in early pregnancy using virtual reality. *Ultrasound in Obstetrics and Gynecology: The Official Journal of the International Society of Ultrasound in Obstetrics and Gynecology* 32, 910–916
- 12. Lomanowska, A. M., Guitton, M. J. (2014) My avatar is pregnant! Representation of pregnancy, birth, and maternity in a virtual world. *Computers in Human Behavior* 31, 322–331
- 13. Öztürk, D. M., Sayıner, F. D., and Çelik, N. (2018) Ebelik Öğrencilerinin Bilgisayarlı Simülasyon Uygulaması Sonrası Görüşlerinin Değerlendirilmesi. *Sağlık Hizmetleri ve Eğitimi Dergisi* 2, 66–71
- 14. Coşar Çetin, F. (2018) in *Doğum Öncesi Dönem I* (İstanbul Tıp Kitap Evleri, İstabul). 1st Ed.
- 15. Marshall, J. E., Raynor, M. D. (2014) Myles Textbook for Midwives (Elservier). 16th Ed.
- 16. Yıldırım, M. (2002) Resimli İnsan Anatomisi Sağlık Yüksek Okulları İçin (Nobel Tıp Kitabevleri)
- 17. Taşkın, L. (2019) Doğum ve Kadın Sağlığı Hemşireliği (Akademisyen Kitabevi)16. Baskı.
- 18. Büyükmumcu, M. (2020) Resimli Sistematik Anatomi. 5th Ed.
- 19. Vural, F., Uzel, M. (2012) İnsan anatomisi (Akademi Basın ve Yayıncılık)2. Baskı.
- 20. Öz, G. (2012) Kadın sağlığı hastalıkları ve bakımı (Rulo Ofset Matbaacılık)
- 21. Çiçek, N., Akyürek, C., Çelik, Ç., Haberal, A. (2004) *Kadın Hastalıkları ve Doğum Bilgisi Cilt 1* (Atlas Kitapçılık, Ankara) BRC Basım.
- 22. Kumcağız, H., Kumcağız, H. (2020) in Cinsel Sağlık Eğitimi (Pegem Akademi, Ankara), pp 87–115.
- 23. Yücel, M. K. (2015) Doğum ve Kadın Sağlığı (Palme Yayınları) Ankara.
- 24. Kocatürk, A. (2018) in *Doğum Öncesi Dönem I* (İstanbul Tıp Kitapevleri). 1st Ed.
- 25. Rathfisch, G. (2015) in *Hemşire ve Ebelere Yönelik Kadın Sağlığı ve Hastalıkları* (Nobel Tıp Kitabevleri), pp 197–213. 1st Ed.
- 26. Barry, J. S., Anthony, R. V. (2008) The pregnant sheep as a model for human pregnancy. *Theriogenology* 69, 55–67
- 27. Pardi, G., Cetin, I. (2006) Human fetal growth and organ development: 50 years of discoveries. *American journal of obstetrics and gynecology* 194, 1088–1099
- 28. Wilcox, A. J., Weinberg, C. R., O'Connor, J. F., Baird, D. D., Schlatterer, J. P., Canfield, R. E., Armstrong, E. G., Nisula, B. C. (1988) Incidence of early loss of pregnancy. *New England Journal of Medicine* 319, 189–194
- 29. Bhattacharya, N., Stubblefield, P. G. (2016) *Human Fetal Growth and Development* (Springer International Publishing, Springer International Publishing Switzerland)
- 30. CFH (2019) If You Are Pregnant: Information on fetal development, abortion and alternatives Woman's Right to Know Act. *Minnesota Department of Health Child & Family Health Division*,
- 31. Keith, L., Moore, P., VN, T., Torchia, M. G. (2013) Developing Human: Clinically Oriented Embryology, (Elsevier India)
- 32. Hill, M. A. (2018) Two web resources linking major human embryology collections worldwide. *Cells Tissues Organs* 205, 293–302

- 33. Webster, S., De Wreede, R. (2016) *Embryology at a Glance* (John Wiley & Sons)
- 34. Webster, S., Atherton, S. (2015) An Augmented Reality Embryology Textbook. *The FASEB Journal* 29, 550–6
- 35. NG (2021) The Biology of Prenatal Development. The Endowment for Human Development,
- 36. Coşkun, A. M. (2012) in Kadın Sağlığı ve Hastalıkları Hemşireliği El Kitabı (Koç Üniversitesi Yayınları).
- 37. Karahan, N., ve Serhatlıoğlu, S. (2019) in *Hemşirelik ve Ebelik İçin Kadın Sağlığı ve Hastalıkları* (Akademisyen Kitabevi), pp 134–171.
- 38. Moore, K. L., Persaud, T. V. N., and Torchia, M. G. (2018) *The developing human-e-book: clinically oriented embryology* (Elsevier Health Sciences)
- 39. Dinçer, S., Doğanay, A. (2016) Öğretim Materyali'ne İlişkin Motivasyon Ölçeği (ÖMMÖ) Türkçe Uyarlama Çalışması. *Ilkogretim Online* 15,
- 40. Turan, F. D. (2020) Sanal Gerçeklik Teknolojisi ile Hazırlanmış Epileptik Nöbet Yönetimi Eğitim Programının Ebeveynlerin Nöbet Yönetimine Etkisi.
- 41. Goldthwaite, L. M., Tocce, K. (2017) Simulation training for family planning procedures. *Current Opinion in Obstetrics and Gynecology* 29, 437–442
- 42. Chang, C.-Y., Sung, H.-Y., Guo, J.-L., Chang, B.-Y., Kuo, F.-R. (2019) Effects of spherical video-based virtual reality on nursing students' learning performance in childbirth education training. *Interactive Learning Environments*, 1–17
- 43. Kayabaşı, Y. (2002) Sanal gerçeklik ve eğitim amaçli kullanılmasi. Turkish Online, 151
- 44. Schroeder, R. (1997) Networked worlds: Social aspects of multi-user virtual reality technology. *Sociological Research Online* 2, 89–99
- 45. Çavaş, B., Huyugüzel, P., Can, B. (2004) Eğitim de Sanal Gerçeklik Uygulamaları.
- 46. Bayram, S. (1999) Eğitimde Sanal Gerçeklik Uygulamaları. *Marmara Üniversitesi Atatürk Eğitim Fakültesi Eğitim Bilimleri Dergisi* 11, 49–54
- 47. Warburton, S. (2009) Second Life in higher education: Assessing the potential for and the barriers to deploying virtual worlds in learning and teaching. *British journal of educational technology* 40, 414–426
- 48. Avcı, A. F., Taşdemir, Ş. (2019) Artırılmış ve Sanal Gerçeklik İle Periyodik Cetvel Öğretimi. *Selcuk University Journal of Engineering Sciences* 18, 68–83
- 49. Rosenblum, L., Durbin, J., Doyle, R., Tate, D. (1997) *The virtual reality Responsive Workbench: applications and experiences* (Naval Research Lab Washington Dc)
- 50. Helsel, S. (1992) Virtual reality and education. Educational Technology 32, 38-42
- 51. Burnett, B. (1993) Virtual reality and technology. T. Hayward, Adventures in Virtual Reality. Carmel, IN: Que Corporation, 231
- 52. Jacobson, R. (1994) Applying the virtual worlds paradigm to mapping and surveying data. *Virtual Reality World* 2, 60–62
- 53. Bayraktar, E., Kaleli, F. (2007) Sanal gerceklik ve uygulama alanlari. Akademik Bilişim, 1-6
- 54. Wodaski, R. (1993) Virtual Reality Madness! (SAMS publishing)
- 55. Abbey, C. (1994) VR Means Virtual Reconstruction. Wired,
- 56. Arat, T., Baltacıoğlu, S. (2016) Sanal gerçeklik ve turizm. *Selçuk Üniversitesi Sosyal Bilimler Meslek Yüksek Okulu Dergisi* 19, 103–118
- 57. Özgüneş, R. E., Bozok, D. (2017) Turizm sektörünün sanal rakibi (mi?): Arttırılmış gerçeklik. *Uluslararası Türk Dünyası Turizm Araştırmaları Dergisi* 2, 146–160
- 58. Demirezen, B. (2019) Artırılmış Gerçeklik ve Sanal Gerçeklik Teknolojisinin Turizm Sektöründe Kullanılabilirliği Üzerine Bir Literatür Taraması. *Uluslararası Global Turizm Araştırmaları Dergisi* 3, 1–26
- 59. VRAC (2006) Virtual Reality Applications Center. Virtual Reality Application Center,
- 60. Göktaş, H. H., Çavuşoğlu, A., Sen, B., Görgünoğlu, S. (2006) Simülasyon Sistemleri İçin 3 Boyutlu Sanal Şehirlerin Sayısal Coğrafik Haritalar Üzerinde Oluşturulması. *Teknoloji* 9,
- 61. Zafer, D. Z. (2015) Mimari tasarım sürecine sanal gerçeklik teknolojilerinin etkisi.
- 62. Süygün, M. S., Bozyiğit, S. (2021) Dış Ticaret ve Lojistik Eğitiminde Sanal Gerçeklik Teknolojisinin Kullanımı. *Journal of the Cukurova University Institute of Social Sciences* 30,
- 63. Papadopoulou, P. (2007) Applying virtual reality for trust-building e-commerce environments. *Virtual Reality* 11, 107–127
- 64. Martínez-Navarro, J., Bigné, E., Guixeres, J., Alcañiz, M., and Torrecilla, C. (2019) The influence of virtual reality in e-commerce. *Journal of Business Research* 100, 475–482
- 65. Chittaro, L., Ration, R. (2000) in *International Conference on Adaptive Hypermedia and Adaptive Web-Based Systems* (Springer), pp 86–97.
- 66. Mass, Y., Herzberg, A. (1999) in Proceedings of the 1st ACM Conference on Electronic Commerce, pp

- 103-109.
- 67. Chittaro, L., Ranon, R. (2000) in *Proceedings of the CHI2000 Workshop on Designing Interactive Systems for 1-to-1 E-Commerce* (Citeseer).
- 68. Kilmon, C. A., Brown, L., Ghosh, S., Mikitiuk, A. (2010) Immersive virtual reality simulations in nursing education. *Nursing education perspectives* 31, 314–317
- 69. Shin, Y.-S. (2002) Virtual reality simulations in web-based science education. *Computer Applications in Engineering Education* 10, 18–25
- 70. Coulter, R., Saland, L., Caudell, T., Goldsmith, T. E., Alverson, D. (2007) The effect of degree of immersion upon learning performance in virtual reality simulations for medical education. *InMedicine Meets Virtual Reality* 15, 155
- 71. Lamb, R. L., Etopio, E. (2019) Virtual reality simulations and writing: A neuroimaging study in science education. *Journal of Science Education and Technology* 28, 542–552
- 72. Tepe, T., Kaleci, D., Tüzün, H. (2016) in 10th International Computer and Instructional Technologies Symposium (ICITS), pp 16–18.
- 73. Kalaycı, İ. (2019) Sanal Gerçeklik Teknolojisiyle İşlenen Tarih Metodolojisi Dersinin Öğrenci Algısına Etkileri. *Turkish Studies-Information Technologies and Applied Sciences* 14, 569–585
- 74. Topuz, Y., and Özdener, N. (2018) Tıp Eğitimde Sanal Gerçeklik Teknolojisi. *Değişen Dünyada Eğitim*, 225
- 75. Demir, R. (2020) "Din Kültürü ve Ahlak Bilgisi Öğretimi Dersi" nde Artırılmış Gerçeklik Uygulamalarının Öğrenci Görüşleri Doğrultusunda Değerlendirilmesi. *Çukurova Üniversitesi İlahiyat Fakültesi Dergisi (ÇÜİFD)* 20, 201–219
- 76. Arıcı, V. A. (2013) Fen eğitiminde sanal gerçeklik programları üzerine bir çalışma:" Güneş sistemi ve ötesi: Uzay bilmecesi" ünitesi örneği.
- 77. Larijani, L. C. (1993) The virtual reality primer (McGraw-Hill, Inc.)
- 78. McGonigle, D., Eggers, R. M. (1998) Stages of virtually: Instructor and student. *TechTrends* 43, 23–26 79. Kandemir, C., Demir, B. A. (2020) Eğitimde Sanal Gerçeklik Uygulamaları Üzerine: "Sınıfta Ben De Varım" Projesi. *The Turkish Online Journal of Design Art and Communication* 10, 339–354
- 80. Roussou, M. (2004) Learning by doing and learning through play: an exploration of interactivity in virtual environments for children. *Computers in Entertainment (CIE)* 2, 10–10
- 81. Başaran, F. (2010) Öğretmen adaylarının eğitiminde sanal gerçeklilk kullanımına ilişkin görüşleri (Sakarya Üniversitesi BÖTE örneği).
- 82. Nooriafshar, M., Williams, R., Maraseni, T. N. (2004) in *Proceedings of the 7th American Society of Business and Behavioral Sciences International Conference (ASBBS 2004)* (American Society of Business and Behavioral Sciences (ASBBS)).
- 83. Tuncer, M., Taşpınar, M. (2008) Sanal Ortamda Eğitim Ve Öğretimin Geleceği Ve Olasi Sorunlar. *Sosyal Bilimler Dergisi* 10, 124
- 84. Tepe, T. (2019) Başa Takılan Görüntüleyiciler İçin Geliştirilmiş Sanal Gerçeklik Ortamlarının Öğrenme ve Buradalık Algısı Üzerine Etkilerinin İncelenmesi.
- 85. Akgün, İ. (2019) Robotik Rehabilitasyonun Inmeli Hastalarda üst Ekstremite fonksiyonları Ve yaşam Kalitesi üzerine Etkisi.
- 86. Kayabınar, B. (2019) Kronik İnmeli Hastalarda Sanal Gerçeklik Eğitiminin İkili Görev Performansı, Denge ve Yürüme Üzerine Etkilerinin İncelenmesi.
- 87. Özkan, F., Zincir, H. (2017) Serebral Palsili Çocukların Rehabilitasyonunda Sanal Gerçeklik Tedavisi: Sistematik Derleme. *Sağlık Bilimleri Dergisi* 26, 181–188
- 88. Yavuzarslan, M., Demirkol, D., Gülseçen, S. (2020) Sanal Gerçeklik Teknolojilerinin İnme Geçiren Hastaların Rehabilitasyonundaki Rolüne İlişkin Bir Literatür Taraması. *Journal of Information Systems and Management Research* 2, 42–49
- 89. Dereli, E. (2010) İnme Geçiren Hastaların Üst Ekstremite Rehabilitasyonunda Sanal Gerçeklik Temelli ve Göreve Yönlendirilmiş Egzersizlerin El Fonksiyonlarına Etkisinin Karşılaştırılması.
- 90. Louvre Müzer turu (2021) Louvre Museum Official Website. Le Louvre,
- 91. KTB (2021) Virtual Tour. Kültür ve Turizm Bakanlığı,
- 92. Dunn, A., Patterson, J., Biega, C. F., Grishchenko, A., Luna, J., Stanek, J. R., Strouse, R. (2019) A novel clinician-orchestrated virtual reality platform for distraction during pediatric intravenous procedures in children with hemophilia: randomized controlled trial. *JMIR serious games* 7, e10902
- 93. Atzori, B., Lauro Grotto, R., Giugni, A., Calabrò, M., Alhalabi, W., Hoffman, H. G. (2018) Virtual reality analgesia for pediatric dental patients. *Frontiers in psychology* 9, 2265
- 94. Binay Yaz, Ş., Bal Yılmaz, H. (2021) Pediatrik Hastalara Yönelik Tıbbi İşlemlerde Sanal Gerçeklik Kullanımının Etkileri: Literatür İncelemesi. *Gümüşhane Üniversitesi Sağlık Bilimleri Dergisi* 10, 138–143
- 95. Javaid, M., Haleem, A. (2020) Virtual reality applications toward medical field. Clinical Epidemiology

- and Global Health 8, 600–605
- 96. Hoffman, H. G., Chambers, G. T., Meyer III, W. J., Arceneaux, L. L., Russell, W. J., Seibel, E. J., Richards, T. L., Sharar, S. R., Patterson, D. R. (2011) Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. *Annals of behavioral medicine* 41, 183–191
- 97. Noben, L., Goossens, S. M. T. A., Truijens, S. E. M., Van Berckel, M. M. G., Perquin, C. W., Slooter, G. D., Van Rooijen, S. J. (2019) A virtual reality video to improve information provision and reduce anxiety before cesarean delivery: randomized controlled trial. *JMIR mental health* 6, e15872
- 98. Mantovani, F., Castelnuovo, G., Gaggioli, A., Riva, G. (2003) Virtual reality training for health-care professionals. *CyberPsychology & Behavior* 6, 389–395
- 99. Gaba, D. M. (2004) The future vision of simulation in health care. BMJ Quality & Safety 13, i2-i10
- 100. Bracq, M.-S., Michinov, E., Jannin, P. (2019) Virtual reality simulation in nontechnical skills training for healthcare professionals: a systematic review. *Simulation in Healthcare* 14, 188–194
- 101. Demirci, Ş. (2018) Sağlık Hizmetlerinde Sanal Gerçeklik Teknolojileri. İnönü Üniversitesi Sağlık Hizmetleri Meslek Yüksek Okulu Dergisi 6, 35–46
- 102. Williams, J., Jones, D., Ebert, L., Williams, C. (2017) Exploring the use of virtual reality technology in neonatal resuscitation simulation for midwifery students. *Women and Birth* 30, 13–14
- 103. Weller, J. M., Nestel, D., Marshall, S. D., Brooks, P. M., Conn, J. J. (2012) Simulation in clinical teaching and learning. *Medical Journal of Australia* 196, 594–594
- 104. Çalım, S. İ., Öztürk, E. (2018) Ebelik Beceri Eğitiminde Simülasyon Kullanımı: Sistematik Derleme. 105. Nehring, W. M., Lashley, F. R. (2009) Nursing simulation: A review of the past 40 years. *Simulation & Gaming* 40, 528–552
- 106. Williams, J., Jones, D., Walker, R. (2018) Consideration of using virtual reality for teaching neonatal resuscitation to midwifery students. *Nurse Education in Practice* 31, 126–129
- 107. Cooper, S., Cant, R., Porter, J., Bogossian, F., McKenna, L., Brady, S., Fox-Young, S. (2012) Simulation based learning in midwifery education: a systematic review. *Women and Birth* 25, 64–78
- 108. Ferguson, C., Davidson, P. M., Scott, P. J., Jackson, D., and Hickman, L. D. (2015) Augmented reality, virtual reality and gaming: an integral part of nursing.
- 109. Mao, J., Horan, B., Forbes, H., Smilevski, S., Bucknall, T., Nagle, C., Phillips, D., and Gibson, I. (2017) in *The International Conference on Design and Technology* (KnowledgeE), pp 44–50.
- 110. McGhee, S. J. A., Bradley, P. J., and McComish, A. G. (2011) Immersive virtual reality: Potential use in an undergraduate nursing & midwifery program in Scotland. *Studies in Learning, Evaluation, Innovation & Development* 8,
- 111. Kyaw, B. M., Saxena, N., Posadzki, P., Vseteckova, J., Nikolaou, C. K., George, P. P., Divakar, U., Masiello, I., Kononowicz, A. A., Zary, N. (2019) Virtual reality for health professions education: systematic review and meta-analysis by the digital health education collaboration. *Journal of medical Internet research* 21, e12959
- 112. Fealy, S., Jones, D., Hutton, A., Graham, K., McNeill, L., Sweet, L., and Hazelton, M. (2019) The integration of immersive virtual reality in tertiary nursing and midwifery education: A scoping review. *Nurse education today* 79, 14–19
- 113. Downer, T., Gray, M., Andersen, P. (2020) Three-dimensional technology: evaluating the use of visualisation in midwifery education. *Clinical Simulation in Nursing* 39, 27–32
- 114. Jones, D., Hazelton, M., Evans, D. J., Pento, V., See, Z. S., Van Leugenhaege, L., and Fealy, S. (2021) in *Digital Anatomy* (Springer), pp 325–342.
- 115. Phillips, D., Duke, M., Nagle, C., Macfarlane, S., Karantzas, G., Patterson, D. (2013) The Virtual Maternity Clinic: A teaching and learning innovation for midwifery education. *Nurse education today* 33, 1224–1229
- 116. Downer, T., Gray, M., and Capper, T. (2021) Online learning and teaching approaches used in midwifery programs: A scoping review. *Nurse Education Today*, 104980
- 117. Öner, S. (2020) Yenidoğanın ilk bakımına yönelik bir sanal gerçeklik simülasyonunun geliştirilmesi ve değerlendirilmesi.
- 118. İsmail, N. H. B. (2019) Fetal Growth Based on al Quran Using Augmented Reality.
- 119. Sielhorst, T., Obst, T., Burgkart, R., Riener, R., and Navab, N. (2004) in *International workshop on augmented environments for medical imaging-MICCAI Satellite Workshop*, pp 11–20.
- 120. Atlantis VR (2010) Development of Pregnancy Simulator Provided With A.I. and Augmented Reality. 121. Random.org (1998) Random.org True Random Number Service.
- 122. Paas, F. G., Van Merriënboer, J. J. (1993) The efficiency of instructional conditions: An approach to combine mental effort and performance measures. *Human factors* 35, 737–743
- 123. Kılıç, A. G. E., Karadeniz, Ö. G. Ş. (2004) Hiper ortamlarda öğrencilerin bilişsel yüklenme ve kaybolma düzeylerinin belirlenmesi. *Kuram ve Uygulamada Eğitim Yönetimi* 40, 562–579

- 124. Witmer, B. G., Jerome, C. J., Singer, M. J. (2005) The factor structure of the presence questionnaire. *Presence: Teleoperators & Virtual Environments* 14, 298–312
- 125. Gökoğlu, S., Çakıroğlu, Ü. (2019) Sanal Gerçeklik Temelli Öğrenme Ortamlarında Bulunuşluk Hissinin Ölçülmesi: Bulunuşluk Ölçeğinin Türkçe'ye Uyarlanması. *Eğitim Teknolojisi Kuram ve Uygulama* 9, 169–188
- 126. Lumen Learning (2021) Stages of Development | Introductory Psychology.
- 127. Musumeci, G., Castrogiovanni, P., Trovato, F. M., Parenti, R., Szychlinska, M. A., and Imbesi, R. (2015) Pregnancy, embryo-fetal development and nutrition: physiology around fetal programming. *J Histol Histopathol* 2, 1
- 128. İÜ (2021) İstanbul Üniversitesi-Cerrahpa Üniversitesi, Sağlık Bilimleri Fakültesi, Ebelik Bölümü, AKTS Bilgi Paketi. İstanbul Üniversitesi-Cerrahpaşa AKTS Bilgi Paketi,
- 129. KBU (2021) Karabük Üniversitesi, Sağlık Bilimleri Fakültesi, Ebelik Bölümü, AKTS Bilgi Paketi.
- 130. MÜ (2021) Medipol Üniversitesi, Sağlık Bilimleri Fakültesi, Ebelik Bölümü, AKTS Bilgi Paketi.
- 131. YÖK (2016) EUÇEP.
- 132. Aquaportail (2021) Couche germinale: définition et explications. AquaPortail,
- 133. Turbosquid (2021) Free 3D fetus 37 development TurboSquid 1329462.
- 134. George, D. (2011) SPSS for windows step by step: A simple study guide and reference, 17.0 update, 10/e (Pearson Education India)
- 135 Dikmen, M., Şimşek, M., Tuncer, M. (2018) Öğrenme stilleri ile öğrenmeye yönelik tutum arasındaki ilişki.
- 136. Demir, M. K. (2006) Sınıf Öğretmeni Adaylarının Öğrenme Stilleri ve Sosyal Bilgiler Öğretimi. Eurasian Journal of Educational Research (EJER),
- 137. Cavas, B. (2010) A Study on Pre-service Science, Class and Mathematics Teachers' Learning Styles in Turkey. *Science Education International* 21, 47–61
- 138. Can, Ş. (2010) Determination of the learning styles of the pre-school teacher candidates (The case of Muğla University, Turkey). *Procedia-Social and Behavioral Sciences* 2, 4137–4141
- 139. Çubukçu, Z. (2004) Öğretmen Adaylarinin Düşünme Stillerinin Öğrenme Biçimlerini Tercih Etmelerindeki Etkisi.
- 140. Özgür, H. (2013) Uzaktan eğitim öğrencilerinin öğrenme stilleri: Trakya Üniversitesi örneği. *Trakya Üniversitesi Eğitim Fakültesi Dergisi* 3,
- 141. Bingöl, F. B., Bal, M. D., Karakoç, A., and Aslan, B. (2020) Ebelik Öğrencilerinin Doğum Simülasyon Eğitimi Deneyimleri. *Acıbadem Üniversitesi Sağlık Bilimleri Dergisi*, 711–718
- 142. Karakoc, A., Bal, M. D., Bingol, F. B., and Aslan, B. (2019) The effects of simulation-based education on initial neonatal evaluation and care skills. *Pakistan journal of medical sciences* 35, 911
- 143. Durmaz, A., Elem, E., Unutkan, A., Keskin, N. (2017) The effect of simulation on vaginal delivery skills and self-sufficiency levels. *J Curr Res Health Secto* 7, 41–52
- 144. Tsai, S.-L., Chai, S.-K., Hsieh, L.-F., Lin, S., Taur, F.-M., Sung, W.-H., and Doong, J.-L. (2008) The use of virtual reality computer simulation in learning Port-A cath injection. *Advances in Health Sciences Education* 13, 71–87
- 145. Gu, Y., Zou, Z., Chen, X. (2017) The Effects of vSIM for Nursing<sup>TM</sup> as a teaching strategy on fundamentals of nursing education in undergraduates. *Clinical Simulation in Nursing* 13, 194–197
- 146. Liaw, S. Y., Chan, S. W.-C., Chen, F.-G., Hooi, S. C., and Siau, C. (2014) Comparison of virtual patient simulation with mannequin-based simulation for improving clinical performances in assessing and managing clinical deterioration: randomized controlled trial. *Journal of medical Internet research* 16, e3322
- 147. Jung, E.-Y., Park, D. K., Lee, Y. H., Jo, H. S., Lim, Y. S., Park, R. W. (2012) Evaluation of practical exercises using an intravenous simulator incorporating virtual reality and haptics device technologies. *Nurse Education Today* 32, 458–463
- 148. Cobbett, S., and Snelgrove-Clarke, E. (2016) Virtual versus face-to-face clinical simulation in relation to student knowledge, anxiety, and self-confidence in maternal-newborn nursing: A randomized controlled trial. *Nurse Education Today* 45, 179–184
- 149. Ismailoglu, E. G., Zaybak, A. (2018) Comparison of the effectiveness of a virtual simulator with a plastic arm model in teaching intravenous catheter insertion skills. *CIN: Computers, Informatics, Nursing* 36, 98–105
- 150. Smith, S. J., Farra, S. L., Ulrich, D. L., Hodgson, E., Nicely, S., Mickle, A. (2018) Effectiveness of two varying levels of virtual reality simulation. *Nursing education perspectives* 39, E10–E15
- 151. LeFlore, J. L., Anderson, M., Zielke, M. A., Nelson, K. A., Thomas, P. E., Hardee, G., and John, L. D. (2012) Can a virtual patient trainer teach student nurses how to save lives—teaching nursing students about pediatric respiratory diseases. *Simulation in Healthcare* 7, 10–17

- 152. Tavşanlı, N. G., Kosova, F., Bolsoy, N., Altıparmak, S., Demirci, H., Selma, Ş., Ulaş, S. C., Çalım, S. İ., Okuyan, Y. Ç., Şimşek, H. N. (2018) Tam Donanımlı Doğum Simulasyon Sisteminin Öğrencilerin Ders Başarısına ve Problem Çözme Yeteneklerine Etkisinin Değerlendirilmesi. *Celal Bayar Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi* 5, 22–27
- 153. Nugraha, A. S., Faza, A. N., Indayani, W., Haryanto, H., Setiawan, A. (2018) in 2018 5th International Conference on Information Technology, Computer, and Electrical Engineering (ICITACEE) (IEEE), pp 142–146.
- 154. Butt, A. L., Kardong-Edgren, S., Ellertson, A. (2018) Using game-based virtual reality with haptics for skill acquisition. *Clinical Simulation in Nursing* 16, 25–32
- 155. Haerling, K. A. (2018) Cost-utility analysis of virtual and mannequin-based simulation. *Simulation in Healthcare* 13, 33–40
- 156. Stepan, K., Zeiger, J., Hanchuk, S., Del Signore, A., Shrivastava, R., Govindaraj, S., Iloreta, A. (2017) in *International forum of allergy & rhinology* (Wiley Online Library), pp 1006–1013.
- 157. Chen, F.-Q., Leng, Y.-F., Ge, J.-F., Wang, D.-W., Li, C., Chen, B., Sun, Z.-L. (2020) Effectiveness of virtual reality in nursing education: meta-analysis. *Journal of medical Internet research* 22, e18290
- 158. Jones, D., Siang See, Z., Billinghurst, M., Goodman, L., and Fealy, S. (2019) in *The 17th International Conference on Virtual-Reality Continuum and its Applications in Industry*, pp 1–2.
- 159. Bryant, R., Miller, C. L., Henderson, D. (2015) Virtual clinical simulations in an online advanced health appraisal course. *Clinical Simulation in Nursing* 11, 437–444
- 160. Solyar, A., Cuellar, H., Sadoughi, B., Olson, T. R., Fried, M. P. (2008) Endoscopic Sinus Surgery Simulator as a teaching tool for anatomy education. *The American journal of surgery* 196, 120–124
- 161. Seixas-Mikelus, S. A., Adal, A., Kesavadas, T., Baheti, A., Srimathveeravalli, G., Hussain, A., Chandrasekhar, R., Wilding, G. E., and Guru, K. A. (2010) Can image-based virtual reality help teach anatomy? *Journal of endourology* 24, 629–634
- 162. Moro, C., Štromberga, Z., Raikos, A., Stirling, A. (2017) The effectiveness of virtual and augmented reality in health sciences and medical anatomy. *Anatomical sciences education* 10, 549–559
- 163. Khot, Z., Quinlan, K., Norman, G. R., Wainman, B. (2013) The relative effectiveness of computer-based and traditional resources for education in anatomy. *Anatomical sciences education* 6, 211–215
- 164.Codd, A. M., Choudhury, B. (2011) Virtual reality anatomy: Is it comparable with traditional methods in the teaching of human forearm musculoskeletal anatomy? *Anatomical sciences education* 4, 119–125
- 165. Ellington, D. R., Shum, P. C., Dennis, E. A., Willis, H. L., Szychowski, J. M., Richter, H. E. (2019) Female pelvic floor immersive simulation: a randomized trial to test the effectiveness of a virtual reality anatomic model on resident knowledge of female pelvic anatomy. *Journal of minimally invasive gynecology* 26, 897–901
- 166. Qian, K., Bai, J., Yang, X., Pan, J., Zhang, J. (2015) in *Proceedings of the 21st ACM Symposium on Virtual Reality Software and Technology*, pp 69–78.
- 167. Zhao, J., Xu, X., Jiang, H.,Ding, Y. (2020) The effectiveness of virtual reality-based technology on anatomy teaching: a meta-analysis of randomized controlled studies. *BMC medical education* 20, 1–10
- 168. De Nicola, M., Salvolini, L., Salvolini, U. (1997) Virtual endoscopy of nasal cavity and paranasal sinuses. *European journal of radiology* 24, 175–180
- 169. Pratiwi, I. G., Hamidiyanti, B. Y. F., Arifin, A., Husin, F., Pandudita, R., Ristrini, R., Bachtiar, A., Putro, G., Dramawan, A., Diarti, M. W. (2021) Virtual Reality Improves The Knowledge of Midwives in IUD (Intra Uterine Device) Training. *Jurnal Kesehatan Prima* 15, 74–82
- 170. Sweller, J., Van Merrienboer, J. J., and Paas, F. G. (1998) Cognitive architecture and instructional design. *Educational psychology review* 10, 251–296
- 171. Van Merrienboer, J. J., Ayres, P. (2005) Research on cognitive load theory and its design implications for e-learning. *Educational Technology Research and Development* 53, 5–13
- 172. Sharma, P., Hannafin, M. J. (2007) Scaffolding in technology-enhanced learning environments. *Interactive learning environments* 15, 27–46
- 173. Paas, F., Renkl, A., Sweller, J. (2003) Cognitive load theory and instructional design: Recent developments. *Educational psychologist* 38, 1–4
- 174. Guttormsen Schär, S., and Zimmermann, P. G. (2007) Investigating means to reduce cognitive load from animations: Applying differentiated measures of knowledge representation. *Journal of Research on Technology in Education* 40, 64–78
- 175. Andersen, S. A. W., Mikkelsen, P. T., Konge, L., Cayé-Thomasen, P., Sørensen, M. S. (2016) Cognitive load in mastoidectomy skills training: virtual reality simulation and traditional dissection compared. *Journal of surgical education* 73, 45–50
- 176. Küçük, S. (2015) Mobil Artırılmış Gerçeklikle Anatomi Öğreniminin Tıp Öğrencilerinin Akademik Başarıları ile Bilişsel Yüklerine Etkisi Ve Öğrencilerin Uygulamaya Yönelik Görüşleri. Yayımlanmamış

- Doktora Tezi.
- 177. Küçük, S., Yỳlmaz, R. M., Gökalp, Y. (2014) Augmented reality for learning English: Achievement, attitude and cognitive load levels of students. *Education & Science/Egitim ve Bilim* 39,
- 178. Lee, E. A.-L., Wong, K. W., Fung, C. C. (2010) How does desktop virtual reality enhance learning outcomes? A structural equation modeling approach. *Computers & Education* 55, 1424–1442
- 179. Weng, C., Otanga, S., Weng, A., Cox, J. (2018) Effects of interactivity in E-textbooks on 7th graders science learning and cognitive load. *Computers & Education* 120, 172–184
- 180. Makransky, G., Terkildsen, T. S., and Mayer, R. E. (2019) Adding immersive virtual reality to a science lab simulation causes more presence but less learning. *Learning and Instruction* 60, 225–236
- 181. Du, X., and Arya, A. (2015) in *International Conference on Learning and Collaboration Technologies* (Springer), pp 75–86.
- 182. Şahin Timar, Z. (2020) Çoklu Ortamla Değerlendirme Materyalinde Duygusal Tasarımın İşe Koşulmasının Bilişsel Yüke ve Motivasyona Etkileri.
- 183. Park, B., Flowerday, T., and Brünken, R. (2015) Cognitive and affective effects of seductive details in multimedia learning. *Computers in Human Behavior* 44, 267–278
- 184. Plass, J. L., Heidig, S., Hayward, E. O., Homer, B. D., and Um, E. (2014) Emotional design in multimedia learning: Effects of shape and color on affect and learning. *Learning and Instruction* 29, 128–140
- 185. Um, E., Plass, J. L., Hayward, E. O., Homer, B. D. (2012) Emotional design in multimedia learning. *Journal of educational psychology* 104, 485
- 186. Bailenson, J. N., Yee, N., Blascovich, J., Beall, A. C., Lundblad, N., Jin, M. (2008) The use of immersive virtual reality in the learning sciences: Digital transformations of teachers, students, and social context. *The Journal of the Learning Sciences* 17, 102–141
- 187. Kılıç, T. (2020) Sanal Gerçeklik Teknolojisinin İç Mimarlık Eğitiminde Kullanılmasına Yönelik Bir Öğretim Modeli Önerisi.
- 188. Gökoğlu, S. (2019) Sanal gerçeklik temelli öğrenme ortamının yangın güvenliğine yönelik davranışsal becerilerin gelişimine etkisi.
- 189. Adams, E. (2004) Postmodernism and the Three Types of Immersion, Gamasutra.
- 190. Blascovich, J., Bailenson, J. (2006) in Virtual Decisions (Routledge), pp 239–263.
- 191. Passig, D., Tzuriel, D., Eshel-Kedmi, G. (2016) Improving children's cognitive modifiability by dynamic assessment in 3D Immersive Virtual Reality environments. *Computers & Education* 95, 296–308 192. Freina, L.,Ott, M. (2015) in *The international scientific conference elearning and software for education*, pp 10–1007.
- 193. Johnson, L. F., Levine, A. H. (2008) Virtual worlds: Inherently immersive, highly social learning spaces. *Theory Into Practice* 47, 161–170
- 194. Stoerger, S. (2008) Virtualworlds, Virtualliteracy. Knowledge Quest 36, 50
- 195. Baños, R. M., Botella, C., Alcañiz, M., Liaño, V., Guerrero, B., and Rey, B. (2004) Immersion and emotion: their impact on the sense of presence. *Cyberpsychology & behavior* 7, 734–741
- 196. Monahan, T., McArdle, G., Bertolotto, M. (2008) Virtual reality for collaborative e-learning. *Computers & Education* 50, 1339–1353
- 197. De Leo, G., Diggs, L. A., Radici, E., Mastaglio, T. W. (2014) Measuring sense of presence and user characteristics to predict effective training in an online simulated virtual environment. *Simulation in Healthcare* 9, 1–6
- 198. Peinl, R., Wirth, T. (2020) Presence in VR experiences—an empirical cost-benefit-analysis. *arXiv* preprint arXiv:2002.07576,
- 199. Servotte, J.-C., Goosse, M., Campbell, S. H., Dardenne, N., Pilote, B., Simoneau, I. L., Guillaume, M., Bragard, I., Ghuysen, A. (2020) Virtual reality experience: immersion, sense of presence, and cybersickness. *Clinical Simulation in Nursing* 38, 35–43
- 200. Saab, M. M., Hegarty, J., Murphy, D., Landers, M. (2021) Incorporating Virtual Reality in Nurse Education: A Qualitative Study of Nursing Students' perspectives. *Nurse Education Today*, 105045
- 201. Hardie, P., Darley, A., Carroll, L., Redmond, C., Campbell, A., Jarvis, S. (2020) Nursing & Midwifery students' experience of immersive virtual reality storytelling: an evaluative study. *BMC nursing* 19, 1–12

### **EKLER**

### EK-1. Kişisel Bilgi Formu

düşünüyorsunuz?

**Sayın Katılımcı,** bu çalışma fetal gelişimin öğretiminde "Sanal Gerçeklik Teknolojisi ile Oluşturulan Fetal Gelişim Uygulaması'nın etkinliğini saptamak amacıyla planlanmıştır. Çalışmaya başlamadan önce sizi tanımayı amaçlayan birkaç soruyu cevaplamanız gerekmektedir. Vereceğiniz cevaplar araştırma dışında kullanılmayacağını temin ederim. Katıldığınız için teşekkür ederim.

Prof. Dr. Saadet YAZICI Öğr. Gör. Reyhan AYDIN DOĞAN

| I. Yaşınız |
|---|
| 2. Cinsiyetiniz a. Erkek b. Kadın |
| 3. Medeni durumunuz a. Bekar b. Evli c. Birlikte yaşıyor d. Diğer |
| 4. En uzun süre yaşadığınız yer a. Şehir merkezi b. İlçe c. Kasaba d. Köy |
| 5. Şu anda kaldığınız yer |
| a. Yurtta b. Aile ile c. Evde, yalnız d. Evde, arkadaşlarla e. Diğer |
| 6. Bölümünüz kaçıncı tercihiniz? |
| 7. Bölümünüzü isteyerek mi seçtiniz? a. Evet b. Hayır |
| 8. Ebelik mesleğini tercih etmenize neden olan faktörler nelerdir? a. Ekonomik nedenler b. İş bulma |
| kolaylığı c. Ailenin isteği d. Diğer |
| 9. Şimdiye kadar aldığınız bütün derslere yönelik genel akademik ortalamanız nedir? |
| 10. Normal Doğum ders devamsızlığınızı saat olarak belirtiniz. a. Teorik ders |
| 11. Okuldan mezun olduktan sonra ne yapmayı planlıyorsunuz? |
| a. Ebe olarak çalışmayı planlıyorum b. Akademisyen olarak çalışmayı planlıyorum c. Herhangi bir planım |
| yok |
| d. Diğer |
| 12. Sanal Gerçeklik (VR) ilgili bir bilginiz var mı? a. Evet b. Hayır |
| 13. Sanal Gerçeklik (VR) yönteminin kullanıldığı herhangi bir uygulamaya katıldınız mı? a. Evet b. Hayır |
| 14. Sanal Gerçeklik (VR) yönteminin kullanıldığı bir uygulamaya katıldıysanız bu uygulama hakkında ne |

# EK-2.Fetal Gelişim Değerlendirme bilgi Ölçeği (FEGBÖ)

| ucundan spinal kord şekillenir 9 | Sıra | Fetal Gelişim Değerlendirme bilgi Ölçeği (FEGBÖ) | Doğru | Yanlış | Bilmiyorum |
|---|---|---|---|---|---|
| kromozomlu yeni bir hücre olan "zigotu" meydana getirir lik mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir Trofoblastların dış tabakası sinsityotrofoblastlardır. Embriyonel evreye organogenezis evresi de denir. Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 5 . haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. R. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. Umblikal kord 12. haftanın sonunda gelişir. Umblikal kord 12. haftanın sonunda gelişir. Umblikal kord 12. haftanın sonunda gelişir. Umblikal kord 13. ve 4. haftalarda oluşmaya başlar. Umblikal kord 15. haftanın sonunda gelişir. Umblikal kord 16. haftadının sonunda gelişir. Laftadanın sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Fetüsün in 4. haftada uyaranlara bilinçli cevap vermeye başlar. Fetüsün in 4. haftada uyaranlara bilinçli cevap vermeye başlar. Fetüsün sekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Fetüsün fetisi gerisinde fetüs sert yakalama refleksi yapar. Fetüs 36-40. haftalarda dış ortama artık uyum | 1 | 1 1 | | | |
| getirir Ilk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir Trofoblastların dış tabakası sinsityotrofoblastlardır. Embriyonel evreye organogenezis evresi de denir. Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13. Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. Umblikal kord 12. haftanın sonunda gelişir. Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. Pağırsakların gelişimi 13. haftada gelişmeye başlar. Pağırsakların gelişimi 13. haftada gelişmeye başlar. Petüsün 14. haftada yutkumma, esneme ve yüz buruşturma hareketleri başlar. Petüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Petüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. Petüsün terkek fetüsün testisleri scrotuma inmeye başlar. Petüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. Petüs 26. haftada erkek fetüsün testisleri scrotuma inmeye başlar. Petüs 36. 40. haftalarda dış ortama artık uyum | | | | | |
| Ilk mitoz bölünme sonucu oluşan iki yavru hücreye Blastomer denir. | | · | | | |
| Blastomer denir. Döllemme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir Trofoblastların dış tabakası sinsityotrofoblastlardır. Embriyonel evreye organogenezis evresi de denir. Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10. Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12. 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13. Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14. Umblikal kord içerisindeki arterler ve ven wharton ielly ile çevrilidir. 15. Umblikal kord içerisindeki arterler ve ven wharton ielly ile çevrilidir. 16. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22. 18. hafta içerisinde fetüs sert yakalama refleksi yapar. 23. Fetüs 36-40. haftalarda dış ortama artık uyum | | <u>.</u> | | | |
| Döllenme sonrası 1-2 haftalık olan oluşuma Blastokist adı verilir Trofoblastların dış tabakası sinsityotrofoblastlardır. Embriyonel evreye organogenezis evresi de denir. Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. Fetüs 36-40. haftalarda dış ortama artık uyum | 2 | , | | | |
| Blastokist adı verilir Trofoblastların dış tabakası sinsityotrofoblastlardır. Embriyonel evreye organogenezis evresi de denir. Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10. Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12. 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13. Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14. Umblikal kord 12. haftanın sonunda gelişir. 15. Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22. Jaftadi çerisinde fetüs sert yakalama refleksi yapar. 23. Fetüs 36-40. haftalarda dış ortama artık uyum | 3 | | | | |
| 4 Trofoblastların dış tabakası sinsityotrofoblastlardır. 5 Embriyonel evreye organogenezis evresi de denir. 6 Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 7 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. 8 Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 1 Fetüs 36-40. haftalarda dış ortama artık uyum | 3 | , | | | |
| 5 Embriyonel evreye organogenezis evresi de denir. 6 Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 7 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. 8 Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 4 | | | | |
| 6 Üçüncü germ yaprağı gebeliğin üçüncü haftasında oluşur. 7 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. 8 Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | • | | | |
| oluşur. 7 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. 8 Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | <b>—</b> | | | | |
| 7 24. günde koryonik villiler ve embriyo arasında kan dolaşımı başlar. 8 Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| 8 Embriyonun anterior ucundan beyin, posterior ucundan spinal kord şekillenir 9 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton ielly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 7 | 24. günde koryonik villiler ve embriyo arasında kan | | | |
| ucundan spinal kord şekillenir 9 | | dolaşımı başlar. | | | |
| 5. haftanın sonunda dış genitaller, ilkel biçimde kol ve bacaklar, göz, burun ve kulaklar belirmeye başlar. Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. Umblikal kord 12. haftanın sonunda gelişir. Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22. 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23. Fetüs 36-40. haftalarda dış ortama artık uyum | 8 | | | | |
| ve bacaklar, göz, burun ve kulaklar belirmeye başlar. 10 Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| başlar. Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. Umblikal kord 12. haftanın sonunda gelişir. Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. Bağırsakların gelişimi 13. haftada gelişmeye başlar. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22. 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | 9 | | | | |
| Nöral tüp, beyin ve omurilik dokusu 6. haftada gelişir. Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 13. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 14. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 15. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22. 38. hafta içerisinde fetüs sert yakalama refleksi yapar. | | | | | |
| gelişir. 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | , | | | |
| 11 Embriyoda dil ve dudak oluşumu 8.haftada tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 10 | | | | |
| tamamlanmış olur. 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 1.1 | | | | |
| 12 8. haftada embriyoda el ve ayak parmakları oluşmuş olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 11 | · | | | |
| olmasına rağmen perdeler ile birbirine bağlıdır. 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 1.2 | | | | |
| 13 Umblikal kord 3. ve 4. haftalarda oluşmaya başlar. 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 12 | | | | |
| 14 Umblikal kord 12. haftanın sonunda gelişir. 15 Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 16 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 12 | | | | |
| Umblikal kord içerisindeki arterler ve ven wharton jelly ile çevrilidir. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 13. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 14. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 15. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 26. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 27. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 28. hafta içerisinde fetüs sert yakalama refleksi yapar. 29. Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| jelly ile çevrilidir. 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 13. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 14. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 15. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 26. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 27. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 28. hafta içerisinde fetüs sert yakalama refleksi yapar. 29. Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| 12. haftadan sonra fetüs amnios sıvısı içerisine idrarını yapmaya başlar. 13. Bağırsakların gelişimi 13. haftada gelişmeye başlar. 14. Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 15. Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 26. 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 27. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 28. hafta içerisinde fetüs sert yakalama refleksi yapar. 29. Fetüs 36-40. haftalarda dış ortama artık uyum | 13 | | | | |
| idrarını yapmaya başlar. 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 16 | | | | |
| 17 Bağırsakların gelişimi 13. haftada gelişmeye başlar. 18 Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| Fetüsün 14. haftada yutkunma, esneme ve yüz buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 17 | | | | |
| buruşturma hareketleri başlar. 19 Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| Fetüsün mekonyum denilen ilk dışkısı 18. haftada oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| oluşmaya başlar. 20 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 10 | | | | |
| 22. haftada erkek fetüsün testisleri scrotuma inmeye başlar. 21. Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22. 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23. Fetüs 36-40. haftalarda dış ortama artık uyum | 17 | | | | |
| başlar. 21 Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 20 | | | | |
| Fetüs 24. haftada uyaranlara bilinçli cevap vermeye başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 20 | · | | | |
| başlar. 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 21 | , | | | |
| 22 38. hafta içerisinde fetüs sert yakalama refleksi yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | | , 1 | | | |
| yapar. 23 Fetüs 36-40. haftalarda dış ortama artık uyum | 22 | | | | |
| Fetüs 36-40. haftalarda dış ortama artık uyum | | | | | |
| | 23 | | | | |
| | | , | | | |

## EK-3.Bilişsel Yük Ölçeği

Bu ölçek ile "Normal Gebelikte Hafta Hafta Fetal Gelişim" konusunu öğrenirken zihninizde oluşan bilişsel yükün belirlenmesi amaçlanmıştır. Vereceğiniz bilgiler sadece bilimsel araştırma amaçlı kullanılacaktır.

Kullandığınız ders materyali ile "Normal Gebelikte Hafta Hafta Fetal Gelişim" konusunu çalışırken zihinsel/bilişsel olarak ne kadar çaba sarfettiniz? (1 ile 9 arasında derecelendirme

| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
|---|---|---|---|---|---|---|---|---|

Az Çok

### EK-4.Bulunuşluk Hissi Ölçeği

Yaşamış olduğunuz sanal gerçeklik deneyimini aşağıdaki şekilde belirtildiği gibi 1'den 5'e kadar puanlayınız. İşaretleme seçeneklerin de geçerli olabileceğini unutmayınız. Soruları dikkatli bir şekilde okuyarak sırasıyla ve birbirinden bağımsız olaral Hiçbir soruyu boş bırakmayınız ve verdiğiniz cevabı değiştirmeyiniz.

#### DENEYİMLEDİĞİN ORTAM İLE İLGİLİ OLARAK;



#### EK-4 (devam)



### EK-4 (devam)

#### ENGELLEDİ

24. Ortamdaki görev veya etkinlikleri yerine getirmek için kullanılan sistemlerden çok verilen görevlere veya etkinliklere ne kadar konsantre olabildin?



26. Nesneleri fiziksel etkileşim yoluyla tanımak (bir nesneye dokunmak, bir yüzeyin üzerinde yürümek veya bir duvar veya nesneye çarpmak) ne kadar kolay oldu?



27. Sanal ortam deneyimi sırasında ortama veya göreve tamamen odaklandığını hissettiğinanlar oldu mu?



28. Sanal ortamla etkileşim kurmak için kullanılan kontrol cihazlarına ne kadar kolay uyum sağladın?



29. Sanal ortamda farklı duyularla sağlanan bilgiler (örneğin; görme, duyma, dokunma) tutarlı mıydı?



### Ek-5. Fetal Gelişimi Değerlendirme Bilgi Ölçeği Etik Kurul Onayı

Evrako Tarib 148875 12.03.2021-18875



#### T.C. SAĞLIK BİLİMLERİ ÜNİVERSİTESİ Hamidiye Bilimsel Araştırmalar Etik Kurulu

Sayı : E-46418926-050.01.04--18875

Konu : Araştırma Projesi Değerlendirme Raporu

(21/196)

Sayın Prof. Dr. Saadet YAZICI

Kurulumuza değerlendirilmek üzere sunulan, 21/196 kayıt numaralı "*Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ)'nin Geliştirilmesi*" başlıklı proje önerisi kurulumuzun 26.02.2021 tarihli toplantısında değerlendirilmiş ve kurul kararında etik açıdan uygun bulunmuştur. İlgili kurul kararı Ek'te sunulmuştur.

Bilgilerinize rica ederim.

Prof. Dr. Fatih GÜLTEKİN Başkan

Ek:Kurul Kararı

Bu belge, güvenli elektronik imza ile imzalanmıştır.

Belge Doğrulama Kodu :\*BEKR4E0DC\* Pin Kodu :86691

Belge Takip Adresi : https://www.turkiye.gov.tr/sbu-ebys Bilgi için: Ayşe OKUTAN Unvanı: Mühendis

Adres:Mekteb-i Tibbiye-i Şahane Kampūsū, Tibbiye Cad. No:38 Selimiye Telefon:0216 346 36 38 Faks:0216 346 36 40 Web:http://sbu.edu.tr Kep Adresi:sbu@hs01.kep.tr



Bu belge,güvenli elektronik imza ile imzanlamıştır.

Evrak Tarih ve Sayısı: 01.03.2021-794





#### T.C. SAĞLIK BİLİMLERİ ÜNİVERSİTESİ HAMİDİYE BİLİMSEL ARAŞTIRMALAR ETİK KURULU

Toplanti Tarihi : 26.02.2021 Toplanti Sayisi : 2021/8 Karar Sayisi : 8/9

Kurulumuza değerlendirilmek üzere sunulan, Prof. Dr. Saadet YAZICI'nın sorumlu araştırmacı, Öğr. Gör. Sebahat Hüseyinoğlu ve Öğr. Gör. Reyhan Aydın Doğan'ın yardımcı araştırmacı olduğu 21/196 kayıt numaralı "Fetal Gelişimi Değerlendirme Bilgi Ölçeği (FEGBÖ)'nin Geliştirilmesi" başlıklı proje önerisi kurulumuzun 26.02.2021 tarihli toplantısında değerlendirilmiş ve kurul kararında etik açıdan uygun bulunmuştur.

#### Aslı Gibidir **e-imzalıdır** Prof. Dr. Fatih GÜLTEKİN Başkan

Prof. Dr. Günseli GÜVEN POLAT Başkan Yardımcısı

Doç.Dr. Yasemin AYDIN KARTAL Etik Kurul Üyesi

Dr. Öğr. Üyesi Elif GÜLTEKİN Etik Kurul Üyesi

Dr. Öğr. Üyesi Eray Metin GÜLER Etik Kurul Üyesi

Dr. Öğr. Üyesi Şükran ÖZDATLI KURTULUŞ Etik Kurul Üyesi

> Dr. Öğr. Üyesi Erhan ALABAY Etik Kurul Üyesi

Doç.Dr. Papatya KELEŞ Etik Kurul Üyesi

Dr. Öğr. Üyesi Banu BAYRAM Etik Kurul Üyesi

Dr. Öğr. Üyesi Semra AÇIKSÖZ Etik Kurul Üyesi

Dr. Öğr. Üyesi Enes AKYÜZ Etik Kurul Üyesi

Dr. Öğr. Üyesi Merve KOLCU Etik Kurul Üyesi

> Ayşe OKUTAN Mühendis

## Ek 6.Literatür doğrultusunda oluşturulan hafta hafta fetal boy, kilo ve gelişim.

| Literatür doğrultu | ısunda oluşturulan hafta hafta fetal boy, kilo ve gelişim- 1 |
|---|---|
| Bebeğin popo | , |
| <ol><li>Bebeğin kord</li></ol> | 2. Bebeğin kordonu başta kısa olacak, bebek yukarıya yaklaşabilir. |
| | 3. Bebek büyürken kordonu da uzayarak bebekle birlikte gelişmiş olacak. |
| 4. Kordon başta | kalın daha sonra incelecek |
| HAFTA | GELİŞİM METNİ |
| 3- 8. Haftalar arası | <ul> <li>Beyin omurilik ve kalbin gelişimi başlar.</li> </ul> |
| | <ul> <li>Kol ve bacaklar daha fazla gelişir.</li> </ul> |
| | <ul> <li>Fetal kalp 5. haftanın ortasında düzenli ve ritmik olarak<br/>atmaya başlar.</li> </ul> |
| | <ul> <li>8. haftada embriyoda el ve ayak parmakları oluşmuş<br/>olmasına rağmen perdeler ile birbirine bağlıdır.</li> </ul> |
| 9-12. Haftalar arası | • Embriyo 12. haftadan sonra fetüs ismini alır. |
| | • El ve ayaklardaki perdelenme 11. haftanın sonunda |
| | ortadan kalkar. |
| 13-16. Haftalar arası | • 13. haftada ince lanugo adı verilen vücut tüyleri oluşmaya |
| | başlamıştır. |
| | <ul> <li>Bağırsakların gelişimi 13. haftada başlar.</li> </ul> |
| | <ul> <li>Anne, bebek hareketlerini 16. haftada hissedebilir.</li> </ul> |
| 17-20. Haftalar arası | <ul> <li>Fetüsün mekonyum denilen ilk dışkısı 18. haftada</li> </ul> |
| | oluşmaya başlar. |
| | <ul> <li>Fetüsün saçları 19. haftada çıkmaya başlar.</li> </ul> |
| 25-28. Haftalar arası | <ul> <li>Fetüs 24.haftada gözlerini açıp kapamaya başlar.</li> </ul> |
| 29-32. Haftalar arası | <ul> <li>Fetal kemikler 29. haftada sertleşmeye başlar.</li> </ul> |
| | <ul> <li>32. haftada saçlar kafanın tamamını kaplar.</li> </ul> |
| | • 32. haftada ayak ve el tırnakları uzamaya başlar. |
| 33-38. Haftalar arası | • 37. haftada fetüs, gerinme, irkilme ve parmak emme |
| | hareketlerini yapar. |
| | • 38. hafta içerisinde fetüs sert yakalama refleksi yapar. |
| 38-40 Haftalar arası | • 39. haftada fetüsün saçları ve tırnakları uzamaya devam |
| | eder. |

## Ek-6 (devam)

| Literatür doğrultusunda oluşturulan hafta hafta fetal boy, kilo ve | | |
|---|---|---|
| | gelişim- 2 | |
| HAFTA | BOY | KİLO |
| 6 Hafta | 0.33 cm | 1,13 gram |
| 7 Hafta | 1.27 cm | 1,13 gram |
| 8 Hafta | 1.6 cm | 1 gram |
| 9 Hafta | 2.3 cm | 2 gram |
| 10 Hafta | 3.1 cm | 4 gram |
| 11 Hafta | 4.1 cm | 7 gram |
| 12 Hafta | 5.4 cm | 14 gram |
| 13 Hafta | 7.4 cm | 23 gram |
| 14 Hafta | 8.7 cm | 43 gram |
| 15 Hafta | 10.1 cm | 70 gram |
| 16 Hafta | 11.6 cm | 100 gram |
| 17 Hafta | 13 cm | 140 gram |
| 18 Hafta | 14.2 cm | 190 gram |
| 19 Hafta | 15.3 cm | 240 gram |
| 20 Hafta | 16.4 cm | 300 gram |
| 20 Hafta | 25.6 cm | 300 gram |
| 21 Hafta | 26.7 cm | 360 gram |
| 22 Hafta | 27.8 cm | 430 gram |
| 23 Hafta | 28.9 cm | 501 gram |
| 24 Hafta | 30 cm | 600 gram |
| 25 Hafta | 34.6 cm | 660 gram |
| 26 Hafta | 35.6 cm | 760 gram |
| 27 Hafta | 36.6 cm | 875 gram |
| 28 Hafta | 37.6 cm | 1005 gram |
| 29 Hafta | 38.6 cm | 1153 gram |
| 30 Hafta | 39.9 cm | 1319 gram |
| 31 Hafta | 41.1 cm | 1502 gram |
| 32 Hafta | 42.4 cm | 1702 gram |
| 33 Hafta | 43.7 cm | 1918 gram |
| 34 Hafta | 45 cm | 2146 gram |
| 35 Hafta | 46.2 cm | 2383 gram |
| 36 Hafta | 47.4 cm | 2622 gram |
| 37 Hafta | 48.6 cm | 2859 gram |
| 38 Hafta | 49.8 cm | 3083 gram |
| 39 Hafta | 50.7 cm | 3288 gram |
| 40 Hafta | 51.2 cm | 3462 gram |

EK-7.Sanal gerçeklik teknolojili fetal gelişim uygulamasının referans görselleri











EK-8. Fetal gelişim uygulamasındaki hologramik saat görseli


# EK-9. Fetal Gelişim Teori Eğitim İçeriği





































18

## EK-9 (devam)



kte bu yapıdak ua adını alır.

20

Im plantasyon - de

zigotun üzerini örten desidusya
Desidus kaputurist,
Altindakine
Desidus kaputurist,
Altindakine
Desidus basarın
Desidus vera denit.
Implantasyon srasında zigot,
desidusi maddeleri absorbe
ederek belenit.
Daha sonra beliemesi maternal
kap yoli dis oli

FETAL GELİŞİM

FETÜSÜN BÜYÜME VE GELİŞMESİ

Birinci Trimester(1-13 hafta)

Fetal Growth From 8 to 40 Weeks

25

22

- Organiar hazim olarak büyür ve işinderinde başlar
   Orayayı belirgindeşir ve 13-18 haftalar aranında tüği ile
   Orayayı belirgindeşir ve 13-18 haftalar aranında tüği ile
   Orayalayını 13-2-6, haftalarılan belevi, hiscedilir (il şiş gebelerinle geckendis)
   New York olaranında başlarılanında b

26

III. trimester ( 27-40 hafta)

27



31





# EK-9 (devam)











51

## EK-10.Bilgilendirilmiş Gönüllü Olur Formu (Araştırmaya katılma onayı için)

## BİLGİLENDİRİLMİŞ GÖNÜLLÜ OLUR FORMU

Araştırma Projesinin Adı: Fetal Gelişimin Öğretiminde Sanal Gerçeklik Uygulamasının

Geliştirilmesi ve Kullanılması

Sorumlu Araştırıcının Adı: Prof. Dr. Saadet YAZICI Diğer Araştırıcıların Adı: Öğr. Gör. Reyhan AYDIN

Destekleyici (varsa): BAP (Etik kurul onayı alındıktan sonra başvurulacaktır).

"Fetal Gelişimin Öğretiminde Sanal Gerçeklik Uygulamasının Geliştirilmesi ve Kullanılması" isimli bir çalışmada yer almak üzere davet edilmiş bulunmaktasınız. Bu çalışmaya davet edilmenizin nedeni ebelik bölümü öğrencisi olmanız ve müfredatta işlenen fetal gelişim ve fetal sağlık bilgisini ders içeriğinizde alıyor olmanızdır. Bu çalışma, araştırma amaçlı olarak yapılmaktadır ve katılım gönüllülük esasına dayalıdır. Çalışmaya katılma konusunda karar vermeden önce araştırma hakkında sizi bilgilendirmek istiyoruz. Çalışma hakkında tam olarak bilgi sahibi olduktan sonra ve sorularınız cevaplandıktan sonra eğer katılmak isterseniz sizden bu formu imzalamanız istenecektir. Bu araştırma, Ebelik Anabilim Dalında, Prof. Dr. Saadet YAZICI sorumluluğu altındadır.

#### Calışmanın amacı nedir; benden başka kaç kişi bu çalışmaya katılacak?

Bu başlık altında aşağıdaki bilgiler yer almalıdır:

- Araştırmanın amacı, sanal gerçeklik ortamında, gebelik oluşumu, fetal ve plasental gelişim için sanal gebeliğin tasarlanması ve tasarlanan sanal gebeliğin ebelik eğitimi üzerine etkinliğinin değerlendirilmesidir.
- Çalışmaya kaç kişinin alınmasının planlandığı (tek ya da çok merkezli ise belirtilmesi):

Çalışma tek merkezli bir çalışmadır. Çalışmaya 1 kontrol 2 deney grubu olmak ve her grupta 35 öğrenci olacak şekilde 105 öğrenci ile yapılması planlanmaktadır.

### Bu çalışmaya katılmalı mıyım? (Bu bölüm aynen korunacaktır)

Bu çalışmada yer alıp almamak tamamen size bağlıdır. Şu anda bu formu imzalasanız bile istediğiniz herhangi bir zamanda bir neden göstermeksizin çalışmayı bırakmakta özgürsünüz. Eğer katılmak istemez iseniz veya çalışmadan ayrılırsanız, doktorunuz tarafından sizin için en uygun tedavi planı uygulanacaktır. Aynı şekilde çalışmayı yürüten doktor çalışmaya devam etmenizin sizin için yararlı olmayacağına karar verebilir ve sizi çalışma dışı bırakabilir, bu durumda da sizin için en uygun tedavi seçilecektir.

## Bu çalışmaya katılırsam beni ne bekliyor?

Bu başlık altında aşağıdaki bilgiler yer almalıdır:

- Çalışmanın hangi yöntemlerle gerçekleştirileceği, Çalışma deney ve kontrol grubu olarak tasarlanmış deneysel bir çalışma olması planlanmaktadır.
- Araştırmanın süresi 12 aydır. 15.03.2020-15.02.2021 tarihleri arasında planlanmaktadır. Siz gönüllülere uygulanacak olan süreç ise
- Tüm gönüllülere müfredatlarında olan fetal gelişim derste anlatılacak ve ölçekler uygulanacaktır bu süre 4 saat sürecektir. 6 ay sonrasında da aynı ölçeklerle değerlendirme yapılacaktır.
- Deney I grubundaki öğrencilere eğitim sonrasında fetüsün hafta hafta gelişim evrelerini içeren araştırmacılar tarafından hazırlanan bilgisayar destekli ve yönergeli sanal gerçeklik uygulaması izletilecektir. 6 ay sonrasında da aynı ölçeklerle değerlendirme yapılacaktır.
- Deney II öğrencilere eğitim sonrasında fetüsün hafta hafta gelişim evrelerini içeren araştırmacılar tarafından hazırlanan bilgisayar desteksiz ve yönergesiz sanal gerçeklik uygulaması izletilecektir. 6 ay sonrasında da aynı ölçeklerle değerlendirme yapılacaktır.
- Hastaya ait biyolojik bir materyal ya da görüntü materyali üzerinde çalışılacaksa tam olarak ne bakılacağı,

(Örnek: Hastalığınız nedeni ile yapılan rutin tetkik ve tedavi işlemleriniz sırasında sizden alınan kanda (.... ml) ...... isimli maddelerin düzeyinin nasıl değiştiği araştırılacaktır.)

### Çalışmanın riskleri ve rahatsızlıkları var mıdır?

1- Herhangi bir risk bulunmamaktadır.

### Örnek:

- 1. ......
- 2. Araştırmadan dolayı göreceğiniz olası bir zararda gerekli her türlü tıbbi girişim tarafımızdan yapılacaktır; bu konudaki tüm harcalamalar da tarafımızdan karşılanacaktır

## Çalışmada yer almamın yararları nelerdir?

Tez başarı ile tamamlandığında, dünyada ve Türkiye'de ilk defa sanal gerçeklik gözlüğü tasarlanmış bir sanal gebelik uygulaması oluşturulmuş olacaktır.

Elde edilen sanal gebelik hem ebelik öğrencileri hem de tüm ebelerin hizmet içi eğitimlerinde kullanılabilen bir uygulama olacaktır. Aynı zamanda bir sonraki sanal gerçeklik uygulamalarına temel hazırlayacaktır.

Ebelik eğitiminde sanal gerçeklik uygulamaların temelini oluşturarak tüm dünyada kullanılabilecek etkin bir yöntem olarak kullanılması hedeflenmektedir.

Ebelik eğitiminde oluşturulacak simülasyon merkezlerinin temelini oluşturacaktır.

### Bu çalışmaya katılmamın maliyeti nedir? (Bu bölüm aynen korunacaktır)

Çalışmaya katılmakla parasal yük altına girmeyeceksiniz ve size de herhangi bir ödeme yapılmayacaktır.

## Kişisel bilgilerim nasıl kullanılacak? (Bu bölüm aynen korunacaktır)

Çalışma doktorunuz kişisel bilgilerinizi, araştırmayı ve istatiksel analizleri yürütmek için kullanacaktır ancak kimlik bilgileriniz gizli tutulacaktır. Yalnızca gereği halinde, sizinle ilgili bilgileri etik kurullar ya da resmi makamlar inceleyebilir. Çalışmanın sonunda, kendi sonuçlarınızla ilgili bilgi istemeye hakkınız vardır. Çalışma sonuçları çalışma bitiminde tıbbi literatürde yayınlanabilecektir ancak kimliğiniz açıklanmayacaktır.

#### Daha fazla bilgi için kime başvurabilirim?

Çalışma ile ilgili ek bilgiye gereksiniminiz olduğunuzda aşağıdaki kişi ile lütfen iletişime geçiniz.

ADI : Öğr. Gör. Reyhan AYDIN GÖREVİ : Yardımcı araştırmacı TELEFON : 0542 266 65 68

## (Katılımcının/Hastanın Beyanı)

Ebelik Anabilim dalında, Prof. Dr. Saadet Yazıcı tarafından tıbbi bir araştırma yapılacağı belirtilerek bu araştırma ile ilgili yukarıdaki bilgiler bana aktarıldı ve ilgili metni okudum. Bu bilgilerden sonra böyle bir araştırmaya "katılımcı" olarak davet edildim.

Araştırmaya katılmam konusunda zorlayıcı bir davranışla karşılaşmış değilim. Eğer katılmayı reddedersem, bu durumun tıbbi bakımıma ve hekim ile olan ilişkime herhangi bir zarar getirmeyeceğini de biliyorum. Projenin yürütülmesi sırasında herhangi bir neden göstermeden araştırmadan çekilebilirim. (*Ancak araştırmacıları zor durumda bırakmamak için araştırmadan çekileceğimi önceden bildirmemim uygun olacağının bilincindeyim*). Ayrıca tıbbi durumuma herhangi bir zarar verilmemesi koşuluyla araştırmacı tarafından araştırma dışı da tutulabilirim.

Araştırma için yapılacak harcamalarla ilgili herhangi bir parasal sorumluluk altına girmiyorum. Bana da bir ödeme yapılmayacaktır.

Araştırmadan elde edilen benimle ilgili kişisel bilgilerin gizliliğinin korunacağını biliyorum.

Araştırma uygulamasından kaynaklanan nedenlerle meydana gelebilecek herhangi bir sağlık sorunumun ortaya çıkması halinde, her türlü tıbbi müdahalenin sağlanacağı konusunda gerekli güvence verildi. (Bu tıbbi müdahalelerle ilgili olarak da parasal bir yük altına girmeyeceğim).

Araştırma sırasında bir sağlık sorunu ile karşılaştığımda; herhangi bir saatte, Öğr. Gör. Reyhan AYDIN, 0542 266 65 68, Karabük Üniversitesi Sağlık bilimleri Fakültesi Ebelik Bölü Kat 3 Oda no M327'den arayabileceğimi biliyorum.

Bana yapılan tüm açıklamaları ayrıntılarıyla anlamış bulunmaktayım. Bu koşullarla söz konusu klinik araştırmaya kendi rızamla, hiçbir baskı ve zorlama olmaksızın, gönüllülük içerisinde katılmayı kabul ediyorum.

İmzalı bu form kağıdının bir kopyası bana verilecektir.

| a |
|------------------------|
| Görüşme tanığ |
| Adı, soyadı:<br>Adres: |
| Tel: |
| İmza: |
| Tarih: |

Not: Aydınlatma ve katılımcının beyanı <u>birbirlerinin devamı</u> şeklinde olmalı ve <u>aynı</u> sayfada yer almalıdır.

# EK-11. Eğitici Eğitimi Sertifikası

| | ENSTİTÜ<br>Öğrenmek Pahalıdır. |
|---|---|
| SERTİFİKA | |
| CERTIFICATE OF ACHIEVEMENT | |
| CERTIFICATE OF ACHIEVEMENT | |
| Reyhan Aydın | |
| Reynan Ayani | |
| Eğiticinin Eğitimi | |
| eğitimini başarıyla tamamlamıştır. | |
| Eğitim Tarihi: 2019-12-15 | |
| Sertifika Kodu: 151293840033 | |
| $\wedge$ $\wedge$ | |
| SILAL S NTÜRK | |
| Enstitü Vönet cisi | |
| HENSTITU Ltd - Enstitü ÖÜ | |
| Türkiye- Estonia | |
| · a.m.y · arrang | |
| Bu sertifika şu URL ile doğrulanabilir: https://www.lienstitu.com/sertifika-sorgulama/sertifika/151293840033 | |

## EK-12. Etik Kurul Onayı



#### T.C. KARABÜK ÜNİVERSİTESİ GİRİŞİMSEL OLMAYAN KLİNİK ARAŞTIRMALAR ETİK KURULU

9/6/2020

Karar No: 2020/263

Sayın Prof. Dr. Saadet YAZICI

Girişimsel Olmayan Klinik Araştırmalar Etik Kurulumuza sunmuş olduğunuz "FETAL GELİŞİMİN ÖĞRETİMİNDE SANAL GERÇEKLİK UYGULAMASININ GELİŞTİRİLMESİ VE KULLANILMASI" başlıklı araştırma projeniz amaç, gerekçe, yaklaşım ve yöntemle ilgili açıklamaları açısından Girişimsel Olmayan Etik Kurulu yönergesine göre incelenmiştir. Etik açıdan bir sakınca olmadığına oy birliği ile karar verilmiş ve uygun görülmüştür. Bilgilerinize rica ederim.

Prof. Dr. Orhan ÖNALAN Girişimsel Olmayan Klinik Araştırmalar Etik Kurulu Başkanı

Ekler:

1-Kurul Üyeleri Değerlendirme Formları

## T.C. KARABÜK ÜNİVERSİTESİ GİRİŞİMSEL OLMAYAN KLİNİK ARAŞTIRMALAR ETİK KURULU PROJE DEĞERLENDİRME FORMU

| Başvuru id: | 263 | Geliş Tarihi: | 2/6/2020 |
|---|---|---|---|
| Araştırma Yürütücüsü: | Prof. Dr. Saadet YAZ | ICI | |
| Araştırmanın Başlığı: | FETAL GELİŞİMİ<br>UYGULAMASININ GI | N ÖĞRETİMİNDE S<br>ELİŞTİRİLMESİ VE KUL | ANAL GERÇEKLİK<br>LANILMASI |
| Araştırmaya dahil edile | | 105 | |

| Araştırma daha önce yapılmış mıdır? | Evet | Hayır X |
|---|---|---|
| Araştırma bir hipotezi test etmek üzere planlanmış mıdır? | Evet X | Hayır |
| Araştırma sonucunda ölçülebilir bir hedefe ulaşmak olası mıdır? | Evet X | Hayır |
| Araştırma çağdaş bilime katkıda bulunacak nitelikte midir? | Evet X | Hayır |
| Araştırma metodolojik yönden doyurucu olarak planlanmış mıdır? | Evet X | Hayır |
| Arastırma protokolünde gönüllü sayıları gercekci midir? | Evet X | Havir |
| Araştırmanın istatistik bilgileri yeterli midir? | Evet X | Hayır |
| Araştırma için en uygun sayıda gönüllü kullanımı amaçlanmış mıdır? | Evet X | Hayır |
| Araştırma gönüllülerin aydınlatılmış onamı alınmış mıdır? | Evet X | Hayır |
| Araştırma uygun yer ve koşullarda yapılacak midir? | Evet X | Hayır |
| Araştırmacı(lar) çalışma ile ilgili yeterli bilgi ve deneyime sahip midir? | Evet X | Hayır |
| Araştırmada çevre ve/veya insan sağlığını tehdit edecek toksik<br>rezidü, kimyasal, biyolojik, radyoaktif maddelerin bulaşma riski<br>var mıdır? | Evet | Hayır X |
| Araştırma sonunda yayın çıkarabilecek nitelikte midir? | Evet X | Hayır |
| Gerekli görülen diğer açıklamalar: | | |
| Değerlendirme Sonucu: | uygun görülmüstür. | |

## EK-13.Bulunuşluk Hissi Ölçeği (BHÖ) Ölçek kullanım izni



## EK-14.Bilişsel Yük Ölçeği (BYÖ) Ölçek kullanım izni





# EK-15.Araştırma Kurum İzni

21/01/2020

Sayın İlgili,

Sorumlu araştırmacısı Prof. Dr. Saadet YAZICI ve Öğr. Gör. Reyhan AYDIN olan "Fetal Gelişimin Öğretiminde Sanal Gerçeklik Uygulamasının Geliştirilmesi ve Kullanılması" isimli projenin veri toplama aşamasını içeren kısmının bölümümüzde yapılması uygundur. Bilgilerinize saygılarımla arz ederim.

Doç. Dr. İşil İşik ANDSOY

EK-16.Bilgilendirilmiş Gönüllü Olur Formu (Uygulamadaki Görüntülerin

Kullanımı İçin)

BİLGİLENDİRİLMİŞ GÖNÜLLÜ ONAM FORMU

(UYGULAMASIRASINDA FOROGRAF ÇEKİLMESİ VE ARAŞTIRMADA

**KULLANILMASI İZNİ)** 

Sayın Katılımcı;

Çalışmayı kabul edip zaman ayırdığınız için teşekkür ederiz. Çalışma kapsamında sanal

gerçeklik uygulamasını deneyimlerken ki fotoğrafınızı, araştırmada görsel olarak

kullanmak için, isminizi ve yüzünüzü görselde görünmeyecek şekilde kullanmak

istiyoruz. Elde edilen bilgiler yalnızca araştırma amacı için kullanılacak, başka bir amaçla

kullanılmayacaktır. Bu araştırmaya katılmanız dahilinde isminiz kullanılmayacak ve

kimlik haklarınız korunacaktır. Bu araştırmaya katılmanız için sizden herhangi bir ücret

istenmeyecektir. Araştırma gönüllülük esasına dayanmaktadır ve istediğiniz zaman

görsellerinizin kullanılmamasını isteme ve çalışmayı bırakma hakkına sahipsiniz.

Bilgilendirilmiş Gönüllü Onam Formundaki tüm açıklamaları okudum.

Araştırmaya gönüllü olarak katıldığımı, istediğim zaman gerekçeli ya da gerekçesiz

olarak araştırmadan ayrılabileceğimi biliyorum. Söz konusu araştırmaya, hiçbir baskı ve

zorlama olmaksızın kendi isteğimle uygulamayı deneyimlerken görsellerimin

kullanılmasını kabul ediyorum

Tarih: ..../20...

Gönüllünün İmzası: